
#### The GlaxoSmithKline group of companies

208466/ADP-04511

| Division | : Worldwide Development |
|------------------|-------------------------------------|
| Information Type | : Reporting and Analysis Plan (RAP) |

Title : A Pilot Study of Genetically Engineered NY-ESO-1 Specific NY-ESO 1c259T in HLA-A2+ Patients with Synovial Sarcoma

Compound Number : GSK3377794

Effective Date : 07-NOV-2019

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 208466/ADP-04511.
- This RAP is intended to describe the planned efficacy and safety analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

#### RAP Author(s):

| Author | Date |
|-----------------------------------------------------------|------------|
| Principal Biostatistician (Oncology, Clinical Statistics) | 28-Oct2019 |

Copyright 2019 the GlaxoSmithKline group of companies. All rights reserved. Unauthorized copying or use of this information is prohibited.


## The GlaxoSmithKline group of companies

208466/ADP-04511

| Reviewer (Method: Email) | Date |
|------------------------------------------------------------|------------|
| Global Medical Director (Oncology, Clinical Development) | 02-Nov2019 |
| Principal Programmer (Oncology, Clinical Programming) | 01-Nov2019 |
| Clinical Development Head (Oncology, Clinical Development) | 04-Nov2019 |
| Clinical Development Lead (Oncology, Clinical Development) | 01-Nov2019 |

## Clinical Statistics and Clinical Programming Line Approvals: (Method: Pharma TMF eSignature)

| Approver | Date |
|---|---|
| Statistics Director (Oncology Clinical Statistics) On behalf of PPD (Senior Statistics Director, Clinical Statistics) | 07-Nov2019 |
| Programming Manager (Oncology Clinical Programming) | 07-Nov2019 |

## 1. TABLE OF CONTENTS

| | | | | PAGE |
|---|---|---|---|---|
| 1. | TABL | E OF CON | NTENTS | 3 |
| 2. | LIST | OF TABLE | ES | 5 |
| 3. | LIST | OF ABBR | EVIATIONS & TRADE MARKS | 6 |
| 4. | INTRO | DDUCTIO | DN | 8 |
| 5. | OVER | ALL STIL | JDY DESIGN AND OBJECTIVES | Ω |
| J. | 5.1. | | Objectives | |
| | 0.1. | 5.1.1. | | |
| | | 5.1.2. | | |
| | | 5.1.3. | Exploratory Objectives | |
| | 5.2. | | sign and Study Procedures | |
| | | 5.2.1. | | |
| | | 5.2.2. | | |
| | 5.3. | Sample | Size | |
| | | • | | |
| 6. | GENE | | ALYSIS CONVENTIONS | |
| | 6.1. | | Periods | |
| | 6.2. | Visit Wir | ndows | 12 |
| 7 | A N I A I . | V010 D01 | DI II ATIONO | 40 |
| 7. | | | PULATIONS | |
| | 7.1. | | o-Treat Population | |
| | 7.2. | | d Intent-to-Treat Population | |
| | 7.3. | Per-Proi | tocol Population | 13 |
| 8. | SUBJ | ECT DISF | POSITION | 13 |
| 9. | PR∩T | | EVIATIONS | 13 |
| ٥. | 11101 | OCOL DI | LVIATIONO | |
| 10. | DEMO | GRAPHI | IC AND BASELINE CHARACTERISTICS | 14 |
| | 10.1. | | raphic Characteristics | |
| | 10.2. | | History | |
| | 10.3. | | ancer Therapy | |
| | _ | | | |
| 11. | | | METHODS FOR EFFICACY | |
| | 11.1. | • | Efficacy Analysis | |
| | 11.2. | Seconda | ary Efficacy Analyses | 16 |
| 12 | CTAT | ICTICAL // | ANALYTICAL ISSUES | 21 |
| 12. | | | | |
| | 12.1.<br>12.2. | | g of Dropouts or Missing Dataof Centers in Multi-Center Studies | |
| | 12.2. | | Comparisons/Multiplicity | |
| | 12.3.<br>12.4. | | ation of Subgroups | |
| | 12.4. | | Analysis and Data Monitoring | |
| | 12.0. | intollin F | , analysis and Data Montoning | |
| 13. | STAT | ISTICAL N | METHODS FOR SAFETY ENDPOINTS | 22 |
| | | | rua Exposure | |


| | 13.2. | Adverse Events | |
|---|---|---|---|
| | 13.3. | Adverse Events of Special Interest (AESI) | |
| | 13.4. | Laboratory Tests | 25 |
| | | 13.4.1. Clinical Laboratory Tests | 25 |
| | | 13.4.2. Persistence of NY-ESO-1 c259T and Replication | 0.0 |
| | | Competent Lentivirus (RCL) | |
| | 13.5. | Vital Signs | |
| | 13.6. | Physical Exams | |
| | 13.7. | Electrocardiograms | 29 |
| | 13.8. | Eastern Cooperative Oncology Group (ECOG) Performance Status | |
| | 13.9. | Concomitant Medications | 29 |
| 14. | QUAL | ITY CONTROL | 30 |
| 15. | TABLE | ES AND LISTINGS CONVENTIONS | 30 |
| 16. | REFE | RENCES | 32 |
| 17. | PRELI | MINARY LIST OF TABLES, LISTINGS, AND FIGURES TO BE | |
| | PROG | RAMMED | |
| | 17.1. | | |
| | 17.2. | Data Listings | |
| | 17.3. | Figures | 41 |
| 18. | APPE | NDICES | 43 |
| | 18.1. | | |
| | | Appendix 2 List of PTs to Be Combined | |
| | 18.3. | Appendix 3 Specification for Collapsing Adverse Event Segments | 48 |
| 1. | COLL | APSING AE SEGMENTS WITH A COMMON AE PREFERRED | |
| | TERM | (PT) INTO UNIQUE EVENTS BASED ON THE START AND END | |
| | | S | 48 |
| | 1.1 | Multiple AE Segments with Overlapped or Continuous Start/End | 48 |
| | 1.2 | Dates | |
| | 1.3 | Create Derived Variables in ADAE ADaM SAS Dataset | |
| 2 | A D D I T | TIONIAL NOTES | |
| 2. | ADDII | TONAL NOTES | 52 |
| 3. | DATA | EXAMPLES | |
| | 3.1 | Case #1: Previous AE End Date is Same as Next AE Start Date | |
| | 3.2 | Case #2: Previous AE Start Date is Same as Next AE Start Date | 54 |
| | 3.3 | Case #3: Next AE Start Date is One Day after Previous AE End Date | 55 |
| | 3.4 | Case #4: Previous AE End Date is Greater Than Next AE Start | |
| | | Date | 55 |

## CONFIDENTIAL

## 2. LIST OF TABLES

| Table 1 | Definition of Baseline | 10 |
|---|---|---|
| Table 2 | Partial or Missing Date Algorithms | 11 |
| Table 3 | Best Overall Response per RECIST v1.1. | 19 |
| Table 4 | Sensitivity Analyses for NE Responses | 21 |
| Table 5 | Potentially Clinically Significant Elevations in Hepatic Parameters | 26 |
| Table 6 | Potentially Clinically Significant Vital Signs Values | 29 |

## 3. LIST OF ABBREVIATIONS & TRADE MARKS

| Abbreviation | Description |
|--------------|------------------------------------------------|
| AE | Adverse Event |
| ATC-2 | Anatomical Therapeutic Chemical 2nd level |
| ATC-3 | Anatomical Therapeutic Chemical 3rd level |
| BMI | Body Mass Index |
| BOR | Best Overall Response |
| BSA | Body Surface Area |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CMV | Cytomegalovirus |
| CR | Complete Response |
| CRP | C-reactive protein |
| CRS | Cytokine Release Syndrome |
| CTCAE | Common Toxicity Criteria for Adverse Events |
| DOR | Duration of Respond |
| DOSD | Duration of Stable Disease |
| ECG | Electrocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | Electronic Case Report Form |
| eCTD | Electronic Common Technical Document |
| GVHD | Graft Versus Host Disease |
| ICH | International Conference on Harmonisation |
| ITT | Intent-to-treat |
| KM | Kaplan-Meier |
| LTFU | Long-Term Follow-Up |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mITT | Modified Intent-to-Treat |
| NCI | National Cancer Institute |
| NE | Not Evaluable |
| ORR | Overall Response Rate |
| OS | Overall Survival |
| PCR | Polymerase Chain Reaction |
| PD | Progression of Disease |
| PFS | Progression-Free Survival |
| PP | Per-protocol |
| PR | Partial Response |
| PT | Preferred Term |
| QTc | QT Interval Corrected for Heart Rate |
| RECIST | Response Evaluation Criteria in Solid Tumors |
| RCL | Replication Competent Lentovirus |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SD | Stable Disease |
| SOC | System Organ Class |

## CONFIDENTIAL

208466/ADP-04511

| Abbreviation | Description |
|--------------|---------------------------|
| TTR | Time to Complete Response |
| ULN | Upper Limit of Normal |
| WHO | World Health Organization |

| Trademarks of the Glaz<br>Group of Comp |
|-----------------------------------------|
| None |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| SAS |

#### 4. INTRODUCTION

This statistical analysis plan (SAP) describes the efficacy and safety analyses that will be performed for Study 208466/ADP-04511, based on the study protocol Version 15, dated 15OCT2018. The SAP should be used in conjunction with the protocol and electronic case report form (eCRF).

#### 5. OVERALL STUDY DESIGN AND OBJECTIVES

## 5.1. Study Objectives

## 5.1.1. Primary Objectives

- Determine the response rate in subjects with unresectable, metastatic or recurrent synovial sarcoma treated with lymphodepletion and Treg depletion followed by adoptive immunotherapy with T cells engineered to recognize an HLA-A2 restricted NY-ESO-1 derived peptide (Cohort 1).
- Determine the response rate and duration of response of adoptive immunotherapy with NY-ESO-1<sup>c259</sup>T cells in subjects with synovial sarcoma and low-level expression of NY-ESO-1 (Cohort 2).
- Determine the response rate and duration of response of adoptive immunotherapy with NY-ESO-1<sup>c259</sup>T cells in subjects with synovial sarcoma treated with a lymphodepleting conditioning regimen containing cyclophosphamide as a single cytotoxic agent (Cohort 3).
- Determine the response rate and duration of response of adoptive immunotherapy with NY-ESO-1<sup>c259</sup>T cells in subjects with synovial sarcoma treated with a lymphodepleting regimen containing cyclophosphamide and fludarabine cytotoxic agents at reduced total doses (Cohort 4).

## 5.1.2. Secondary Objectives

- Determine the safety of treatment with adoptively transferred NY-ESO-1<sup>c259</sup>T cells.
- When possible, assess whether subjects with progressive disease following NY-ESO-1<sup>c259</sup>T cell infusion or who do not respond experience a response following a second dose.

## 5.1.3. Exploratory Objectives

- Evaluate persistence, phenotype, and functionality of adoptively transferred NY-ESO-1<sup>c259</sup>T cells and correlate with clinical response.
- Evaluate mechanisms of resistance and sensitivity to NY-ESO-1<sup>c259</sup>T cells.
- Evaluate antigen spreading as a mechanism of response.

#### 5.2. Trial Design and Study Procedures

#### 5.2.1. Study Design

This open-label trial was designed as a four Cohort study as of Protocol Amendment 15. Study implementation (including study design) is described in detail in Section 3 of the protocol.

Subjects are eligible for the study if they test positive for HLA-A\*02:01, HLA-A\*02:05, and/or HLA-A\*02:06; are ≥4 years of age; and have NY-ESO-1 expressing unresectable, metastatic or recurrent synovial sarcoma.

Efficacy, safety, and biomarker assessments to be conducted as each visit are outlined in the Schedule of Procedures in Section 10.2 (Appendix 2) of the protocol.

#### 5.2.2. Treatments and Assignment to Treatment

Drug administration details for each of the four cohorts are described in Section 3.3. of the protocol. Subjects in each cohort received lymphodepletion followed by infusion of transduced NY-ESO-1<sup>c259</sup>T cells, then were followed for toxicity, antitumor effects, and immune endpoints. The target dose administered was  $5x10^9$  with a minimum of  $1x10^9$  to a maximum of  $6x10^9$  transduced NY-ESO-1<sup>c259</sup>T cells for subjects  $\geq$ 40 kg. Subjects  $\leq$ 40 kg were dosed per body weight with a minimum  $0.025x10^9$  transduced cells/kg, with a target dose of  $0.125x10^9$  transduced cells/kg.

Second infusions can occur in two settings:

- 1. Patients enrolled onto any cohort who have a confirmed response, or have stable disease for >3 months, then progress, were eligible for a second infusion of NY-ESO-1c259T, provided eligibility criteria are met. Patients with confirmed responses or stable disease that qualify for a second infusion will receive lymphodepleting chemotherapy and T cell infusion as received for the first infusion.
- 2. Patients in Cohort 3 and 4 who have progressive disease or stable disease  $\leq$  3 months as best response, may receive a 2nd treatment of NY-ESO-1c259T using the Regimen A lymphodepletion to determine if more intense lymphodepletion can result in an improved best response.

Patients may receive a maximum of two treatments with NY-ESO-1c259T. The second cycle (i.e. re-treatment) can be given no sooner than 60 Days from the first infusion and no later than 2 years after the first infusion. Decisions to retreat with a second infusion will be discussed with the Sponsor and Investigators.

## 5.3. Sample Size

The sample size for each cohort is based on clinical judgment. The study is not statistically powered to conduct hypothesis testing between cohorts.

#### 6. GENERAL ANALYSIS CONVENTIONS

With respect to the primary objectives and endpoints, no specific statistical hypotheses will be evaluated. All analyses will be descriptive and exploratory.

In the protocol and eCRF, the date of the first T cell infusion is referred to as Day 0.For the tables, listings, and figures, the date of the first T cell infusion will be referred to as Day 1 to be consistent with CDISC data standards.

Data collected in this study will be documented using summary tables and subject data listings. Continuous variables will be summarized using descriptive statistics (number of subjects, mean, median, standard deviation, minimum, and maximum). Categorical variables will be summarized using frequencies and proportions. Time-to-event data will be summarized via Kaplan-Meier (KM) methodology using the 25th, 50th (median), and 75th percentiles with associated 2-sided 95% confidence intervals (CIs) using the complementary log-log transformation, as well as the proportion of censored observations. The 95% CIs for proportions will be calculated using Wilson and exact confidence limits.

Because of the small number of expected subjects receiving a second infusion, only select adverse events tables will be prepared for data on subjects who receive a second infusion. Efficacy data will be summarized in tables and listings.

Assessments will be displayed for each Cohort and for all Cohorts combined (i.e., overall).

Unless specified otherwise, baseline measurements should be the most recent value prior to initiating lymphodepletion and should occur within 7 days prior to initiating lymphodepletion (Table 1). If an assessment is not available, then the last assessment prior to that visit would be used.

Table 1 Definition of Baseline

| Assessment/Test | Visit |
|---|---|
| Target and Non-target Lesions | Baseline within 7 days prior to initiating |
| | lymphodepletion |
| Demography | Date of Screening Informed Consent |
| Hematology, Chemistry, C-reactive | Baseline within 7 days prior to initiating |
| protein (CRP), CMV PCR, Additional | lymphodepletion |
| Lab | |
| Vital Signs, Physical Exam, ECOG | Baseline within 7 days prior to initiating |
| | lymphodepletion |
| Electrocardiograms | Baseline within 7 days prior to initiating |
| | lymphodepletion |
| Cytokines | Baseline within 7 days prior to initiating |
| | lymphodepletion |

Algorithms for imputing partial or missing dates are shown in Table 2. If a period determination cannot be made for an adverse event, it will be attributed to the post-lymphodepletion period (described in Section 6.1), with missing dates imputed as explained in Table 2. AE end dates are imputed to facilitate calculation of AE duration. Note: Only SAEs are collected prior to leukapheresis.

Table 2 Partial or Missing Date Algorithms

| Variable | Missing Day | Missing Day, Month | Missing Day, Month,<br>Year |
|---|---|---|---|
| Date of Last Systemic<br>Therapy/Date of Initial<br>Diagnosis | Assign 1 | Assign January 1 if prior<br>to date of informed<br>consent, otherwise use<br>date of informed consent | Missing (do not impute) |
| Adverse Event Start Date | Assign first day of month unless it is the month of start of lymphodepletion. Otherwise, assign date lymphodepletion started. | Assign January 1 unless<br>the year is year of start<br>of lymphodepletion<br>Otherwise, assign date<br>lymphodepletion started. | Assign date lymphodepletion started. |
| Adverse Event End Date | Assign the last day of<br>the month or end of<br>study date, whichever is<br>earlier. | Assign December 31 or end of study date, whichever is earlier. | If ongoing, end date is missing. Otherwise, assign end of study date. |

Missing date information for concomitant medication will not be imputed.

Medical history, adverse events and concurrent procedures will be coded using Medical Dictionary for Regulatory Activities (MedDRA), Version 22.0 or higher. Prior and concomitant medications will be coded using the World Health Organization (WHO) Drug Dictionary (December 2015 or later).

Data for all subjects in the clinical database will be included in the data listings. Calculated (derived) variables will be listed as appropriate. All tables, listings, and figures will be programmed using SAS Version 9.3 or higher.

A list of proposed statistical tables, data listings, and figures is provided in Section 17.

BSA (m<sup>2</sup>) will be presented as reported on the eCRF.

BMI will be computed as weight in kg/height in m^2

#### 6.1. Study Periods

Subjects undergo leukapheresis within 7 days of the screening visit. Following leukapheresis, cells are transduced. A baseline visit occurs within 7 days prior to initiating chemotherapy for lymphodepletion. The T cell infusion occurs at most 7 days

following chemotherapy depending on the Cohort. The interventional phase is the period from initiation of chemotherapy for lymphodepletion through the date of discontinuation or up to 5 years after the last T cell infusion, whichever is earlier Subjects are followed for 15 years after infusion, or until death, lost to follow-up, or withdrawal of consent, whichever comes first.

For the purposes of adverse event reporting, the following visit intervals will apply:

- Pre-leukapheresis Period: Date screening ICF signed to the date before leukapheresis – only serious adverse events (SAEs) will be reported for screened subjects
- Date informed consent signed (Screening) to end of study (Period 1)
- Day 1 of lymphodepletion to end of study (Period 2)

Period 1 adverse events will be summarized for the intent-to-treat population unless otherwise specified. Period 2 adverse events will be summarized for the modified intent-to-treat population.

Period 2 is clinically relevant for summarizing safety in the context of lymphodepletion and T-cell therapy because Period 1 includes safety results prior to lymphodepletion and T-cell therapy.

#### 6.2. Visit Windows

Study visits are expected to occur according to the protocol schedule. All data will be tabulated per the evaluation visit as recorded on the eCRF even if the assessment is outside of the visit window. In data listings, dates and study day relative to T cell infusion (Study Day 1) will be presented. Note: for time-to-event analyses, evaluations will be based on the actual date of the event rather than on the visit on which the event was reported.

#### 7. ANALYSIS POPULATIONS

The number of subjects in each study population will be summarized.

## 7.1. Intent-to-Treat Population

The intent-to-treat (ITT) population will include all subjects who were enrolled in the trial (i.e., underwent leukapheresis). The ITT population will be used to assess the efficacy and safety of the T cell therapy regimen.

## 7.2. Modified Intent-to-Treat Population

The modified intent-to-treat (mITT) population will include all subjects who receive NY-ESO-1<sup>c259</sup>T cell infusion. The mITT population is the primary analysis population for both safety and efficacy. If the ITT and mITT populations are the same, only analyses associated to the ITT population will be reported.

## 7.3. Per-Protocol Population

A per-protocol population (PP) may be included if there are subjects in the mITT population who have protocol deviations that are expected to affect efficacy assessments (e.g., subjects enrolled who do not meet key eligibility criteria) during the trial. Exclusions from the per protocol population will be identified and documented prior to database lock.

#### 8. SUBJECT DISPOSITION

Subject disposition will be summarized by Cohort, Cohorts 2-4 combined and overall for all subjects who entered the study (i.e., signed the informed consent for the study) and will include the number of subjects in each population (ITT, mITT, PP if applicable) and reasons subjects were removed from a population. The number of subjects receiving lymphodepleting chemotherapy will also be summarized. The number and proportion of subjects who complete the trial, as well as those exiting the interventional phase for each reason specified on the eCRFs will also be summarized. A subject will be considered to have completed the trial when he/she has confirmed progression of disease or death, or when the subject is in the trial for 5 years after the last T cell infusion. Reasons for early termination from the study are:

- Disease Progression
- Unacceptable toxicity and other safety reasons
- Death
- Investigator discretion
- Subject withdrew consent
- Protocol deviation
- Lost to follow-up
- Termination by Sponsor
- Failed manufacture of cell product
- Pregnancy
- Failed to meet eligibility criteria for the second infusion.

Leukapharesed or T-cell infused subjects excluded from analysis populations will be presented in a data listing.

#### 9. PROTOCOL DEVIATIONS

Subjects will be excluded from the per protocol population if they have protocol deviations expected to affect efficacy assessments, these may include the following, and possibly others not listed here:

- Did not meet key inclusions criteria (e.g., did not meet disease requirements)
- Received less than 1 billion transduced NY-ESO-1<sup>c259</sup>T cells (or less than 0.025x10<sup>9</sup> cells/kg if <40kg).
- Had a post baseline tumor resection
- Took prohibited medication

- Developed withdrawal criteria during the study but were not withdrawn
- Did not have at least one post-treatment tumor assessment
- Had different imaging methods for baseline and post-baseline assessments

Protocol deviations will be presented by Cohort and subject in a data listing.

#### 10. DEMOGRAPHIC AND BASELINE CHARACTERISTICS

#### 10.1. Demographic Characteristics

Demographic and baseline characteristics at study entry will be summarized by Cohort and overall for the ITT and mITT populations. Variables to be summarized are:

- Continuous variables
  - Age (years) at time of screening informed consent
  - Weight (kg, converted from pounds if necessary)
  - Height (cm, converted from inches if necessary)
  - Body surface area (BSA) (m<sup>2</sup>)
  - BMI [(weight in kg)/(height in m)<sup>2</sup>]
- Categorical variables
  - Sex
  - Race
  - Ethnicity
  - NY-ESO status
  - HLA status (HLA-A\*0201, HLA-A\*0205, HLA-A\*0206, Other)
  - ECOG performance status at baseline
  - Primary disease site at enrollment
  - Disease stage at enrollment
  - Histology grade at enrollment

Demographic and baseline characteristics will be presented by Cohort and subject in data listings.

## 10.2. Medical History

Medical history will be summarized by Cohort and overall for the ITT population. Medical history information will be presented by Cohort and subject in a data listing.

## 10.3. Prior Cancer Therapy

All prior cancer therapies should have an end date prior to screening Informed Consent date. Additionally, all prior cancer therapies taken from after apheresis and before lymphodepletion (i.e., bridging therapies) will be summarized.

Prior systemic therapy, radiotherapy, surgery history, and bridging therapies will be summarized for the ITT and mITT populations by Cohort and overall. The following variables will be summarized:

• Prior systemic therapy (yes/no)

- Type of systemic therapy
- Time since last systemic therapy (days)
- Time since initial diagnosis (days)
- Best response to last systemic therapy
- Prior radiotherapy (yes/no)
- Prior cancer-related surgery (yes/no)
- Bridging therapy (yes/no)
- Type of bridging therapy (chemotherapy, radiation, other)

Bridging therapy is therapy administered on or after apheresis and before lymphodepletion.

Time since last systemic therapy is calculated as the date the informed consent was signed minus the latest therapy end date, expressed in days, and will be summarized using descriptive statistics. Time since initial diagnosis is calculated as the date the informed consent was signed minus the date of initial diagnosis, expressed in days, and will be summarized using descriptive statistics. Partial dates for date of last systemic therapy and time since initial diagnosis will be imputed as described in Section 6. Only positive values will be summarized for time since last systemic therapy and time since initial diagnosis. Number of lines of prior systemic therapy will be summarized using descriptive statistics and will also be categorized and summarized using counts and percentages. All other variables listed above will be summarized using counts and percentages.

Yes/no variables for prior systemic therapy, prior radiotherapy, and prior cancer-related surgery will be derived from the presence or absence of this information in the raw datasets, as there is no specific question on the eCRF for these variables.

Prior systemic therapy, radiotherapy, and surgery history information will be presented by Cohort and subject in a data listing.

#### 11. STATISTICAL METHODS FOR EFFICACY

The study objectives are described in Section 5.1.

## 11.1. Primary Efficacy Analysis

The primary analysis population for primary and secondary efficacy endpoints will be the mITT population. ITT will be used as the secondary population for analysis of the primary endpoint. The primary efficacy endpoint is the overall response rate (ORR). ORR is defined as the proportion of subjects with a confirmed complete response (CR) or partial response (PR) relative to the total number of subjects in the corresponding analysis population per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) as determined by the local investigators. To be assigned a status of a CR or PR, changes in tumor measurements must be confirmed by repeat assessments that should be performed

at least 4 weeks after the criteria for response are first met. Subjects with unknown or missing response will be treated as non-responders, that is, they will be included in the denominator when calculating the proportion.

Response categories are confirmed CR, confirmed PR, stable disease (SD), and progressive disease (PD). Response confirmation will be handled according to Table 3 (RECIST v1.1) in the next section.

Sensitivity analyses to be performed for ORR defined by RECIST v1.1 include:

- Two-sided 95% CIs for ORR will be calculated using both the Wilson and Clopper-Pearson methods
- ORR analyses repeated for the PP population (if a PP population is defined)
- Investigator assessed response

Listings of response data and lesion measurements per RECIST v1.1 will also be provided.

## 11.2. Secondary Efficacy Analyses

The key secondary efficacy endpoints are

- Time to confirmed response (TTR)
- Duration of response (DOR)
- Progression-free survival (PFS)
- Overall survival (OS)

Additional clinically relevant endpoints include best overall response (BOR) duration of stable disease (DOSD), and time on study (defined as date of last visit in study – date of informed consent +1).

The secondary efficacy analyses will be performed for the mITT population, that is, subjects who received T-cell infusion, which is the primary population for efficacy analysis. Efficacy endpoints will be based on RECIST v1.1.

Time to confirmed response (CR or PR) (reported in weeks) is defined as the interval between the date of first T-cell infusion and the earliest date of first documented confirmed CR or confirmed PR among participants with a confirmed PR or CR.

Duration of response (reported in weeks) is defined as the time from first documented evidence of confirmed CR or confirmed PR until first documented date of disease progression or death due to any cause or surgical resection or start of prohibited medications. For responders who are still alive and who do not have documented disease progression, surgical resection, or prohibited medication the date of the last disease assessment is used.

PFS (reported in weeks) is defined as the interval between the date of first T cell infusion and the earliest documented evidence of disease progression or death due to any cause or surgical resection or start of prohibited medications. Subjects who do not have a

documented date of progression, death, surgical resection, or prohibited medication will be censored at the date of the last disease assessment.

Subject will be censored for PFS and DOSD at the day 1 for the situation the censoring algorithm calls for the subject to be censored at the date of the last disease assessment but no such assessment exists.

#### **Extended Loss to Follow-up**

For the analysis of PFS, if there are two or more consecutive scheduled disease assessments which are missing and are then followed by an assessment demonstrating disease progression or death (due to any cause) or surgical resection or start of prohibited medications, PFS will be censored at the last adequate disease assessment prior to progression or death or surgical resection or start of prohibited medications. For this type of censoring due to extended loss to follow-up, the 'last adequate disease assessment' will be defined as the date of the last radiological assessment prior to the missing assessments that shows no disease progression.

As the assessment schedule changes through the course of the study (i.e. every 4 weeks during the first 12 weeks and then every 3 months until month 24 and then every 6 months after month 24), the following rules will be used for identifying extended loss to follow up.

- If PFS event is on or prior to week 12, then a subject will be identified as an extended loss to follow up if the subject did not have an adequate disease assessment during the time period of 56 days (8 weeks) prior to PFS event;
- Else if PFS event is after week 12 and on or prior to the first scheduled disease assessment date (month 6, day 183) during week 12 to month 24, then a subject will be identified as an extended loss to follow up if the subject missed both week 8 and week 12 disease assessments:
  - o If PFS event is after week 12 and on or prior to day 122 (month 4), then a subject will be identified as an extended loss to follow up if the subject did not have an adequate disease assessment during the time period of 56 days (8 weeks);
  - Else if PFS event is after week 12 and on or prior to day 153 (month 5), then a subject will be identified as an extended loss to follow up if the subject did not have an adequate disease assessment during the time period of 84 days (12 weeks);
  - Else if PFS event is after week 12 and on or prior to day 183 (month 6), then a subject will be identified as an extended loss to follow up if the subject did not have an adequate disease assessment during the time period of 112 days (16 weeks);
- Else if PFS event is after day 183 (month 6) and on or prior to the second scheduled disease assessment date (month 9, day 274) during week 12 to month

- 24, then a subject will be identified as an extended loss to follow up if the subject missed both week 12 and month 6 disease assessments:
  - o If PFS event is after day 183 (month 6) and on or prior to day 214 (month 7), then a subject will be identified as an extended loss to follow up if the subject did not have an adequate disease assessment during the time period of 120 days (4 weeks + 3 months);
  - Else if PFS event is after day 183 (month 6) and on or prior to day 244 (month 8), then a subject will be identified as an extended loss to follow up if the subject did not have an adequate disease assessment during the time period of 150 days (4 weeks + 4 months);
  - Else if PFS event is after day 183 (month 6) and on or prior to day 274 (month 9), then a subject will be identified as an extended loss to follow up if the subject did not have an adequate disease assessment during the time period of 181 days (4 weeks + 5 months);
- Else if PFS event is after day 274 (month 9) and on or prior to day 731 (month 24), then a subject will be identified as an extended loss to follow up if the subject did not have an adequate disease assessment during the time period of 183 days (6 months);
- Else if PFS event is after day 731 (month 24) and on or prior to day 914 (24 months + 6 months), then a subject will be identified as an extended loss to follow up if the subject missed both month 21 and month 24 disease assessments;
  - If PFS event is after day 731 (month 24) and on or prior to day 822 (month 27), then a subject will be identified as an extended loss to follow up if the subject did not have an adequate disease assessment during the time period of 183 days (6 months);
  - Else if PFS event is after day 822 (month 27) and on or prior to day 914 (month 30), then a subject will be identified as an extended loss to follow up if the subject did not have an adequate disease assessment during the time period of 274 days (6 months + 3 months);
- Else if PFS event is after day 914 (month 30) and on or prior to day 1096 (month 36), then a subject will be identified as an extended loss to follow up if the subject missed both month 24 and month 30 disease assessments;
  - o If PFS event is after day 914 (month 30) and on or prior to day 1005 (month 33), then a subject will be identified as an extended loss to follow up if the subject did not have an adequate disease assessment during the time period of 274 days (6 months + 3 months);
  - Else if PFS event is after day 1005 (month 33) and on or prior to day 1096 (month 36), then a subject will be identified as an extended loss to follow

up if the subject did not have an adequate disease assessment during the time period of 366 days (12 months);

• Else if PFS event is after day 1096 (month 36), then a subject will be identified as an extended loss to follow up if the subject did not have an adequate disease assessment during the time period of 366 days (12 months);

Overall survival (reported in weeks) is defined as the interval between the date of the first T-cell infusion and date of death from any cause. Subjects who are still alive or who are lost to follow-up will be censored at the date of last contact.

Best overall response is the best response recorded from the start of treatment (first T cell infusion) until disease progression/recurrence. Response categories from best to worst are: confirmed CR, confirmed PR, SD and confirmed PD. The handling of response confirmation will be handled according Table 3 (RECIST v1.1). Duration of stable disease must be at least 4 weeks to qualify SD as the BOR. If a subject did not have confirmed CR or PR and had stable disease for less than 4 weeks, BOR will be PD.

Table 3 Best Overall Response per RECIST v1.1.

| Overall Response | Overall Response | Best Overall Response |
|---|---|---|
| First time point | Subsequent Time Point | |
| CR | CR | CR |
| CR | PR | SD, PD, or PR* |
| CR | SD | SD provided minimum criteria for SD duration met**, otherwise PD |
| CR | PD | SD provided minimum criteria for SD duration met**, otherwise PD |
| CR | NE | SD provided minimum criteria for SD duration met**, otherwise NE |
| PR | CR | PR |
| PR | PR | PR |
| PR | SD | SD |
| PR | PD | SD provided minimum criteria for SD duration met**, otherwise PD |
| PR | NE | SD provided minimum criteria for SD duration met**, otherwise NE |
| NE<br>*HS GP: 1 | NE | NE NE |

\*If CR is truly met at first time point, then any disease seen at a subsequent time point, even disease meeting PR criteria relative to baseline, makes the disease PD at that point (since disease must have reappeared after CR). Best response would depend on whether minimum duration for SD was met. However, sometimes 'CR' may be claimed when subsequent scans suggest small lesions were likely still present and in fact the patient had PR, not CR at the first time point. Under these circumstances, the original CR should be changed to PR and the best response is PR.

\*\* Minimum criteria for SD disease duration is at least 4 weeks to qualify SD as BOR.

Note: If Best Overall Response is CR or PR, the subject is classified as a responder for the ORR analysis.

Duration of stable disease (reported in weeks) is defined as the interval between the date of first T cell infusion and the earliest documented evidence of PD. Subjects who do not have documented evidence of PD will be censored at the date of the last assessment.

No hypothesis testing is planned for these secondary endpoints. Time to event endpoints will be summarized and displayed graphically using KM methodology to estimate the median, and the 25th and 75th percentiles and associated 2-sided 95% CIs using the complementary log-log transform. Overall survival may be assessed at fixed time points

such as 1 year and 2 years using KM methods. The proportion of censored observations will be summarized.

Sensitivity analyses will be performed for BOR, DOR, and PFS as follows:

- Summaries based on the PP population (if a PP population is defined)
- In cases where a tumor assessment has a value of NE (missing or unknown), sensitivity analyses will be performed assigning values of PD and SD (PFS only)
- For PFS, subjects who received surgical resection or prohibited medications prior to documented disease progression then PFS will be censored at the date of the last adequate disease assessment
- Based on investigator assessment
- In cases where a tumor assessment has a value of NE (missing or unknown), sensitivity analyses will be performed ignoring the assessment with a value of NE
- In cases where a tumor assessment has a value of not evaluable (NE) (i.e., missing or unknown), sensitivity analyses will be performed assigning values of SD if the assessments before and after the NE assessment are CR, PR, or SD. and will assign PD otherwise, except for PR NE CR where the assessment is improving, as shown in Table 4. (per RECIST v1.1.)

| | Sensitivity Analysis 1: SD Replaces NE at the second |
|---|---|
| Responses at Time Points 1, 2, 3 | time point |
| CR-NE-CR | SD |
| CR-NE-PR | SD |
| CR-NE-SD | SD |
| CR-NE-PD | PD |
| CR-NE-NE | PD |
| PR-NE-CR | SD |
| PR-NE-PR | SD |
| PR-NE-SD | SD |
| PR-NE-PD | PD |
| PR-NE-NE | PD |

Other sensitivity analyses may be performed as appropriate.

Subject response characteristics and time on study will be shown on a swim lane plot. Time on study will be calculated as (date of last assessment for ongoing subjects or discontinuation date) – date of first T cell infusion).

Maximal change in target lesions from baseline will be shown in a waterfall plot. Change in target lesions from baseline over time will be shown in a spider plot.

Listings of response data and derivations for secondary endpoints will be provided, along with other relevant data collected on the eCRF.

#### 12. STATISTICAL/ANALYTICAL ISSUES

## 12.1. Handling of Dropouts or Missing Data

Missing dates will be imputed as described in Section 4. Sensitivity analyses for missing data are described in Section 11.1 and Section 11.2.

## 12.2. Pooling of Centers in Multi-Center Studies

Data will not be summarized by study center or for groupings of study centers.

## 12.3. Multiple Comparisons/Multiplicity

No formal statistical testing will be performed; therefore, no adjustments for multiple comparisons or multiplicity are planned.

## 12.4. Examination of Subgroups

No subgroup analyses are planned.

## 12.5. Interim Analysis and Data Monitoring

Futility evaluation was conducted by Adaptimmune for cohorts 2, 3, and 4 after enrolling 5 subjects using stopping criteria described in Section 3.2 of the protocol.

#### 13. STATISTICAL METHODS FOR SAFETY ENDPOINTS

Safety endpoints are:

- Adverse events (AEs), including serious AEs (SAEs) and adverse events of special events (AESI)
- Laboratory assessments, including chemistry, hematology and anti-infused cell (NY-ESO-1<sup>c259</sup>T) antibodies
- Correlation of circulating cytokines with CRS

Other safety assessments include physical exams, vital signs, and concomitant medications.

All safety data will be included in data listings.

## 13.1. Study Drug Exposure

The total number of transduced T cells and a summary of lymphodepleting chemotherapy administration will be summarized for the mITT population by Cohort and overall using descriptive statistics. The number of transduced cells will be summarized overall for subjects with a second T cell infusion.

All dose administration data for lymphodepletion, including cyclophosphamide and fludarabine, and for T cell infusion will be presented by subject in a data listing.

#### 13.2. Adverse Events

Adverse events (AEs) will be summarized separately for each analysis population and Period (as appropriate) as described in Section 6 and as described below. AEs with partial start or end dates will be imputed as described in Section 6.

Adverse events (AEs) will be summarized by Cohort and overall for:

- Period 1: Date informed consent signed (Screening) to end of study for ITT and mITT populations
- Period 2: Day 1 of lymphodepletion to end of study for mITT population only
- Pre-leukapheresis Period: SAEs only for screened subjects.

Adverse events will be summarized by MedDRA (version 22.0) system organ class (SOC) and preferred term (PT) in alphabetic order for SOC and PT within a SOC. AEs will be graded according to the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) version 4.0. Per the request of the clinical team, various Preferred Terms were combined and will be reported together as one term. The combined terms are listed in Appendix 2. Of note, tables that summarize AEs by SOC and PT and fatal AEs will use MedDRA preferred terms. All other AE tables will summarize AEs by the combined terms in Appendix 2.

Only SAEs occurring prior to leukapheresis for screened subjects will be reported for the pre-leukapheresis period.

AEs with partial start or end dates will be imputed as described in Section 4.

An overview summary table of Period 1 (ITT) and Period 2 (mITT) AEs will be presented by Cohort and overall, including the number and proportion of subjects reporting an AE for the following categories:

- Subjects reporting at least one AE
- Subjects reporting at least one treatment-related AE
- Subjects with ≥ Grade 3 AE
- Subjects with  $\geq$  Grade 3 related AEs
- Subjects with ≥ Grade 3 SAE
- Subjects with  $\geq$  Grade 3 related SAEs
- Subjects reporting at least one SAE
- Subjects reporting at least one treatment-related SAE
- Subjects with SAEs with fatal outcome

For subjects who have a second T cell infusion, an overview summary table of post-lymphodepletion AEs associated with the second infusion will be presented, including the number and proportion of subjects reporting an AE for the following categories:

- Subjects reporting at least one AE
- Subjects reporting at least one treatment-related AE
- Subjects reporting at least one SAE
- Subjects reporting at least one treatment-related SAE
- Subjects with SAEs with fatal outcome

The second infusion AE summaries will be summarized across cohorts.

#### 13.2.1. Adverse Events

The number and proportion of subjects by Cohort and overall with the following categories of AEs will be summarized in tables by system organ class and preferred term for Period 1 (ITT and mITT) and Period 2 (mITT):

- Any AE
- Any AE by toxicity grade
- Any AE by relationship to study treatment

- Any  $AE \ge Grade 3$
- Any treatment-related AE  $\geq$  Grade 3
- Any SAE  $\geq$  Grade 3 SAE
- Any treatment-related  $SAE \ge Grade 3$
- Any SAE
- Any treatment-related SAE
- Any SAE with fatal outcome AEs by descending order of PTs (ordered by overall incidence)
- SAEs by descending order of PTs (ordered by overall incidence)

**In addition**, the following summaries will be provided for the pre-leukapheresis period (all screened subjects):

- Any SAE
- Any SAE with fatal outcome
- Any SAE  $\geq$  Grade 3

The number and percentage of subjects who experienced at least one AE will be summarized overall and for each SOC and each PT. The proportion will be based on the number of subjects in the relevant population by Cohort and overall. Each subject will contribute at most one count per summarization category. In other words, if a subject has more than one AE with the same PT, the subject will be counted only once for that PT. Similarly, if a subject has more than one AE for a SOC, the subject will be counted only once in that SOC, listing out all the PTs.

AE toxicity grade will be classified using NCI CTCAE version 4 criteria into 5 categories: Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life threatening and Grade 5 = fatal. If a subject has multiple occurrences of the same SOC or PT, then only the most severe event will be summarized in the tables for that SOC and PT. AEs of grade 3 or higher will also be summarized. A missing toxicity grade will not be imputed.

The relationship of the AE to T cell infusion will be classified into 5 categories: definitely related, probably related, possibly related, unlikely (Cohort 1 only), and not related. AEs will be summarized in the tables as 'related' or 'not related' and listings will display all categories. Treatment-related AEs include definitely related, probably related, unlikely, and possibly related. If a subject has multiple occurrences of the same SOC or PT, only the most related event will be summarized in the tables for that SOC and PT.

For subjects who have a second T cell infusion, the number and proportion of subjects with the following categories of AEs will be summarized in tables by system organ class and preferred term for AEs associated with the second infusion for the postlymphodepletion period.

- Any AE
- Any AE by toxicity grade
- Any AE by relationship to study treatment

#### Any SAE

No formal hypothesis-testing analysis of AE incidence rates will be performed. All reported AEs will be listed in data listings, with a separate listing for AEs associated with a second T cell infusion. By-subject listings also will be provided for all subjects for the following: all AEs, serious AEs, and AEs with intensity grade 3 or above; the listings will identify which AEs are associated with the first T cell infusion and which are associated with the second T cell infusion. In addition, deaths and cause of death will be presented in a data listing.

## 13.3. Adverse Events of Special Interest (AESI)

An adverse event of special interest is a grouping of adverse events that are of scientific and medical concern specific to NY-ESO-1<sup>c259</sup>T cell infusion. As changes to the MeDRA dictionary may occur between the time of the start of the study and the time of the final reporting, the list of terms to be used for each event of interested will be based on the latest listing provided by safety team.

Summaries of the number and percentage of subjects with these events will be provided for each type of events separately. The summary of event characteristics will also be provided, including number of subjects with any event, number of events, number of subjects with any event that is serious, the outcome of the event, maximum grade. The worst-case approach will be applied at subject level for the event outcome, maximum graded, i.e. a subject will only be conted once as the worst case from all the events that subject had. In addition, onset and duration of the first/last occurences for each type of events will be summarized. AE preferred terms will be 'collapsed' (refer to Appendix 3 for the specific rules) when reporting the onset and duration. Of note, if the AE start date is before the lymphodepletion date and the end date is on or after the lymphodepletion date then the start date for calculating the onset of the AE is still the start date of the AE but the start date for calculating the duration of the AE is the lymphodepletion start date.

Additionally, by-subject listings for subjects experiencing AESIs of CRS, GVHD, GBS, Encephalopathy syndrome and Recurrent pancytopenia with bone marrow failure/Aplastic anemia will be provided (MEdDRA preferred terms are listed in Appendix 2). The time course of CRS and Recurrent pancytopenia with bone marrow failure/Aplastic anemia indicating the severity will be graphically displayed.

Boxplots of select cytokines may also be provided for subjects with and without CRS. A timeline plot of CRS indicating the severity of CRS will be created.

## 13.4. Laboratory Tests

## 13.4.1. Clinical Laboratory Tests

Quantitative clinical laboratory results for hematology and clinical chemistry will be summarized at baseline (as defined in Table 1), each scheduled post-baseline visit, and change from baseline to each scheduled visit using descriptive statistics (number of subjects, mean, median, standard deviation, and minimum and maximum values) for each Cohort and overall. Refer to Appendix 1 for a list of safety laboratory tests by category.

Laboratory data will be summarized for the post-lymphodepletion period (mITT population).

Shift tables that present changes from baseline to worst post-baseline values relative to NCI CTCAE version 4 classification ranges will be produced for each Cohort and overall for laboratory parameters with quantitative CTCAE criteria

The number and percentage of subjects with potentially clinically significant post-baseline elevations in hepatic parameters (Table 5) will be summarized by Cohort and overall.

A listing of the subjects with clinically significant post-baseline hepatic elevations will be provided. The listing will contain all of a subject's values for parameters meeting the criteria.

Table 5 Potentially Clinically Significant Elevations in Hepatic Parameters

| Parameter* | Criterion |
|---|---|
| | Criterion |
| ALT, AST and Total Bilirubin Elevations | ≥3 xULN AST and/or ALT and ≥2 xULN total BIL |
| | ≥3 xULN AST and/or ALT and ≥1.5 xULN total BIL |
| | ≥20 xULN |
| ALT Elevations | ≥10 xULN |
| ALT Elevations | ≥5 xULN |
| | ≥3 xULN |
| Total Bilirubin Elevations | >2 xULN |
| Total Billiudii Elevations | >1.5 xULN |

<sup>\*</sup>ALT = Alanine aminotransferase, ALK = Alkaline Phosphatase, AST = Aspartate aminotransferase, BIL = Total bilirubin, ULN = upper limit of normal.

All laboratory parameters will be included in data listings, and values outside of the reference range will be flagged as high or low on the listings.

## 13.4.2. Persistence of NY-ESO-1 <sup>c259</sup>T and Replication Competent Lentivirus (RCL)

Persistence of gene-modified cells is an indicator of exposure and expansion of T cell therapy. Persistence will be monitored in peripheral blood mononuclear cell (PBMC) samples using a PCR-based method for the presence of the specific WPRE or Psi sequences, which are part of the lentiviral vector used to transduce the T cells. Note, vector with WPRE sequence utilized for subjects dosed before 12-Dec-2016 with exception of Subject PPD , who was dosed with Psi vector.

Persistence data is reported from the analysis vendor as:

- Copies/well
- Copies/ug DNA
- Copies/cell

Copies/ug DNA and copies/cell are calculated by analysis vendor as follows:

- copies/μg DNA=copies per well/μg DNA per well
- copies/cell=(copies/µg)x(0.0000063 µg DNA/cell)

In addition, the following calculations will be performed, where Psi is the persistence result from the eCRF:

Cell Persistence = Absolute peripheral gene-marked cell number /  $\mu$ L = (Psi result number / 151515) x (lymphocyte count + monocyte count) x 1000

Percent of gene marked cells per total lymphocyte compartment =  $((Absolute\ peripheral\ gene\ marked\ cell\ number\ /\ \mu L)\ /\ (Lymphocyte\ count\ x\ 1000))\ x\ 100$ 

OF note, for the data directly from vendor post GSK-Adaptimmune transition, the following calculation will be performed: Cell persistence=Absolute peripheral genemarked cell number/ $\mu$ L= copies/cell × (lymphocyte count + monocyte count) × 1000, where copies/cell is reported by analysis vendor.

For persistence value below LLOQ, the following rules will be applied:

| | Reported Copies per<br>ug DNA Result | | Copies per cell | Set Value for<br>Copies per ug<br>DNA |
|---|---|---|---|---|
| <0.0003 | <50.0 | Negative | 0 | 0 |
| <0.0003 | <50.0 | Detectable, <lloq< td=""><td>0.0003</td><td>50</td></lloq<> | 0.0003 | 50 |

Note, sometimes values for copies per cell and copies per ug DNA might be different than above as it depends on the input of DNA, but rule would be the same:

- If interpretive reported result is negative, set values at 0.
- If interpretive reported result is "Detectable, <LLOQ", set values at LLOQ (If <XXX, set at XXX)

Spider plots of persistence (copies/ug DNA) will be used to graphically summarize persistence over time for each subject by responders and non-responders. Maximum persistence during the study and time to maximum persistence will be summarized overall and for responders and non-responders using descriptive statistics and boxplots.

A listing of persistence will be provided and will include coefficient of variation, number of positive replicates, copies/DNA, interpretive result, duration of detectible persistence and time to loss of 25%/50%/75% peak persistence.

Duration of detectable persistence is defined as time from T-cell infusion until persistence is no longer detectable. Persistence above the assay limit of detection but below the lower limit of quantitation is considered for the duration determination, i.e. the time window from infusion until the first instance persistence falls below the detection limit and the interpretive reported result is "Negative." If persistence for a given subject

remains detectable at their last sample collection timepoint, the last observed time is reported and considered as right-censored with a "+" appended to the numerical result. Note, transduced T-cells frequently persist beyond the follow-up period, and hence, the reported duration is directly influenced by length of time the patient is on-study.

Time to loss of 25% of peak persistence will be calculated as the time since T-cell infusion corresponding to observing at least 25% loss of peak persistence. If time to 25% loss of peak persistence is not observed, the last observed time will be reported with a "+". The same procedure will be followed for 50% and 75%.

The proportion of subjects who are RCL positive will be summarized for the mITT population. RCL is reported as "Negative" if copies of VSV-G are <50 copies/ugDNA

RCL and persistence results (raw and derived) will be presented by Cohort and subject in a data listing.

#### 13.4.3. Cytokines

Boxplots of the maximum post-baseline value for select cytokines including IFN gamma IL6, IL8, IL12, IL13, and TNF alpha will be provided for subjects with none or non-serious CRS vs. serious CRS for the mITT population and for responders vs. non-responders. One spider plot and boxplot will be presented per cytokine.

Cytokine results will be presented by subject in a data listing. Subjects with an adverse event of cytokine release symptom (CRS) will be flagged in the listing. If the reported result is "Fail QC" or "CV>25%", then the value will be set to missing. For values deemed < lower limit of quantitation, a value of the laboratory specified lower limit of quantitation divided by 3 will be used. Laboratory specified upper limit of quantitation values will be used for values > upper limit of quantitation. If there are multiple baseline values, the earliest value will be used as baseline.

The missing data rules for cytokines are as follows:

| Reported Result | Set Value |
|---|---|
| Fail QC | Missing |
| CV>25% | Missing |
| <lloq (ex.="" <0.25)<="" td=""><td>LLOQ/3 (ex: 0.0833 calculated from 0.25/3)</td></lloq> | LLOQ/3 (ex: 0.0833 calculated from 0.25/3) |

## 13.5. Vital Signs

A listing of the subjects with potentially clinically significant post-baseline vital signs will be provided. The listing will contain all of a subject's values for parameters meeting the criteria (Table 6).

## Table 6 Potentially Clinically Significant Vital Signs Values

| Parameter | Criterion |
|-------------------------|------------|
| | < 60 bpm |
| Heart Rate | > 100 bmp |
| Systolic blood pressure | ≥ 140 mmHg |
| Diastolic | ≥ 90 mmHg |

Vital signs will be presented by Cohort and subject in a data listing.

## 13.6. Physical Exams

Physical exam results will be presented by Cohort and subject in a data listing.

## 13.7. Electrocardiograms

All ECG, ECHO, MUGA results will be presented by Cohort and subject in data listings.

## 13.8. Eastern Cooperative Oncology Group (ECOG) Performance Status

ECOG performance status results will be summarized by Cohort and overall at baseline, each scheduled post-baseline visit with counts and proportion of subjects with each score for the mITT population. For subjects less than 10 years of age, Lansky scores will be listed instead of ECOG.

If there are multiple assessments on the same visit the worst ECOG status will be used.

#### 13.9. Concomitant Medications

Concomitant medications will be summarized by the WHO Drug Dictionary Anatomical Therapeutic Chemical 3rd level (ATC-3) and preferred name by Cohort and overall for the mITT population. If the 3rd level term is not available, the next available level (e.g., ATC-2) will be used.

The number and proportion of the subjects who took each medication will be tabulated by the ATC-3 level and preferred name for concomitant medications. A subject will only be counted once within each ATC-3 code and within each preferred name.

All concomitant medication data will be listed by subject.

#### 14. QUALITY CONTROL

All data displays and analyses will adhere to the International Conference on Harmonisation (ICH) *Harmonized Tripartite Guideline: Structure and Content of Clinical Study Reports (ICH Topic E3)*.

GSK will review all tables, listings, and figures prior to final database lock. Final SAS datasets, programs and outputs will be transferred to GSK at project completion.

#### 15. TABLES AND LISTINGS CONVENTIONS

Mock-ups for statistical tables and listings will be provided. Final formats for the statistical tables and listings may deviate from these mock-ups upon agreement with GSK.. Footnotes will be used as needed to clarify the information that is presented in the tables and listings. Unless otherwise requested by GSK the term 'subject' will be used in all tables and listings, in accordance with CDISC standards.

The general layout of tables and listings will be as follows:

| GlaxoSmithKline | Page x of y |
|---|---|
| Protocol: GSK208466/ADP-04511 | Run Date: DDMMMYY-HH:MM |
| <population></population> | |
| Listing 16.2_x (or Table 14.x_x | <b>x</b> ) |
| <title>&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;Col 1 Col 2 Col 3 etc&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;Any footnotes&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;File Name: &lt;pathname for SAS program&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;/tbody&gt;&lt;/table&gt;</title> | |

All tables and listings will use landscape orientation. Margins will be at least 2.0 cm at the top and bottom and at least 0.8 cm on the left and right, excluding headers and

footers, in accordance with electronic Common Technical Document (eCTD) guidelines. Font will be Courier New, unless otherwise specified, with an 8-point font size in most cases. Page numbering will be sequential within each table, listing, and figure. Column headers should be in initial capital letters. Units for numeric data will be included when appropriate.

Tables and data listings will be created from different SAS programs. A single program may produce multiple tables or multiple data listings from the same dataset (e.g., all clinical chemistry data listings may be generated by a single program).

#### **Statistical Table Conventions**

Mock-ups for statistical tables will include headers, title numbers, titles, column headers and footers, and a proposed layout for the display of data. The final decision on the precision (i.e., number of decimal places) for presentation of descriptive statistics will be made by GSK after review of draft statistical tables and before database freeze.

#### **Data Listing Conventions**

Mock-ups for data listings will include headers, title numbers, titles, column headers, and footers. Data listings will provide all data collected on the corresponding eCRF page or provided by external vendors, unless otherwise indicated. If there are too many fields to be fit into a single page, data should be grouped logically and the listings will be generated as Part I, Part II, etc.

In general, data listings should include all subjects with data. However, if only subjects who meet a certain condition are listed (e.g., subjects with SAEs) and no subjects meet the condition, the data listing will so indicate.

The sort order for data presented in data listings will be Cohort and subject ID, unless otherwise requested by Updated... Within a subject, data will be listed in chronological order. Whenever possible, formatted values will be displayed (i.e., decoded). Where applicable, calendar date and study day of evaluations/events will be provided in the data listings.

## 16. REFERENCES

Eisenhauer EA, et al. New response evaluation criteria in solid tumors: Revised RECIST guideline (version 1.1) 2009; Eur J Ca 45:228-247.

Wolchok JD, Hoos A, O'Day S, Weber JS, Hamid O, Lebbé C et al. Guidelines for the Evaluation of Immune Therapy Activity in Solid Tumors: Immune-Related Response Criteria Clin Cancer Res 2009;15:7412-7420.

# 17. PRELIMINARY LIST OF TABLES, LISTINGS, AND FIGURES TO BE PROGRAMMED

## 17.1. Statistical Tables

| Table Number | Table Title | Analysis<br>Population |
|---|---|---|
| 6.1001 | Subject Enrollment and Disposition | ITT |
| 6.2001 | Demographic and Baseline Characteristics | ITT |
| 6.2002 | Demographic and Baseline Characteristics | mITT |
| 6.3001 | Summary of Medical History | ITT |
| 6.4001 | Summary of Prior Cancer Therapy | ITT |
| 6.4002 | Summary of Prior Cancer Therapy | mITT |
| 7.1001 | Summary of Overall Response Rate and Best<br>Overall Response for the First Infusion | mITT |
| 7.1002 | Summary of Overall Response Rate and Best<br>Overall Response for the Second Infusion | Subjects with a<br>Second T Cell<br>Infusion |
| 7.2001 | Time in Study, Time to Response, Duration of Response, and Kaplan-Meier Estimate of Duration of Stable Disease | mITT |
| 7.2002 | Kaplan-Meier Estimate of Progression-Free<br>Survival and Overall Survival | mITT |
| 7.2101 | Sensitivity Analyses for Best Overall Response for the First Infusion | mITT |
| 7.2103 | Sensitivity Analyses for Progression-Free<br>Survival | mITT |
| 8.0001 | Summary of Lymphodepleting Chemotherapy Administration for the First Infusion | mITT |
| 8.0002 | Summary of the First T Cell Infusion | mITT |
| 8.0003 | Summary of the Second T Cell Infusion | Subjects with a<br>Second T Cell<br>Infusion |
| 8.1001 | Overall Summary of Adverse Events for Period 1 | ITT |
| 8.1003 | Overall Summary of Adverse Events for Period 2 | mITT |
| 8.1101 | Incidence of Adverse Events by System Organ<br>Class and Preferred Term for Period 1 | ITT |
| 8.1103 | Incidence of Adverse Events by System Organ<br>Class and Preferred Term for Period 2 | mITT |
| 8.1104 | Summary of Adverse Events Grouped by<br>Similarity of Preferred Terms for Period 1 | ITT |
| 8.1106 | Summary of Adverse Events Grouped by<br>Similarity of Preferred Terms for Period 2 | mITT |

| Table Number | Table Title | Analysis<br>Population |
|---|---|---|
| 8.1201 | Incidence of Adverse Events by Toxicity Grade and Preferred Term for Period 1 | ITT |
| 8.1203 | Incidence of Adverse Events by Toxicity Grade and Preferred Term for Period 2 | mITT |
| 8.1204 | Incidence of Treatment Related Adverse Events<br>by Toxicity Grade and Preferred Term for<br>Period 2 | mITT |
| 8.1205 | Incidence of Treatment Related Adverse Events<br>by System Organ Class and Preferred Term for<br>Period 1 | mITT |
| 8.1206 | Incidence of Treatment Related Adverse Events<br>by System Organ Class and Preferred Term for<br>Period 2 | mITT |
| 8.1301 | Incidence of Adverse Events with Toxicity Grade >= 3 by System Organ Class and Preferred Term for Period 1 | ITT |
| 8.1303 | Incidence of Adverse Events with Toxicity Grade >= 3 by System Organ Class and Preferred Term for Period 2 | mITT |
| 8.1305 | Incidence of Treatment Related Adverse Events with Toxicity Grade >=3 by System Organ Class and Preferred Term for Period 1 | mITT |
| 8.1306 | Incidence of Treatment Related Adverse Eventswith Toxicity Grade >= 3 by System Organ Class and Preferred Term for Period 2 | mITT |
| 8.1401 | Incidence of Serious Adverse Events by System Organ Class and Preferred Term for the Pre- leukapheresis Period | ITT |
| 8.1402 | Incidence of Serious Adverse Events by System Organ Class and Preferred Term for Period 1 | ITT |
| 8.1404 | Incidence of Serious Adverse Events by System<br>Organ Class and Preferred Term for Period 2 | mITT |
| 8.1502 | Incidence of Treatment Related Serious Adverse Events by System Organ Class and Preferred Term for Period 1 | mITT |
| 8.1503 | Incidence of Treatment Related Serious Adverse Events by System Organ Class and Preferred Term for Period 2 | mITT |
| 8.1504 | Incidence of Serious Adverse Events by Toxicity Grade and Preferred Term for Period 1 | ITT |
| 8.1505 | Incidence of Serious Adverse Events by Toxicity Grade and Preferred Term for Period 2 | mITT |
| 8.1506 | Incidence of Treatment Related Serious<br>Adverse Events by Toxicity Grade and | mITT |

| Table Number | Table Title | Analysis<br>Population |
|---|---|---|
| | Preferred Term for Period 2 | |
| 8.1601 | Incidence of Serious Adverse Events with Toxicity Grade >=3 by System Organ Class and Preferred Term for the Pre-leukapheresis Period | ITT |
| 8.1602 | Incidence of Serious Adverse Events with Toxicity Grade >=3 by System Organ Class and Preferred Term for Period 1 | ITT |
| 8.1604 | Incidence of Serious Adverse Events with Toxicity Grade >= 3 by System Organ Class and Preferred Term for Period 2 | mITT |
| 8.1606 | Incidence of Treatment Related Serious Adverse Events with Toxicity Grade >=3 by System Organ Class and Preferred Term for the Period 1 | mITT |
| 8.1607 | Incidence of Treatment Related Serious Adverse Events with Toxicity Grade >=3 by System Organ Class and Preferred Term for the Period 2 | mITT |
| 8.1608 | Incidence of Serious Adverse Events Resulting in Death by System Organ Class and Preferred Term for the Pre-leukapheresis Period | ITT |
| 8.2101 | Incidence of Serious Adverse Events Resulting in Death by System Organ Class and Preferred Term for Period 1 | ITT |
| 8.2103 | Incidence of Serious Adverse Events Resulting in Death by System Organ Class and Preferred Term for Period 2 | mITT |
| 8.3001 | Overall Summary of Adverse Events for the Post-lymphodepletion Period for the Second T Cell Infusion | Subjects with a<br>Second T Cell<br>Infusion |
| 8.3002 | Incidence of Adverse Events by System Organ<br>Class and Preferred Term for the Post-<br>lymphodepletion Period for the Second T Cell<br>Infusion | Subjects with a<br>Second T Cell<br>Infusion |
| 8.3003 | Incidence of Adverse Events by Toxicity Grade and Preferred Term for the Post-lymphodepletion Period for the Second T-Cell Infusion | Subjects with a<br>Second T-Cell<br>Infusion |
| 8.3004 | Incidence of Treatment Related Adverse Events<br>by System Organ Class and Preferred Term for<br>the Post- lymphodepletion Period for the<br>Second T-Cell Infusion | Subjects with a<br>Second T-Cell<br>Infusion |
| 8.3005 | Incidence of Serious Adverse Events by System Organ Class and Preferred Term for the Post- | Subjects with a Second T-Cell |

| Table Number | Table Title | Analysis<br>Population |
|---|---|---|
| | lymphodepletion Period for the Second T-Cell Infusion | Infusion |
| 8.3006 | Incidence of Treatment Related Adverse Events<br>by Toxicity Grade and Preferred Term for the<br>Post- lymphodepletion Period for the Second T-<br>Cell Infusion | Subjects with a<br>Second T-Cell<br>Infusion |
| 8.3007 | Incidence of Serious Adverse Events by Toxicity Grade and Preferred Term for the Post- lymphodepletion Period for the Second T- Cell Infusion | Subjects with a<br>Second T-Cell<br>Infusion |
| 8.3008 | Incidence of Treatment Related Serious Adverse Events by Toxicity Grade and Preferred Term for the Post- lymphodepletion Period for the Second T-Cell Infusion | Subjects with a<br>Second T-Cell<br>Infusion |
| 8.3101 | Summary of Adverse Events of Special Interest by Cohort (All Infusions) | mITT |
| 8.3102 | Summary of Adverse Events of Special Interest for the First Infusion | mITT |
| 8.3103 | Summary of Adverse Events of Special Interest<br>by Cohort for the Second Infusion | Subjects with a<br>Second T-Cell<br>Infusion |
| 8.3104 | Summary of Characteristics of Guillain-Barre<br>Syndrome (All Infusions) | mITT |
| 8.3105 | Summary of Characteristics of Graft versus<br>Host Disease (All Infusions) | mITT |
| 8.3106 | Summary of Characteristics of Cytokine<br>Release Syndrome (All Infusions) | mITT |
| 8.3107 | Summary of Characteristics of Recurrent Pancytopenia/Aplastic Anaemia (All Infusions) | mITT |
| 8.3108 | Summary of Characteristics of Encephalopathy (All Infusions) | mITT |
| 8.3109 | Summary of Characterisics of Guillain-Barre<br>Syndrome (Second Infusion) | Subjects with a<br>Second T-Cell<br>Infusion |
| 8.3110 | Summary of Characteristics of Graft versus<br>Host Disease (Second Infusion) | Subjects with a<br>Second T-Cell<br>Infusion |
| 8.3111 | Summary of Characteristics of Cytokine<br>Release Syndrome (Second Infusion) | Subjects with a<br>Second T-Cell<br>Infusion |
| 8.3112 | Summary of Characteristics of Recurrent<br>Pancytopenia/Aplastic Anaemia (Second<br>Infusion) | Subjects with a<br>Second T-Cell<br>Infusion |
| 8.3113 | Summary of Characteristics of Encephalopathy | Subjects with a |
| Table Number | le Number Table Title | |
|---|---|---|
| | (Second Infusion) | Second T-Cell<br>Infusion |
| 8.3114 | Summary of Onset and Duration of the First<br>Occurrence of Guillain-Barre Syndrome | mITT |
| 8.3115 | Summary of Onset and Duration of the First<br>Occurrence of Graft versus Host Disease | mITT |
| 8.3116 | Summary of Onset and Duration of the First<br>Occurrence of Cytokine Release Syndrome | mITT |
| 8.3117 | Summary of Onset and Duration of the First<br>Occurrence of Recurrent Pancytopenia/Aplastic<br>Anaemia | mITT |
| 8.3118 | Summary of Onset and Duration of the Last<br>Occurrence of Encephalopathy | mITT |
| 8.3119 | Summary of Onset and Duration of the Last<br>Occurrence of Guillain-Barre Syndrome | mITT |
| 8.3120 | Summary of Onset and Duration of the Last<br>Occurrence of Graft versus Host Disease | mITT |
| 8.3121 | Summary of Onset and Duration of the Last<br>Occurrence of Cytokine Release Syndrome | mITT |
| 8.3122 | Summary of Onset and Duration of the Last<br>Occurrence of Recurrent Pancytopenia/Aplastic<br>Anaemia | mITT |
| 8.3123 | Summary of Onset and Duration of the Last<br>Occurrence of Encephalopathy | mITT |
| 8.3124 | Summary of Adverse Events of Special Interest by Cohort (Comprehensive List - All Infusions) | mITT |
| 8.3125 | Summary of Adverse Events of Special Interest for the First Infusion (Comprehensive List) | mITT |
| 8.3126 | Summary of Adverse Events of Special Interest<br>by Cohort for the Second Infusion<br>(Comprehensive List) | Subjects with a<br>Second T-Cell<br>Infusion |
| 8.3127 | Summary of Characteristics of Haematopoietic Cytopenias (Comprehensive List-All Infusions) | mITT |
| 8.3128 | Summary of Characteristics of Haematopoietic Cytopenias (Comprehensive List-Second Infusion) | Subjects with a<br>Second T-Cell<br>Infusion |
| 8.3129 | Summary of Onset and Duration of the First<br>Occurrence of Haematopoietic Cytopenias<br>(Comprehensive List) | mITT |
| 8.3201 | Time to Resolution of Grade >= 3 Haematopoietic Cytopenias (Comprehensive List) | mITT |
| 8.3202 | Time to Resolution of Grade >=3 Recurrent Pancytopenia/Aplastic Anaemia | mITT |

| Table Number | Table Title | Analysis<br>Population |
|---|---|---|
| 8.3203 | Time to Resolution of Grade >=3 Graft versus Host Disease | mITT |
| 8.3204 | Time to Resolution of Grade >=3 Cytokine Release Syndrome | mITT |
| 8.4101 | Change from Baseline to Each Scheduled Visit for Hematology Parameters for the Post-lymphodepletion Period | mITT |
| 8.4102 | Change from Baseline to Each Scheduled Visit for Chemistry Parameters for the Post-lymphodepletion Period | mITT |
| 8.4201 | Shifts from Baseline to Worst Post-Baseline NCL-CTCAE Grade for Hematology | |
| 8.4202 | Shifts from Baseline to Worst Post-Baseline<br>NCI-CTCAE Grade for Chemistry Parameters<br>for the Post-lymphodepletion Period | mITT |
| 8.4301 | Number and Proportion of Subjects with<br>Potentially Clinically Significant Hepatic Post-<br>Baseline Results for the Post-lymphodepletion<br>Period | mITT |
| 8.5001 | Maximum Persistence and Time to Maximum Persistence for Responders, Non-responders, and Overall | mITT |
| 8.5002 | Number and Proportion of RCL Positive<br>Subjects | mITT |
| 8.5003 | Number and Percentage of Subjects with<br>Potentially Clinically Significant Post-Baseline<br>Vital Signs Results | mITT |
| 8.6101 | Summary of ECOG Performance Status at Each Visit | mITT |

# 17.2. Data Listings

| Number | Title |
|---|---|
| 26.0001 | Subject Disposition |
| 26.0002 | Study Visits |
| <b>Protocol Deviations</b> | |
| 26.1401 | Inclusion and Exclusion Criteria Not Met Prior to Leukapheresis |
| 26.1403 | Protocol Deviations |

| Number | Title |
|---|---|
| Demographic Data | |
| 26.1101 | Demographics and Baseline Characteristics |
| 26.3101 | Medical History |
| 26.3102 | HLA and NY-ESO Antigen |
| 26.2101 | Disease Characteristics |
| 26.4001 | Prior Cancer Surgery |
| 26.4002 | Prior Oncology Treatment |
| Study Drug Adminis | stration |
| 28.0001 | Dates of Leukapheresis, Lymphodepleting Chemotherapy, and T-Cell Infusion |
| 28.0002 | Lymphodepleting Chemotherapy |
| 28.0003 | T Cell Infusion |
| Individual Efficacy | Response Data |
| 27.0001 | Lesion Measurements and Assessments by RECIST 1.1 |
| 27.0003 | Response Assessments and Overall Response by RECIST v1.1 for the First Infusion |
| 27.0004 | Response Assessments and Overall Response by RECIST v1.1 Following a Second T Cell Infusion |
| 27.0005 | Investigator RECIST v1.1 Response Assessments and Overall Response for the First Infusion |
| 27.00051 | Investigator RECIST v1.1 Response Assessments and Overall Response Following a Second T Cell Infusion |
| 27.0007 | Progression-Free Survival and Overall Survival |
| 27.0008 | Time to Confirmed Response, Duration of Response, and Duration of Stable Disease, and Best Overall Response |
| Adverse Event Listin | ngs |
| 28.1001 | Adverse Events for First T-Cell Infusion |
| 28.1002 | Adverse Events for Second T-Cell Infusion |
| 28.1003 | Adverse Events with CTCAE Grade 3 or Higher |
| 28.2001 | Serious Adverse Events |
| 28.3001 | Cytokine Release Syndrome (CRS) |
| 28.3002 | Graft Versus Host Disease (GVHD) |
| 28.3003 | Recurrent pancytopenia with bone marrow failure/Aplastic anemia |
| 28.3004 | Guillain-Barre syndrome |
| 28.3005 | Encephalopathy syndrome |
| Listings of Individua | al Laboratory Measurements |
| 28.3101 | Hematology Evaluations - Part 1 |
| 28.3111 | Hematology Evaluations - Part 2 |

# 208466/ADP-04511

| Number | Title |
|---|---|
| 28.3121 | Hematology Evaluations - Part 3 |
| 28.3131 | Clinically Significant Hematology Findings |
| 28.3132 | Listing of Subjects with Potentially Clinically Significant Hepatic Post-Baseline Results the Post-lymphodepletion Period |
| 28.3201 | Clinical Chemistry Evaluations - Part 1 |
| 28.3211 | Clinical Chemistry Evaluations – Part 2 |
| 28.3221 | Clinical Chemistry Evaluations – Part 3 |
| 28.3231 | Clinically Significant Clinical Chemistry Findings |
| 28.3301 | Urinalysis Evaluations – Part 1 |
| 28.3311 | Urinalysis Evaluations – Part 2 |
| 28.3321 | Urinalysis Evaluations – Part 3 |
| 28.3331 | Clinically Significant Urinalysis Findings |
| 28.3341 | Additional Laboratory Assessments |
| 28.3342 | Clinically Significant Additional Laboratory Findings |
| 28.3343 | Renal Function Findings |
| 28.4001 | Replication Competent Lentivirus (RCL) |
| 28.4002 | Persistence |
| 28.4101 | Cytokines – Part 1 |
| 28.4102 | Cytokines – Part2 |
| 28.4201 | Biopsy – Tumor Antigen Results |
| 28.4301 | Flow Cytometry |
| 28.5001 | Pregnancy Test Results |
| 28.5101 | Vital Signs |
| 28.5102 | Listing of Subjects with Potentially Clinically Significant Post-<br>Baseline Vital Signs Results |
| 28.5201 | ECOG Performance Status, Karnofsky Score, and Lansky Score |
| 28.6101 | Electrocardiogram |
| 28.6201 | Physical Examination |
| 28.6301 | Concomitant Medications |
| 28.6401 | Bridging Therapies |
| 28.6402 | On-study Surgery |
| 28.6403 | On-study Oncology Treatment |
| 28.6404 | Echocardiogram or Multigated Acquisition Scan (MUGA) |
| 28.6502 | EBV and Anti-CMV Status |
| 28.6503 | Infectious Disease Testing |

# 17.3. Figures

| Number | Figure Title | Analysis<br>Population |
|---|---|---|
| 17.0001 | Maximal Reduction in Sum of Diameters of Target Lesions from Baseline through Progression or Prior to Subsequent Anti-Cancer Therapy for the First Infusion | mITT |
| 17.0002 | Maximal Reduction in Sum of Diameters of Target Lesions from the Second Infusion through Progression or Subsequent Anti-Cancer Therapy | mITT |
| 17.1001 | Kaplan-Meier Plot of Progression-Free Survival | mITT |
| 17.1002 | Kaplan-Meier Plot of Overall Survival | mITT |
| 17.2001 | Response Characteristics via RECIST 1.1 and Follow-up | mITT |
| 17.3001 | Boxplots for Peak Expansion by Responders vs. Non-<br>Responders for the First Infusion | mITT |
| 17.4001 | Spider Plots for Persistence Results over Time (Truncated at 60 Days) for Responders vs. Non-Responders for the First Infusion | mITT |
| 17.4002 | Spider Plots for Persistence Results over Time (Truncated at 100 Days) by Responders vs. Non-Responders for the First Infusion | mITT |
| 17.4003 | Spider Plots for Persistence Results over Time by<br>Responders vs. Non-Responders for the First Infusion | mITT |
| 17.4004 | Spider Plots of Change from Baseline in Target Lesion<br>through Progression and Prior to Subsequent Anti-Cancer<br>Therapy Over Time by Response Status for the First Infusion | mITT |
| 17.4005 | Spider Plots for Persistence Results over Time (Truncated at 60 Days) by Responders vs. Non-Responders for the Second Infusion | mITT |
| 17.4006 | Spider Plots for Persistence Results over Time (Truncated at 100 Days) by Responders vs. Non-Responders for the Second Infusion | mITT |
| 17.4007 | Spider Plots for Persistence Results over Time by<br>Responders vs. Non-Responders for the Second Infusion | mITT |
| 17.4008 | Spider Plots of Change from Baseline in Target Lesion<br>through Progression and Prior to Subsequent Anti-Cancer<br>Therapy Over Time by Response Status for the Second<br>Infusion | mITT |
| 18.5003 | Characteristics of CRS Plot for the First Infusion | mITT |
| 18.5004 | Characteristics of CRS Plot for the Second Infusion | Subjects with<br>a Second T-<br>Cell Infusion |
| 18.5005 | Characteristics of Recurrent Pancytopenia with Bone<br>Marrow Failure/Aplastic Anemia Plot for the First Infusion | mITT |
| 18.5006 | Characteristics of Recurrent Pancytopenia with Bone<br>Marrow Failure/Aplastic Anemia Plot for the Second | Subjects with a Second T- |

# 208466/ADP-04511

| Number | Figure Title | Analysis<br>Population |
|---|---|---|
| | Infusion | Cell Infusion |
| 18.5101 | Profile of INF-Gamma by CRS Status and Subject (First Infusion) | mITT |
| 18.5102 | Profile of IL-6 by CRS Status and Subject (First Infusion) | mITT |
| 18.5103 | Profile of IL-8 by CRS Status and Subject (First Infusion) | mITT |
| 18.5104 | Profile of IL-12 by CRS Status and Subject (First Infusion) | mITT |
| 18.5105 | Profile of IL-13 by CRS Status and Subject (First Infusion) | mITT |
| 18.5106 | Profile of TNF-Alpha by CRS Status and Subject (First Infusion) | mITT |
| 18.5107 | Profile of INF-Gamma by Response and Subject (First Infusion) | mITT |
| 18.5108 | Profile of IL-6 by Response and Subject (First Infusion) | mITT |
| 18.5109 | Profile of IL-8 by Response and Subject (First Infusion) | mITT |
| 18.5110 | Profile of IL-12 by Response and Subject (First Infusion) | mITT |
| 18.5111 | Profile of IL-13 by Response and Subject (First Infusion) | mITT |
| 18.5112 | Profile of TNF-Alpha by Response and Subject (First Infusion) | mITT |
| 18.5113 | Peak Cytokine Expression of INF-Gamma by CRS Status (First Infusion) | mITT |
| 18.5114 | Peak Cytokine Expression of IL-6 by CRS Status (First Infusion) | mITT |
| 18.5115 | Peak Cytokine Expression of IL-8 by CRS Status (First Infusion) | mITT |
| 18.5116 | Peak Cytokine Expression of IL-12 by CRS Status (First Infusion) | mITT |
| 18.5117 | Peak Cytokine Expression of IL-13 by CRS Status (First Infusion) | mITT |
| 18.5118 | Peak Cytokine Expression of TNF-Alpha by CRS Status (First Infusion) | mITT |
| 18.5119 | Peak Cytokine Expression of INF-Gamma by Response (First Infusion) | mITT |
| 18.5120 | Peak Cytokine Expression of IL-6 by Response (First Infusion) | mITT |
| 18.5121 | Peak Cytokine Expression of IL-8 by Response (First Infusion) | mITT |
| 18.5122 | Peak Cytokine Expression of IL-12 by Response (First Infusion) | mITT |
| 18.5123 | Peak Cytokine Expression of IL-13 by Response (First Infusion) | mITT |
| 18.5124 | Peak Cytokine Expression of TNF-Alpha by Response (First Infusion) | mITT |

### 18. APPENDICES

## 18.1. Appendix 1 Safety Laboratory Tests by Category

#### Urinalysis

- Specific gravity
- Urine glucose
- Urine protein
- Urine biliburin
- Urine ketones
- Urine blood
- PH
- Urine leukocytes

#### Hematology

- WBC
- RBC
- Hemaglobin
- Hematocrit
- Platelet count
- Absolute neturophil count
- Absolute lymphocyte count
- Absolute monocyte count
- Absolute eosinophil count
- Reticulocyte count

#### Chemistry

- Creatinine clearance
- BUN
- Creatinine
- Sodium
- Potassium
- Chloride
- CO2
- Calcium
- Magnesium
- Albumin
- Total Bilirubin
- Alkaline Phosphatase
- AST
- ALT
- LDH
- Phosphorus

# 208466/ADP-04511

- Ferritin
- C-reactive protein
- Direct Bilirubin
- Uric Acid
- Amylase
- Lipase

# Coagulation

- PT
- PTT

# Pregnancy Test

- Urine pregnancy test
- serum pregnancy test

#### Additional Lab

- TSH
- T3
- T4

# 18.2. Appendix 2 List of PTs to Be Combined

The following synonyms will be combined under the PT as shown below. The combined term will be used when reporting AE data in tables by PT.

Synonymous terms will be combined regardless of body system.

| Synonym | MedDRA Preferred terms (System Organ Class) |
|---|---|
| Anaemia/Red blood cell count decreased | Anaemia (Blood and lymphatic system disorders) |
| Cytokine Release Syndrome (CRS) | Cytokine Release Syndrome (Immune System Disorders) |
| | Cytokine Storm (Immune System Disorders) |
| Acute GVHD – Skin | Acute graft versus host disease in skin |
| Acute GVHD - Gut (Liver and Intestine) | Acute graft versus host disease in liver Acute graft versus host disease in intestine |
| Acute GVHD - Other (Lung, Bone Marrow, not specified) | Acute graft versus host disease |
| Chronic GVHD - Skin | Chronic graft versus host disease in skin |
| Acute GVHD - Gut (Liver and Intestine) | Acute graft versus host disease in liver |
| | Acute graft versus host disease in intestine |
| Acute GVHD - Other (Lung, Bone Marrow, not specified) | Acute graft versus host disease |
| Chronic GVHD - Skin | Chronic graft versus host disease in skin |
| Chronic GVHD - Gut (Liver and Intestine) | Chronic graft versus host disease in liver |

| Synonym | MedDRA Preferred terms (System Organ<br>Class) |
|---|---|
| | Chronic graft versus host disease in intestine |
| Chronic GVHD Other - (Lung, Bone Marrow, not specified) | Chronic graft versus host disease |
| Unspecified GVHD - Skin | Graft versus host disease in skin |
| Unspecified GVHD - Gut (Liver and Intestine) | Graft versus host disease in liver Graft versus host disease in gastrointestinal tract |
| Unspecified GVHD - Other (Lung, Bone Marrow, not specified) | Graft versus host disease Graft versus host disease in eye Graft versus host disease in lung Prophylaxis against graft versus host disease Transfusion associated graft versus host disease Engraftment syndrome |
| Leukopenia/WBC decreased | White blood cell count decreased (Investigations) Leukopenia (Blood and lymphatic system disorders) |
| Lymphopenia/Lymphocyte count decreased | Lymphopenia (Investigations) Lymphocyte count decreased (Investigations) CD4 lymphocytes decreased (Investigations) CD8 lymphocytes decreased |
| Neutropenia/Neutrophil count decreased | Neutrophil count decreased (Investigations) Neutropenia (Blood and lymphatic system disorders) |

208466/ADP-04511

| Synonym | MedDRA Preferred terms (System Organ<br>Class) |
|---|---|
| Rash/Rash maculo-papular | Rash maculo-papular |
| | Rash |
| | Rash erythematous |
| Thrombocytopenia/Platelet count decreased | Platelet count decreased (Investigations) |
| | Thrombocytopenia (Blood and lymphatic system disorders) |

MedDRA Version 22

The AE listing will not combine these PTs but list them out as they are reported.

# 18.3. Appendix 3 Specification for Collapsing Adverse Event Segments

This section provides the specification for collapsing the segments of adverse events with common preferred term and with either overlapped/or continuous start/end dates into unique adverse events (AEs) based on ADAE ADaM SAS dataset.

# 1. COLLAPSING AE SEGMENTS WITH A COMMON AE PREFERRED TERM (PT) INTO UNIQUE EVENTS BASED ON THE START AND END DATES

For each unique subject, the AE records (segments) with the same AE preferred term will be collapsed into one unique AE event based on the start and end dates below.

# 1.1 Multiple AE Segments with Overlapped or Continuous Start/End Dates

Multiple AE segments with a common preferred term (PT, variable=ADAE.AEDECOD) that occurred around the same time; defined as:

If a segment starts no more than one day (i.e.,  $\leq 1$  day) prior, on, or after the previous segment's end date, it is considered as an 'event'.

If the gap between the start date of a segment and the end date of previous segment is greater than one complete day (i.e., > 1 day), then consider these segments as different events.

If partial start or end dates for any AE segments, then consider these segments as separate events.

### \*\*\* NOTE: Handling of partial dates or completely missing dates

Partial dates or completely missing dates will not be imputed.

The reason for not using imputed dates is due to the small number of partial / or completely missing dates. Furthermore, using imputed dates might create additional error of up to 30 days off for the AE start or AE end dates, and can be up to 60 days off for the duration of AE.

## 1.2 Sort Adverse Events (AE)

For any AE event identified above:

 Sort the AEs segments by study ID (ADAE.STUDYID), unique subject ID (ADAE.USUBJID), AE preferred term (ADAE.AEDECOD), AE start date (ADAE.AESTDTC), and AE end date (ADAE.AEENDTC). The sorting will include all AE segments with complete or partial start / end dates.

#### 1.3 Create Derived Variables in ADAE ADaM SAS Dataset

Based on the ADAE dataset sorted above under Section 1.2, for each unique subject, create the following derived variables in the ADAE ADaM SAS data set:

#### 1) ANL01FL: Flag for the unique AE

#### a) Collapsed AE Segments

For collapsed AE segments. based on the ADAE data set sorted above under Section 1.2:

- o derive the flag variable: <u>ANL01FL="Y" on the first record for each collapsed AE (i.e. the earliest segment within each collapsed AE with the same ADAE.AEDECOD)</u>.
- Otherwise ANL01FL="" (Missing).

#### b) AE Events Comprised of a Single Row (No Collapsing Needed)

derive the flag variable: <u>ANL01FL="Y" for each single segment AE</u> event.

#### 2) EVTSEQ: Sequence number of each unique AE with the same PT

Create a sequence number, EVTSEQ, for each unique AE within the same ADAE.AEDECOD.

For each unique subject within each unique AE preferred term, this variable will be recorded as the sequential number to identify all unique adverse events (including both single segment events (i.e., no collapsing needed) and collapsed events from multiple segments) based on the sorting order chronologically addressed above under Section 1.2.

#### a) Collapsed AE Segments

Each collapsed AE and its corresponding composed segments will have the same sequence numbers (i.e., if multiple segments/records are qualified for being collapsed into one unique AE (i.e, all those records will have same value for the derived variable EVTSEQ for that corresponding subject within the same collapsed AE).

#### b) Single Segment AE Records

Each single segment AE event (i.e., un-collapsed event) will have different unique sequence number separately

#### c) AE Segments with partial start or end dates

Each AE segment with partial start or end dates will have different unique sequence number starting from 99XXX, where

XXX=001, 002, ....

#### \* NOTE:

For those subjects who received 2 T-cell infusions, the sequential number will be based on both infusion periods combined

(i.e., the assigned sequential number will be independent of T-cell infusion periods).

#### - Example:

#### **Original ADAE Dataset:**

| SUBJID | ADECODE | APERIOD | ASTDT | AENDT |
|--------|------------------------------|---------|-------|-------|
| PPD | Cytokine Release<br>Syndrome | 1 | PPD | PPD |
| | Cytokine Release<br>Syndrome | 1 | PPD | PPD |
| | Cytokine Release<br>Syndrome | 1 | PPD | PPD |
| | Cytokine Release<br>Syndrome | 2 | PPD | PPD |

#### **Derived ADAE Dataset:**

| SUBJID | ADECODE | APERIOD | ASTDT | AENDT | ANL01FL | EVTSEQ |
|---|---|---|---|---|---|---|
| PPD | Cytokine<br>Release<br>Syndrome | 1 | PPD | PPD | Y | 1 |
| | Cytokine<br>Release<br>Syndrome | 1 | PPD | PPD | | 1 |
| | Cytokine<br>Release<br>Syndrome | 1 | PPD | PPD | | 1 |
| | Cytokine<br>Release<br>Syndrome | 2 | PPD | PPD | Y | 2 |

#### 3) EVTENDT: End Date for each unique AE

- a) Collapsed AE Segments
  - =ADAE.AENDT (end date) of the last segment of the collapsed
     event (i.e., the segment with the latest ADAE.AENDT within the same collapsed AE for each unique subject)
  - This should be populated on the segment with ANL01FL='Y' only (i.e., the segment with earliest ADAE.ASTDT of each collapsed AE).
  - o Note:

If any of the segments have missing end date (i.e., unresolved) then the derived EVTENDT will be missing, and hence cannot calculate duration of event (please see derived variable: EVTDUR under item 4) below).

b) Single Segment AE Records

=ADAE.AENDT (end date) of each single segment event (i.e. uncollapsed record).

#### 4) EVTDUR: Duration of each unique AE

- a) Collapsed AE Segments
  - Where ANL01FL='Y' then EVTDUR = AESTDT-EVTENDT+1
  - = Missing, if missing end date for the derived variable EVTENDT (i.e., AEOUT=unresolved with missing AEENDTC for any of the segments within the same collapsed AE)

#### b) Single Segment AE records

- EVTDUR = AESTDT-EVTENDT (i.e., = AEENDT) + 1
- = Missing, if missing end date (i.e., missing AEENDT and hence EVTENDT due to AEOUT=unresolved for the corresponding, single segment record (i.e., un-collapsed AE record).

#### 2. ADDITIONAL NOTES

- For any collapsed AEs and single segment records with missing or partial start and/or end dates,
  - EVTDUR= missing and will be excluded from the calculation for the summary statistics of AE duration.
- AOCCPFL: Flag for the first occurrence of preferred term
  - This variable is a GSK standard variable in the ADAE ADaM SAS data set, which can be used to capture the first AE onset date for each unique AE preferred term.

#### 3. DATA EXAMPLES

# 3.1 Case #1: Previous AE End Date is Same as Next AE Start Date

#### **Original ADAE Dataset**

| USUBJID | AEDECO<br>D | ASTD<br>T | AEND<br>T | APERIO<br>D | ATOXGR<br>N | AREL<br>1 | AEOUT | AEACN |
|---|---|---|---|---|---|---|---|---|
| PPD | Cytokine<br>release<br>syndrome | PPD | PPD | 1 | 1 | Y | RECOVERED/RESOLV<br>ED | NOT<br>APPLICABL<br>E |
| | Cytokine<br>release<br>syndrome | PPD | PPD | 1 | 2 | Y | RECOVERED/RESOLV<br>ED | NOT<br>APPLICABL<br>E |
| | Cytokine<br>release<br>syndrome | PPD | PPD | 2 | 2 | N<br>Y | RECOVERED/RESOLV<br>ED | NOT<br>APPLICABL<br>E |
| | Cytokine<br>release<br>syndrome | PPD | PPD | 2 | 3 | Y | RECOVERED/RESOLV<br>ED | NOT<br>APPLICABL<br>E |

In the above example, this subject had 4 CRS records with the first two occurred after the 1<sup>st</sup> T-cell infusion, and the last two occurred after the 2<sup>nd</sup> T-cell infusion. The first two segments can be collapsed into one single CRS event since the 2<sup>nd</sup> segment started on the same date as the end date of the 1<sup>st</sup> segment. Similarly, the 3<sup>rd</sup> and 4<sup>th</sup> segment post the 2<sup>nd</sup> T-cell infusion can be collapsed into one other CRS event due to the same reason.

Below please see the derived variables added into ADAE ADaM SAS dataset.

# **Derived ADAE Dataset**

| USUB<br>JID | AED<br>ECO<br>D | AS<br>TD<br>T | AE<br>ND<br>T | APE<br>RIO<br>D | ATO<br>XGR<br>N | AR<br>EL<br>1 | AEOUT | AEAC<br>N | ANL<br>01FL | EVT<br>SEQ | EVT<br>END<br>T | EVT<br>DUR | AOC<br>CPF<br>L |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PPD | Cytok<br>ine<br>releas<br>e<br>syndr<br>ome | PPD | PPD | 1 | 1 | Y | RECOVERE<br>D/RESOLVE<br>D | NOT<br>APPLI<br>CABL<br>E | Y | i | PPD | 3 | |
| | Cytok<br>ine<br>releas<br>e<br>syndr<br>ome | PPD | PPD | 1 | 2 | Y | RECOVERE<br>D/RESOLVE<br>D | NOT<br>APPLI<br>CABL<br>E | | i | | | |
| | Cytok<br>ine<br>releas<br>e<br>syndr<br>ome | PPD | PPD | 2 | 2 | N | RECOVERE<br>D/RESOLVE<br>D | NOT<br>APPLI<br>CABL<br>E | Y | 2 | PPD | 14 | |
| | Cytok<br>ine<br>releas<br>e<br>syndr<br>ome | PPD | PPD | 2 | 3 | Y | RECOVERE<br>D/RESOLVE<br>D | NOT<br>APPLI<br>CABL<br>E | | 2 | | | |

# 3.2 Case #2: Previous AE Start Date is Same as Next AE Start Date

| Unique<br>Subject<br>Identifier | Dictionary-<br>Derived Term | Sequence<br>Number | Outcome of Adverse<br>Event | Standard<br>Toxicity<br>Grade | Action Taken<br>with Study<br>Treatment | Causality | Start Date/Time<br>of Adverse<br>Event | End Date/Time<br>of Adverse<br>Event | ANL01FL | evtseq | evtendt | evtdur |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PPD | Nausea | 22 | RECOVERED/RESOLVED | 1 | | NOT<br>RELATED | PPD | PPD | Υ | 1 | PPD | 9 |
| PPD | Nausea | 25 | RECOVERED/RESOLVED | 1 | | NOT<br>RELATED | PPD | PPD | | 1 | | |
| PPD | Nausea | 23 | RECOVERED/RESOLVED | 1 | | NOT<br>RELATED | PPD | PPD | Υ | 2 | PPD | 18 |
| PPD | Nausea | 24 | RECOVERED/RESOLVED | 1 | | NOT<br>RELATED | PPD | PPD | | 2 | | |
| PPD | Nausea | 26 | RECOVERED/RESOLVED | 1 | | NOT<br>RELATED | PPD | PPD | | 2 | | |
| PPD | Nausea | 27 | RECOVERED/RESOLVED | 1 | | NOT<br>RELATED | PPD | PPD | | 2 | | |
| PPD | Vomiting | 43 | RECOVERED/RESOLVED | 1 | | NOT<br>RELATED | PPD | PPD | Υ | 1 | PPD_ | 9 |
| PPD | Vomiting | 46 | RECOVERED/RESOLVED | 1 | | NOT<br>RELATED | PPD | PPD | | 1 | | |

# 3.3 Case #3: Next AE Start Date is One Day after Previous AE End Date

| Unique Subject | Dictionary-Derived<br>Term | Sequence<br>Number | Outcome of Adverse Event | Standard<br>Toxicity<br>Grade | Action Taken<br>with Study<br>Treatment | Causality | Start<br>Date/Time<br>of Adverse<br>Event | End<br>Date/Time<br>of Adverse<br>Event | ANL01FL | evtseq | evtendt | evtdur |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PPD | Neutrophil count<br>decreased | 14 | RECOVERED/RESOLVED | 4 | NOT<br>APPLICABLE | NOT<br>RELATED | PPD | PPD | Y | 1 | PPD | 9 |
| PPD | Neutrophil count decreased | 15 | RECOVERED/RESOLVED | 3 | NOT<br>APPLICABLE | NOT<br>RELATED | PPD | PPD | | 1 | | |
| PPD | White blood cell count decreased | 21 | RECOVERED/RESOLVED | 4 | DOSE NOT<br>CHANGED | NOT<br>RELATED | PPD | PPD | Y | 1 | PPD | 16 |
| PPD | White blood cell count decreased | 22 | RECOVERED/RESOLVED | 3 | NOT<br>APPLICABLE | NOT<br>RELATED | PPD | PPD | | 1 | | - |
| PPD | Neutrophil count<br>decreased | 12 | RECOVERED/RESOLVED | 3 | DOSE NOT<br>CHANGED | NOT<br>RELATED | PPD | PPD | Y | 1 | PPD | 6 |
| PPD | Neutrophil count decreased | 13 | RECOVERED/RESOLVED | 4 | DOSE NOT<br>CHANGED | NOT<br>RELATED | PPD | PPD | | 1 | - | - |

# 3.4 Case #4: Previous AE End Date is Greater Than Next AE Start Date.

| Unique Subject<br>Identifier | Dictionary-Derived<br>Term | Sequence<br>Number | Outcome of Adverse<br>Event | Standard<br>Toxicity<br>Grade | Action Taken<br>with Study<br>Treatment | Causality | Start<br>Date/Time of<br>Adverse<br>Event | End<br>Date/Time of<br>Adverse<br>Event | ANL01FL | evtseq | evtendt | evtdur |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PPD | Dyspnoea | 20 | RECOVERED/RESOLVED | 1 | | NOT<br>RELATED | PPD | PPD | Υ | 2 | PPD | 183 |
| PPD | Dyspnoea | 17 | RECOVERED/RESOLVED | 1 | | NOT<br>RELATED | PPD | PPD | | 2 | | |
| PPD | Dyspnoea | 18 | RECOVERED/RESOLVED | 2 | | POSSIBLE | PPD | PPD | | 2 | | |
| PPD | Skin disorder | 60 | RECOVERED/RESOLVED | 1 | | NOT<br>RELATED | PPD | PPD | Υ | 1 | PPD | 8 |
| IPPD | Skin disorder | 58 | RECOVERED/RESOLVED | 1 | | NOT<br>RELATED | PPD | PPD | | 1 | | - |
| PPD | Decreased appetite | 32 | RECOVERED/RESOLVED | 3 | | NOT<br>RELATED | PPD | PPD | Y | 1 | PPD | 52 |
| PPD | Decreased appetite | 34 | RECOVERED/RESOLVED | 3 | | POSSIBLE | PPD | PPD_ | | 1 | | |


Protocol: GSK208466/ADP-04511 Population: Intent-To-Treat (Data as of: 24APR2018)

Table 6.1001

Subject Enrollment and Disposition

ITT Population

| | | | | | Cohort 2-4 | |
|---|---|---|---|---|---|---|
| | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total | Overall |
| ITT Population | XX | XX | XX | XX | XX | XX |
| MITT Population | xx | xx | XX | XX | XX | xx |
| Lymphodepleted | xx | xx | xx | XX | xx | XX |
| Subject Status at the End of the First Infusion | | | | | | |
| Disease progression | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Unacceptable toxicity and other safety reasons | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| death | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| INVESTIGATOR DISCRETION | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| subject withdrew consent | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| protocol violation | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| lost to follow-up | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| termination by sponsor | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| failed manufacture of cell product | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| pregnancy | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| FAILED TO MEET ELIGIBILITY CRITERIA FOR THE SECOND INFUSION | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

ITT = Intent-to-treat, mITT = Modified ITT.

ITT Population = all subjects who were enrolled in the trial (i.e., underwent leukapheresis).

MITT Population = all subjects in the ITT population who received at least one T cell infusion.

Note 1: Denominator for percentages is based on the ITT Population.

Note 2: Subjects who have disease progression are considered to have completed the interventional phase.

Note 3: If withdrawn less than or equal to 60 days since the first infusion, the subject cannot be re-enrolled into the  $2^{nd}$  infusion and only required to provide the status at the end of the study.

File Name: S:\.....\&prog name

#### 208466/ADP-04511


(Data as of: 24APR2018)

Protocol: GSK208466/ADP-04511 Population: Intent-To-Treat

Table 6.1001

Subject Enrollment and Disposition

ITT Population

| | | | | | Cohort 2-4 | |
|---|---|---|---|---|---|---|
| | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total | Overall |
| Subject Status at the End of the Study | | | | | | |
| Disease progression | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Unacceptable toxicity and other safety reasons | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| death | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| INVESTIGATOR DISCRETION | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| subject withdrew consent | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| protocol violation | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| lost to follow-up | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| termination by sponsor | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| failed manufacture of cell product | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| pregnancy | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| FAILED TO MEET ELIGIBILITY CRITERIA FOR THE SECOND INFUSION | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

ITT = Intent-to-treat, mITT = Modified ITT.

ITT Population = all subjects who were enrolled in the trial (i.e., underwent leukapheresis).

MITT Population = all subjects in the ITT population who received at least one T cell infusion.

Note 1: Denominator for percentages is based on the ITT Population.

Note 2: Subjects who have disease progression are considered to have completed the interventional phase.

Note 3: If withdrawn less than or equal to 60 days since the first infusion, the subject cannot be re-enrolled into the 2nd infusion and only required to provide the status at the end of the study.

File Name: S:\.....\&prog name

#### 208466/ADP-04511

Page 1 of 3 (Data as of: 24APR2018)

Protocol: GSK208466/ADP-04511 Population: Intent-To-Treat

Table 6.2001

Demographic and Baseline Characteristics

ITT Population

| Sex | Parameter | Category | Statistic | Cohort 1 (N=xx) | Cohort 2<br>(N=xx) | Cohort 3<br>(N=xx) | Cohort 4<br>(N=xx) | Cohort 2-4<br>Total<br>(N=xx) | Overall (N=xx) |
|---|---|---|---|---|---|---|---|---|---|
| MALE | Sex | FEMAI.E | n (%) | x (xx x%) | x (xx x%) | x (xx x%) | x (xx x%) | x (xx x%) | x (xx x%) |
| Mean | DCA | | | | , , | | , , | | |
| Mean | Age (vears) | | N | Х | Х | Х | Х | Х | Х |
| Median Min, Max Min, Min, Max Min, Min, Max Min, Min, Max Min, Ma | 2 (4 / | | | | | | | | |
| Min, Max xx, xx | | | SD | | XX.XX | | | | |
| Race | | | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| AMERICAN INDIAN OR ALASKA N(%) x (xx.x%) x (xx | | | Min,Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| NATIVE ASIAN | Race | BLACK OR AFRICAN AMERICAN | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| NATIVE HAWAIIAN OR OTHER n(%) x (xx.x%) x (xx. | | | n(%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| PACIFIC ISLANDER WHITE | | ASIAN | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| OTHER n(%) x (xx.x%) x (xx.x | | | n(%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| DTHER N(%) X (XX.X%) X | | WHITE | n(%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| NOT HISPANIC OR LATINO n(%) x (xx.x%) x (xx.xx) x (xx.xx) x (xx.xx) x (xx.xx) | | OTHER | | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Screening N x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x | Ethnicity | HISPANIC OR LATINO | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Height (cm) N x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x <th< td=""><td>_</td><td>NOT HISPANIC OR LATINO</td><td>n(%)</td><td>x (xx.x%)</td><td>x (xx.x%)</td><td>x (xx.x%)</td><td>x (xx.x%)</td><td>x (xx.x%)</td><td>x (xx.x%)</td></th<> | _ | NOT HISPANIC OR LATINO | n(%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Height (cm) N x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x x <th< td=""><td>Screening</td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td></th<> | Screening | | | | | | | | |
| SD xx.xxx | _ | | N | Х | X | Х | X | Х | Х |
| Median xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx xx.xx | | | Mean | XX.XX | XX.XX | xx.xx | XX.XX | XX.XX | xx.xx |
| | | | SD | XX.XXX | XX.XXX | xx.xxx | XX.XXX | XX.XXX | XX.XXX |
| Min, Max xx.x, xx.x xx.x, xx.x xx.x, xx.x xx.x | | | Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | xx.xx |
| | | | Min,Max | xx.x,xx.x | xx.x,xx.x | xx.x, xx.x | xx.x,xx.x | xx.x,xx.x | xx.x,xx.x |

BMI = Body Mass Index, BSA = Body Surface Area, ECOG = Eastern Cooperative Oncology Group, SD = Standard Deviation.

Note 1: Age is the age at informed consent, baseline weight is within 7 days prior to lymnphodepletion, and BMI is calculated using the baseline weight and the height at the Screening visit.

Note 2: ECOG Score: 0 - Fully active and able to carry on all pre-disease activities without restriction, 1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light sedentary nature, 2 - Ambulatory and capable of all self-care but unable to carry out any work activities, 3 - Capable of only limited self-care, 4 - Completely disabled, 5 - Dead. Subjects had to have an ECOG score of 0 or 1 to be enrolled in the study.

File Name: S:\.....\&prog name

Protocol: GSK208466/ADP-04511 Population: Intent-To-Treat Page 2 (Data as of: 24APR2018)

Table 6.2001

Demographic and Baseline Characteristics

ITT Population

| Parameter | Category | Statistic | Cohort 1 (N=xx) | Cohort 2<br>(N=xx) | Cohort 3 (N=xx) | Cohort 4<br>(N=xx) | Cohort 2-4<br>Total<br>(N=xx) | Overall<br>(N=xx) |
|---|---|---|---|---|---|---|---|---|
| Weight (kg) | | N | х | х | х | х | x | X |
| weight (kg) | | Mean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | SD | | | XX.XXX | | | XX.XXX |
| | | Median | XX.XXX | xx.xxx | | xx.xxx | XX.XXX | |
| | | | XX.XX | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX |
| | | Min,Max | xx.x, xx.x | xx.x, xx.x | xx.x,xx.x | xx.x,xx.x | xx.x, xx.x | XX.X,XX.X |
| BMI(kg/m^2) | | N | х | Х | X | X | X | X |
| | | Mean | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | xx.xx |
| | | SD | xx.xxx | xx.xxx | XX.XXX | XX.XXX | XX.XXX | xx.xxx |
| | | Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | xx.xx |
| | | Min,Max | xx.x,xx.x | xx.x,xx.x | xx.x, xx.x | xx.x, xx.x | XX.X,XX.X | xx.x,xx.x |
| BSA (m^2) | | N | Х | X | X | X | X | X |
| | | Mean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | SD | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | xx.xxx |
| | | Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | xx.xx |
| | | Min,Max | xx.x, xx.x | xx.x,xx.x | xx.x,xx.x | xx.x,xx.x | xx.x, xx.x | xx.x, xx.x |
| HLA Status | HLA-A*0201 | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | HLA-A*0205 | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | HLA-A*0206 | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | Other | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| NY-ESO Status | Positive High | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | Positive Low | n (응) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | Negative | n (응) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | Not Evaluable | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |

BMI = Body Mass Index, BSA = Body Surface Area, ECOG = Eastern Cooperative Oncology Group, SD = Standard Deviation.

Note 1: Age is the age at informed consent, baseline weight is within 7 days prior to T-cell infusion, and BMI is calculated using the baseline weight and the height at the Screening visit.

Note 2: ECOG Score: 0 - Fully active and able to carry on all pre-disease activities without restriction, 1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light sedentary nature, 2 - Ambulatory and capable of all self-care but unable to carry out any work activities, 3 - Capable of only limited self-care, 4 - Completely disabled, 5 - Dead. Subjects had to have an ECOG score of 0 or 1 to be enrolled in the study. File Name: S:\.....\&prog name

(Data as of: 24APR2018)

Protocol: GSK208466/ADP-04511

Page 3 of 3 Population: Intent-To-Treat

Table 6.2001

Demographic and Baseline Characteristics

ITT Population

| Parameter | Category | Statistic | Cohort 1 (N=xx) | Cohort 2<br>(N=xx) | Cohort 3 (N=xx) | Cohort 4 (N=xx) | Cohort 2-4<br>Total<br>(N=xx) | Overall (N=xx) |
|---|---|---|---|---|---|---|---|---|
| Disease Stage at<br>Enrollment | Stage I<br>Stage II<br>Stage III | n(%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | Stage IV | n(%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | OTHER<br>MISSING | n(%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Type of Histology | MONOPHASIC | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | BIPHASIC | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | OTHER | n(%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Screening ECOG Performance | 2 | | | | | | | |
| Status | 0 | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | 1 | n(%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |

BMI = Body Mass Index, BSA = Body Surface Area, ECOG = Eastern Cooperative Oncology Group, SD = Standard Deviation.

Note 1: Age is the age at informed consent, baseline weight is within 7 days prior to T-cell infusion, and BMI is calculated using the baseline weight and the height at the Screening visit.

Note 2: ECOG Score: 0 - Fully active and able to carry on all pre-disease activities without restriction, 1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light sedentary nature, 2 - Ambulatory and capable of all self-care but unable to carry out any work activities, 3 -Capable of only limited self-care, 4 - Completely disabled, 5 - Dead. Subjects had to have an ECOG score of 0 or 1 to be enrolled in the study. File Name: S:\.....\&prog name

208466/ADP-04511

Repeat 6.2001 format for:

Table 6.2002 Demographic and Baseline Characteristics mITT Population

Note: mITT tables will be provided only if mITT and ITT populations differ.

Protocol: GSK208466/ADP-04511 Population: Intent-To-Treat 
 (Data as of: 24APR2018)

Table 6.3001

Summary of Medical History

ITT Population

| System Organ Class/<br>Preferred Term | Cohort 1<br>(N=xx) | Cohort 2<br>(N=xx) | Cohort 3<br>(N=xx) | Cohort 4<br>(N=xx) | Cohort 2-4<br>Total<br>(N=xx) | Overall<br>(N=xx) |
|---|---|---|---|---|---|---|
| Any Medical History | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| SOC 1 | | | | | | |
| Preferred Term 1 | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Preferred Term 2 | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Etc. | | | | | | |
| SOC 2 | | | | | | |
| Preferred Term 1 | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Preferred Term 2 | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Etc. | | | | | | |

Etc.

File Name: S:\.....\&prog\_name

Programming note: sort by descending overall SOC and descending overall PT.

(Data as of: 24APR2018)

Protocol: GSK208466/ADP-04511

 Population: Intent-To-Treat

Table 6.4001

Summary of Prior Cancer Therapy

ITT Population

| | | | | | | Cohort 2-4 | |
|---|---|---|---|---|---|---|---|
| Characteristic/ | | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total | Overall |
| Category | Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Prior Systemic Therapy | | | | | | | |
| YES | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| NO | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Number of Prior Systemic<br>Therapy Regimens | | | | | | | |
| 1 | n(%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| 2 | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Etc. | , , | , , | , , | , , | , , | , , | , , |
| Type of Systemic Therapy \$ | | | | | | | |
| CHEMOTHERAPY | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| IMMUNOTHERAPY | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| HORMONAL | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| VACCINE | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| OTHER | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| OTHER | 11 ( 0 ) | A (AA.A0) | A (AA.A0) | A (AA.A0) | A (AA.A0) | A (AA.A0) | A (AA.A0) |
| Time Since Last Systemic | | | | | | | |
| Therapy (Days) @ | n | X | X | X | Х | X | X |
| | Mean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | xx.xx |
| | SD | xx.xxx | xx.xxx | xx.xxx | xx.xxx | xx.xxx | xx.xxx |
| | Median | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | XX.XX |
| | Min,Max | xx.x,xx.x | xx.x,xx.x | xx.x,xx.x | xx.x,xx.x | xx.x,xx.x | xx.x,xx.x |
| Best Response to Last Syste<br>Therapy | emic | | | | | | |
| COMPLETE RESPONSE | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| PARTIAL RESPONSE | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| STABLE DISEASE | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| DISEASE PROGRESSION | n(%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| UNKNOWN | n (%) | x (xx.x%)<br>x (xx.x%) | x (xx.x%)<br>x (xx.x%) | x (xx.x%)<br>x (xx.x%) | x (xx.x%)<br>x (xx.x%) | x (xx.x%)<br>x (xx.x%) | x (xx.x%)<br>x (xx.x%) |
| NOT DONE | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |

<sup>\$</sup> A subject may have more than one response.

<sup>@</sup> Time Since Last Systemic Therapy is calculated as the date the informed consent was signed minus the latest therapy end date. Time Since Initial Diagnosis is calculated as the date the informed consent was signed minus the date of initial diagnosis.

<sup>#</sup> Bridging therapy is therapy administered on or after apheresis and before lymphodepletion.

File Name: S:\.....\&prog name

(Data as of: 24APR2018)

Protocol: GSK208466/ADP-04511 

Population: Intent-To-Treat

Table 6.4001

Summary of Prior Cancer Therapy

ITT Population

| | | | | | | Cohort 2-4 | |
|---|---|---|---|---|---|---|---|
| Characteristic/ | | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total | Overall |
| Category | Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Prior Radiotherapy | | | | | | | |
| YES | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| NO | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| D ' 0 D 1 + 10 | | | | | | | |
| Prior Cancer-Related Surge | - | | | | | | , , , , |
| YES | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| NO | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Bridging Therapy # | | | | | | | |
| YES | n(%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| NO | n(%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Type of Bridging Therapy # | # | | | | | | |
| CHEMOTHERAPY | n(%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| RADIATION | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| OTHER | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Time Since Initial | | | | | | | |
| Diagnosis(Days) @ | n | X | X | X | X | X | X |
| | Mean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | SD | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| | Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x,xx.x | xx.x, xx.x | xx.x, xx.x | xx.x,xx.x |

<sup>\$</sup> A subject may have more than one response.

<sup>@</sup> Time Since Last Systemic Therapy is calculated as the date the informed consent was signed minus the latest therapy end date. Time Since Initial Diagnosis is calculated as the date the informed consent was signed minus the date of initial diagnosis.

<sup>#</sup> Bridging therapy is therapy administered on or after apheresis and before lymphodepletion.

File Name: S:\.....\&prog name

208466/ADP-04511
Repeat 6.4001 format for:

Table 6.4002 Summary of Prior Cancer Therapy mITT Population Protocol: GSK208466/ADP-04511
Population: Modified Intent-To-Treat 
(Data as of: 24APR2018)

Table 7.1001

Summary of Overall Response Rate and Best Overall Response for the First Infusion

mITT Population

| Parameter/<br>Category or Criterion | Statistic | Cohort 1 (N=xx) | Cohort 2<br>(N=xx) | Cohort 3 (N=xx) | Cohort 4 (N=xx) |
|---|---|---|---|---|---|
| Overall Response Rate (ORR) \$ | | | | | |
| Derived Response derived based on RECIST V1.1 | n (%)<br>95% Clopper Pearson<br>CI<br>95% Wilson CI | x (xx.x%)<br>(xx.x, xx.x)<br>(xx.x, xx.x) | x (xx.x%)<br>(xx.x, xx.x)<br>(xx.x, xx.x) | x (xx.x%)<br>(xx.x, xx.x)<br>(xx.x, xx.x) | x (xx.x%)<br>(xx.x,<br>xx.x)<br>(xx.x,<br>xx.x) |
| Investigator-assessed based on RECIST V1.1 | n (%)<br>95% CI | x (xx.x%)<br>(xx.x, xx.x) | x (xx.x%)<br>(xx.x, xx.x) | x (xx.x%)<br>(xx.x, xx.x) | x (xx.x%)<br>(xx.x,<br>xx.x) |
| Best Overall Response<br>(BOR) derived based on<br>RECIST V1.1 & | | | | | |
| Complete Response | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Partial Response | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Stable Disease | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Progressive<br>Disease | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Unknown or Missing | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |

BOR = Best Overall Response, CI = Confidence Interval, ORR = Overall Response Rate.

<sup>\$</sup> Overall response rate is defined as the proportion of subjects with a confirmed complete response or partial response relative to the total number of subjects in the population.

<sup>&</sup>amp; Best overall response is the best response recorded from the time of first T cell infusion until disease progression, use of prohibited medications, or surgical resection. If unconfirmed complete or partial response, then the best overall response is stable disease.

Note 1: Subject PPD had a day 3 assessment of PD that is not included in this summary because assessments prior to week 4 were not used in determination of PD. Note 2: In cohort 2 subject PPD's derived BOR based on RECIST 1.1 is SD but PD per investigator-assessed.

File Name: S:\.....\&prog name

208466/ADP-04511

#### Repeat Table 7.1001 template for:

Table 7.1002 Summary of Overall Response Rate and Best Overall Response for the Second Infusion Subjects Who Received Second Infusion Protocol: GSK208466/ADP-04511

 Population: Modified Intent-To-Treat (Data as of: 24APR2018)

Table 7.2001

Time in Study, Time to Response, Duration of Response, and Kaplan-Meier Estimate of Duration of Stable Disease mITT Population

| Parameter/<br>Category | Statistic | Cohort 1<br>(N=xx) | Cohort 2<br>(N=xx) | Cohort 3<br>(N=xx) | Cohort 4<br>(N=xx) |
|---|---|---|---|---|---|
| category | Statistic | (N-XX) | (N-XX) | (IV-XX) | (IV-XX) |
| Cime to Response<br>(weeks)& | n | Х | x | х | x |
| | Mean | X.X | X.X | x.x | x.x |
| | SD | X.XX | x.xx | x.xx | X.XX |
| | Median | X.X | X.X | x.x | x.x |
| | Min, Max | х, х | х, х | x, x | x, x |
| Ouration of Response<br>(weeks) @ | n | х | х | х | х |
| | Mean | X.X | X.X | X • X | X . X |
| | SD | X.XX | x.xx | X.XX | X.XX |
| | Median | X • X | X.X | X • X | x.x |
| | Min, Max | x, x | x, x | x, x | x, x |

CI = Confidence interval, DOR = Duration of Response, TTR = Time to Response, DOSD = Duration of Stable Disease, Q1=25th percentile, Q3=75th percentile, CR = Complete Response, PR = Confirmed Response, PD = Progressive Disease.

Note: Quartiles and 95% CI are from Kaplan-Meier estimate. CIs are from complementary log-log transformation.

<sup>&</sup>amp; TTR is defined as the interval between the date of first T cell infusion and the earliest date of confirmed complete response (CR) or partial response (PR), and is summarized for those subjects with a confirmed CR or PR.

<sup>@</sup> DOR is defined as the time from first documented confirmed CR or PR until first documented disease progression or death due to any cause or surgical resection or start of prohibited medications from any cause. For responders without these events, date of the last study assessment is used.

<sup>#</sup> DOSD is defined as the interval between the date of first T cell infusion and the first documented disease progression. Subjects who do not have documented disease progression are censored at the date of last disease assessment.

File Name: S:\.....\&prog name

Protocol: GSK208466/ADP-04511
Population: Modified Intent-To-Treat (Data as of: 24APR2018)

Table 7.2001

Time in Study, Time to Response, Duration of Response, and Kaplan-Meier Estimate of Duration of Stable Disease mITT Population

| Parameter/ | | | | | |
|---|---|---|---|---|---|
| | | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 |
| Category | Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Duration of Stable<br>Disease (DOSD) # | | | | | |
| Subjects with Event | n (응) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Number Censored | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Duration of Stable<br>Disease (weeks) | N | X | Х | X | Х |
| | Q1 (95% CI) | xx.x ( $xx.x$ , $xx.x$ ) | xx.x ( $xx.x$ , $xx.x$ ) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Median<br>(95% CI) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Q3 (95% CI) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| Time in Study(Days) | | | | | |
| | n | х | Х | Х | х |
| | Mean | XX.XX | XX.XX | XX.XX | XX.XX |
| | SD | xx.xxx | xx.xxx | xx.xxx | xx.xxx |
| | Median | xx.xx | xx.xx | xx.xx | xx.xx |
| | Min,Max | xx.x,xx.x | xx.x,xx.x | xx.x,xx.x | xx.x,xx.x |

CI = Confidence interval, DOR = Duration of Response, TTR = Time to Response, DOSD = Duration of Stable Disease, Q1= $25^{th}$  percentile, Q3= $75^{th}$  percentile, CR = Complete Response, PR = Confirmed Response, PD = Progressive Disease.

File Name: S:\.....\&prog name

Note: Quartiles and 95% CI are from Kaplan-Meier estimate. CIs are from complementary log-log transformation.

<sup>&</sup>amp; TTR is defined as the interval between the date of first T cell infusion and the earliest date of confirmed complete response (CR) or partial response (PR), and is summarized for those subjects with a confirmed CR or PR.

<sup>@</sup> DOR is defined as the time from first documented confirmed CR or PR until first documented disease progression or death due to any cause or surgical resection or start of prohibited medications from any cause. For responders without these events, date of the last study assessment is used.

<sup>#</sup> DOSD is defined as the interval between the date of first T cell infusion and the first documented disease progression. Subjects who do not have documented disease progression are censored at the date of last disease assessment.

 (Data as of: 24APR2018)

Protocol: GSK208466/ADP-04511

Population: Modified Intent-To-Treat

Table 7.2002
Kaplan-Meier Estimate of Progression-Free Survival and Overall Survival mITT Population

| Parameter/ | | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 |
|---|---|---|---|---|---|
| Category | Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Progression-Free<br>Survival (PFS) & | | | | | |
| Subjects with Event | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Number Censored | n (응) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| PFS (weeks) | N<br>Q1 (95%<br>CI)<br>Median<br>(95% CI) | X<br>xx.x (xx.x, xx.x)<br>xx.x (xx.x, xx.x) | X xx.x (xx.x, xx.x) xx.x (xx.x, xx.x) | X xx.x (xx.x, xx.x) xx.x (xx.x, xx.x) | X<br>xx.x (xx.x, xx.x)<br>xx.x (xx.x, xx.x) |
| | Q3 (95%<br>CI) | xx.x (xx.x, xx.x) | xx.x (xx.x,<br>xx.x) | xx.x (xx.x,<br>xx.x) | xx.x (xx.x, xx.x) |
| Reason for PD/Death<br>Increased Tumor Burden<br>Death<br>Surgical Resection<br>Prohibited Medication | n (%) n (%) n (%) n (%) | x (xx.x%)<br>x (xx.x%)<br>x (xx.x%)<br>x (xx.x%) | x (xx.x%)<br>x (xx.x%)<br>x (xx.x%)<br>x (xx.x%) | x (xx.x%)<br>x (xx.x%)<br>x (xx.x%)<br>x (xx.x%) | x (xx.x%)<br>x (xx.x%)<br>x (xx.x%)<br>x (xx.x%) |
| Overall Survival (OS) @<br>Subjects with Event<br>Number Censored | n (%)<br>n (%) | x (xx.x%)<br>x (xx.x%) | x (xx.x%)<br>x (xx.x%) | x (xx.x%)<br>x (xx.x%) | x (xx.x%)<br>x (xx.x%) |
| OS (weeks) | N<br>Q1 (95%<br>CI)<br>Median<br>(95% CI)<br>Q3 (95% | X xx.x (xx.x, xx.x) xx.x (xx.x, xx.x) xx.x (xx.x, xx.x) | X xx.x (xx.x, xx.x) xx.x (xx.x, xx.x) xx.x (xx.x, | X xx.x (xx.x, xx.x) xx.x (xx.x, xx.x) xx.x (xx.x, xx.x) | X<br>xx.x (xx.x, xx.x)<br>xx.x (xx.x, xx.x)<br>xx.x (xx.x, |
| | CI) | | xx.x) | | xx.x) |

CI = Confidence interval, OS = Overall Survival, PFS = Progression-Free Survival, Q1=25<sup>th</sup> percentile, Q3=75<sup>th</sup> percentile.

Note: Quartiles and 95% CI are from Kaplan-Meier estimate. CIs are from complementary log-log transformation.

<sup>&</sup>amp; PFS is defined as the interval between the date of first T cell infusion and first documented disease progression or death due to any cause or surgical resection or start of prohibited medication. Subjects without any of the aforementioned events are censored at the date of last adequate assessment.

208466/ADP-04511

@ OS is defined as the interval between the date of first T cell infusion and date of death due to any cause. Subjects who are still alive or lost to follow-up are censored at the date of last contact.

File Name: S:\.....\&prog name

Note to programmer: Denominator for each reason is number fo subjects with event.

 (Data as of: 24APR2018)

Protocol: GSK208466/ADP-04511
Population: Modified Intent-To-Treat (

Table 7.2101

Sensitivity Analyses for Best Overall Response for the First Infusion

mITT Population

| Sensitivity Analysis/<br>Response Category | Statistic | Cohort 1<br>(N=xx) | Cohort 2<br>(N=xx) | Cohort 3<br>(N=xx) | Cohort 4<br>(N=xx) |
|---|---|---|---|---|---|
| Progressive Disease | | | | | |
| Based on Last Tumor<br>Assessment \$ | | | | | |
| Complete Response | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Partial Response | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Stable Disease | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Progressive<br>Disease | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Unknown or Missing | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Investigator Assessment of Response | | | | | |
| Complete Response | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Partial Response | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Stable Disease | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Progressive<br>Disease | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Unknown or Missing | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |

BOR = Best Overall Response, CR = Complete Response, PR = Partial Response, SD = Stable Disease, PD = Progressive Disease, NE = Not Evaluable (Unknown or Missing), N/A = Not Applicable.

Note: Best overall response is the best response recorded from the time of first T cell infusion until disease progression, use of prohibited medications, or surgical resection, whichever came first, except as noted in \$ footnote.

Note: Subject PPD had a day 3 assessment of PD that is not included in this summary because assessments prior to week 4 were not used in determination of PD.

File Name: S:\.....\&prog name

<sup>\$</sup> Date of last assessment is used as date of progressive disease in place of start date of prohibited medications or surgical resection.

<sup>@</sup> Assign values of SD if the assessments before and after the NE assessment are CR, PR, or SD. Assign PD otherwise, except for PR NE CR where the assessment is improving.
Protocol: GSK208466/ADP-04511

Population: Modified Intent-To-Treat

 (Data as of: 24APR2018)

Table 7.2101

Sensitivity Analyses for Best Overall Response for the First Infusion

mITT Population

| Sensitivity Analysis/<br>Response Category | Statistic | Cohort 1 (N=xx) | Cohort 2<br>(N=xx) | Cohort 3<br>(N=xx) | Cohort 4<br>(N=xx) |
|---|---|---|---|---|---|
| Replace NE with SD | | | | | |
| or PD @ | | | | | |
| Complete Response | n (%) | N/A | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Partial Response | n (%) | N/A | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Stable Disease | n (%) | N/A | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Progressive | n (%) | N/A | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Disease | n (2) | N / A | v (vv v <sup>2</sup> ) | v (vv v2) | v (vv v?) |
| Unknown or Missing | n (%) | N/A | x (xx.x%) | x (xx.x%) | x (xx.x%) |

BOR = Best Overall Response, CR = Complete Response, PR = Partial Response, SD = Stable Disease, PD = Progressive Disease, NE = Not Evaluable (Unknown or Missing), N/A = Not Applicable.

Note: Best overall response is the best response recorded from the time of first T cell infusion until disease progression, use of prohibited medications, or surgical resection, whichever came first, except as noted in \$ footnote.

Note: Subject PPD had a day 3 assessment of PD that is not included in this summary because assessments prior to week 4 were not used in determination of PD.

File Name: S:\.... \&prog name

<sup>\$</sup> Date of last assessment is used as date of progressive disease in place of start date of prohibited medications or surgical resection.

<sup>@</sup> Assign values of SD if the assessments before and after the NE assessment are CR, PR, or SD. Assign PD otherwise, except for PR NE CR where the assessment is improving.


(Data as of: 24APR2018)

Protocol: GSK208466/ADP-04511

Population: Modified Intent-To-Treat

Table 7.2103

Sensitivity Analyses for Progression-Free Survival

mITT Population

| Sensitivity Analysis/<br>Response Category | Statistic | Cohort 1 (N=xx) | Cohort 2<br>(N=xx) | Cohort 3<br>(N=xx) | Cohort 4<br>(N=xx) |
|---|---|---|---|---|---|
| Progressive Disease | | | | | |
| Based on Last Tumor | | | | | |
| Assessment \$ | | | | | |
| Subjects with Event | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Number Censored | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Progression-Free | | | | | |
| Survival(weeks) | N | X | X | X | X |
| | Q1 (95% CI) | xx.x (xx.x, xx.x) | xx.x ( $xx.x$ , $xx.x$ ) | xx.x ( $xx.x$ , $xx.x$ ) | xx.x ( $xx.x$ , $xx.x$ ) |
| | Median<br>(95% CI) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Q3 (95% CI) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x ( $xx.x$ , $xx.x$ ) | xx.x (xx.x, xx.x) |

CR = Complete Response, PR = Partial Response, SD = Stable Disease, PD = Progressive Disease, NE = Not Evaluable (Unknown or Missing).

File Name: S:\.....\&prog name

<sup>&</sup>amp; PFS is defined as the interval between the date of first T cell infusion and first disease progression, death due to any cause, surgical resection, or start of prohibited medication, except as noted in \$ footnote. Subjects without any of the aforementioned events are censored at the date of last study assessment. \$ Subjects are censored at first surgical resection or start of prohibited medications, whichever came first.

<sup>@</sup> Assign values of SD if the assessments before and after the NE assessment are CR, PR, or SD. Assign PD otherwise, except for PR NE CR where the assessment is improving.

<sup>^</sup> Subjects who discontinued for disease progression but did not meet RECIST criteria for PD are classified as PD at the date of discontinuation.


(Data as of: 24APR2018)

Protocol: GSK208466/ADP-04511

Population: Modified Intent-To-Treat

Table 7.2103

Sensitivity Analyses for Progression-Free Survival

mITT Population

| Sensitivity Analysis/<br>Response Category | Statistic | Cohort 1 (N=xx) | Cohort 2<br>(N=xx) | Cohort 3<br>(N=xx) | Cohort 4<br>(N=xx) |
|---|---|---|---|---|---|
| Investigator Assessment of | | | | | |
| Response | | | | | |
| Subjects with Event | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Number Censored | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Progression-Free | | | | | |
| Survival(weeks) | N | X | X | X | X |
| | Q1 (95% CI) | xx.x ( $xx.x$ , $xx.x$ ) | xx.x ( $xx.x$ , $xx.x$ ) | xx.x ( $xx.x$ , $xx.x$ ) | xx.x ( $xx.x$ , $xx.x$ ) |
| | Median | xx.x ( $xx.x$ , $xx.x$ ) | xx.x ( $xx.x$ , $xx.x$ ) | xx.x (xx.x, xx.x) | xx.x ( $xx.x$ , $xx.x$ ) |
| | (95% CI) | | | | |
| | Q3 (95% CI) | xx.x ( $xx.x$ , $xx.x$ ) | xx.x ( $xx.x$ , $xx.x$ ) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| Ignore Assessments of NE | | | | | |
| Subjects with Event | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Number Censored | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Progression-Free | | | | | |
| Survival(weeks) | N | X | X | X | X |
| | Q1 (95% CI) | xx.x ( $xx.x$ , $xx.x$ ) | xx.x ( $xx.x$ , $xx.x$ ) | xx.x (xx.x, xx.x) | xx.x ( $xx.x$ , $xx.x$ ) |
| | Median<br>(95% CI) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Q3 (95% CI) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |

CR = Complete Response, PR = Partial Response, SD = Stable Disease, PD = Progressive Disease, NE = Not Evaluable (Unknown or Missing).

<sup>&</sup>amp; PFS is defined as the interval between the date of first T cell infusion and first disease progression, death due to any cause, surgical resection, or start of prohibited medication, except as noted in \$ footnote. Subjects without any of the aforementioned events are censored at the date of last study assessment. \$ Subjects are censored at first surgical resection or start of prohibited medications, whichever came first.

<sup>@</sup> Assign values of SD if the assessments before and after the NE assessment are CR, PR, or SD. Assign PD otherwise, except for PR NE CR where the assessment is improving.

<sup>^</sup> Subjects who discontinued for disease progression but did not meet RECIST criteria for PD are classified as PD at the date of discontinuation. File Name: S:\.....\&prog name

(Data as of: 24APR2018)

Protocol: GSK208466/ADP-04511 

Population: Modified Intent-To-Treat

Table 7.2103

Sensitivity Analyses for Progression-Free Survival

mITT Population

| Sensitivity Analysis/<br>Response Category | Statistic | Cohort 1<br>(N=xx) | Cohort 2<br>(N=xx) | Cohort 3<br>(N=xx) | Cohort 4<br>(N=xx) |
|---|---|---|---|---|---|
| Replace NE with SD or | | | | | |
| PD @ | . (0) | / 0 N | ( | ( | 4 |
| Subjects with Event | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Number Censored | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Progression-Free | | | | | |
| Survival(weeks) | N | X | X | X | X |
| | Q1 (95% CI) | xx.x (xx.x, xx.x) | xx.x ( $xx.x$ , $xx.x$ ) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Median | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (95% CI) | | | | |
| | Q3 (95% CI) | xx.x ( $xx.x$ , $xx.x$ ) | xx.x ( $xx.x$ , $xx.x$ ) | xx.x ( $xx.x$ , $xx.x$ ) | xx.x (xx.x, xx.x) |
| Replace NE with SD | | | | | |
| Subjects with Event | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Number Censored | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Progression-Free | | | | | |
| Survival(weeks) | N | X | X | X | X |
| , | Q1 (95% CI) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Median | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | (95% CI) | , | , , , , , , | , , , , , , | , , , |
| | Q3 (95% CI) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |

CR = Complete Response, PR = Partial Response, SD = Stable Disease, PD = Progressive Disease, NE = Not Evaluable (Unknown or Missing).

File Name: S:\.... \&prog name

<sup>&</sup>amp; PFS is defined as the interval between the date of first T cell infusion and first disease progression, death due to any cause, surgical resection, or start of prohibited medication, except as noted in \$ footnote. Subjects without any of the aforementioned events are censored at the date of last study assessment. \$ Subjects are censored at first surgical resection or start of prohibited medications, whichever came first.

<sup>@</sup> Assign values of SD if the assessments before and after the NE assessment are CR, PR, or SD. Assign PD otherwise, except for PR NE CR where the assessment is improving.

<sup>^</sup> Subjects who discontinued for disease progression but did not meet RECIST criteria for PD are classified as PD at the date of discontinuation.


(Data as of: 24APR2018)

Protocol: GSK208466/ADP-04511

Population: Modified Intent-To-Treat

Table 7.2103

Sensitivity Analyses for Progression-Free Survival

mITT Population

| Sensitivity Analysis/ | | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 |
|---|---|---|---|---|---|
| Response Category | Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Replace NE with PD | | | | | |
| Subjects with Event | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Number Censored | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Progression-Free | | | | | |
| Survival(weeks) | N | X | X | X | X |
| | Q1 (95% CI) | xx.x ( $xx.x$ , $xx.x$ ) | xx.x ( $xx.x$ , $xx.x$ ) | xx.x ( $xx.x$ , $xx.x$ ) | xx.x ( $xx.x$ , $xx.x$ ) |
| | Median<br>(95% CI) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Q3 (95% CI) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| Progressive Disease<br>Based on Discontinuation Date<br>for Unconfirmed<br>PD ^ | | | | | |
| Subjects with Event | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Number Censored | n (%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Progression-Free | | | | | |
| Survival(weeks) | N | X | X | X | X |
| | Q1 (95% CI) | xx.x ( $xx.x$ , $xx.x$ ) | xx.x ( $xx.x$ , $xx.x$ ) | xx.x ( $xx.x$ , $xx.x$ ) | xx.x ( $xx.x$ , $xx.x$ ) |
| | Median<br>(95% CI) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| | Q3 (95% CI) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |

CR = Complete Response, PR = Partial Response, SD = Stable Disease, PD = Progressive Disease, NE = Not Evaluable (Unknown or Missing).

<sup>&</sup>amp; PFS is defined as the interval between the date of first T cell infusion and first disease progression, death due to any cause, surgical resection, or start of prohibited medication, except as noted in \$ footnote. Subjects without any of the aforementioned events are censored at the date of last study assessment. \$ Subjects are censored at first surgical resection or start of prohibited medications, whichever came first.

<sup>@</sup> Assign values of SD if the assessments before and after the NE assessment are CR, PR, or SD. Assign PD otherwise, except for PR NE CR where the assessment is improving.

<sup>^</sup> Subjects who discontinued for disease progression but did not meet RECIST criteria for PD are classified as PD at the date of discontinuation. File Name: S:\.....\&prog name

208466/ADP-04511

Protocol: GSK208466/ADP-04511 

Population: Modified Intent-To-Treat (Data as of: 24APR2018)

Table 8.0001 Summary Lymphodepleting Chemotherapy Administration for the First Infusion mITT Population

| Regimen | Statistic | Cohort 1<br>(N=xx) | Cohort 2<br>(N=xx) | Cohort 3<br>(N=xx) | Cohort 4<br>(N=xx) | Cohort 2-4 Total (N=xx) | Overall<br>(N=xx) |
|---|---|---|---|---|---|---|---|
| Initial<br>Treatment @ | | | | | | | |
| Regimen A | n/N | xx/XX | xx/XX | xx/XX | xx/XX | xx/XX | xx/XX |
| Regimen B | n/N | xx/XX | xx/XX | xx/XX | xx/XX | xx/XX | xx/XX |
| Regimen C | n/N | xx/XX | xx/XX | xx/XX | xx/XX | xx/XX | xx/XX |

File Name: S:\.....\&prog name

Note 1: n = number of subjects with the regimen, N = total number of subjects receiving treatment.

Note 2: Regimen A = Fludarabine 30 mg/m $^2$  on Days -5 to -2 and Cyclophosphamide 1800 mg/m $^2$  on Days -5 and -3. Regimen B = Cyclophosphamide 1800 mg/m $^2$  on Days -3 and -2. Regimen C = Fludarabine 30 mg/m $^2$  and Cyclophosphamide 600 mg/m $^2$  on Days -7 to -5.

<sup>@</sup> Subjects in Cohort 1 received Regimen A, subjects in Cohort 2 received Regimen A or C, subjects in Cohort 3 received Regimen B, and subjects in Cohort 4 received Regimen C.


(Data as of: 24APR2018)

Protocol: GSK208466/ADP-04511

Population: Modified Intent-To-Treat

Table 8.0002

Summary of the First T Cell Infusion

mITT Population

| Parameter | Statistic | Cohort 1 (N=xx) | Cohort 2<br>(N=xx) | Cohort 3 (N=xx) | Cohort 4<br>(N=xx) | Cohort 2-4<br>Total<br>(N=xx) | Overall<br>(N=xx) |
|---|---|---|---|---|---|---|---|
| Total Number of<br>Transduced Cells<br>(x 10^9) | N | х | Х | х | x | х | х |
| | Mean | XXX.X | XXX.X | xxx.x | xxx.x | xxx.x | xxx.x |
| | SD | XX.XX | XX.XX | xx.xx | XX.XX | xx.xx | xx.xx |
| | Median | XXX | Xxx | XXX | xxx | XXX | XXX |
| | Min,Max | XXX,XXX | xxx,xxx | xxx,xxx | xxx,xxx | xxx,xxx | xxx,xxx |

File Name: S:\.....\&prog\_name


Protocol: GSK208466/ADP-04511

Population: Modified Intent-To-Treat (Data as of: 24APR2018)

Table 8.0003

Summary of Second T Cell Infusion (Subjects with a Second T Cell Infusion)

| Parameter | Statistic | Cohort 1 (N=xx) | Cohort 2<br>(N=xx) | Cohort 3<br>(N=xx) | Cohort 4<br>(N=xx) | Cohort 2-4<br>Total<br>(N=xx) | Overall<br>(N=xx) |
|---|---|---|---|---|---|---|---|
| Total Number of<br>Transduced Cells<br>(x 10^9) | N | х | х | х | х | x | x |
| | Mean | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X | xxx.x |
| | SD | XX.XX | XX.XX | xx.xx | xx.xx | xx.xx | xx.xx |
| | Median | XXX | Xxx | xxx | xxx | xxx | xxx |
| | Min,Max | XXX, XXX | XXX,XXX | xxx,xxx | xxx,xxx | xxx,xxx | xxx,xxx |

File Name: S:\.....\&prog\_name

Protocol: GSK208466/ADP-04511 Population: Intent-To-Treat  (Data as of: 24APR2018)

Table 8.1001
Overall Summary of Adverse Events for Period 1
ITT Population
ADAE.PER01FL = 'Y'
ITTFL = 'Y'
Do not use treatment-emergent flag.
Use ARM

| Category | Cohort 1 (N=xx) | Cohort 2<br>(N=xx) | Cohort 3<br>(N=xx) | Cohort 4<br>(N=xx) | Cohort 2-4 Total (N=xx) | Overall (N=xx) |
|---|---|---|---|---|---|---|
| | , , | | , , | , , | | |
| Subjects with Any AEs | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Subjects with Any AEs Related& to T Cell Therapy RELGR1 = 'Related' | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Subjects with Any AEs >= Grade 3 TOXGGR1 = 'Grade 3 or Higher' | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Subjects with Any AEs Related& T Cell Therapy and Grade >= 3 RELGR1 = 'Related', TOXGGR1 = 'Grade 3 or Higher' | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| TOAGGRI - Grade 3 Or Higher | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Subjects with Any AEs Related& T Cell Therapy and Fatal Outcome | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Subjects with Any Serious AEs (SAE) AESER = 'Y' | | | | | | |
| Subjects with Any SAEs Related& to T Cell Therapy AESER = 'Y', RELGR1 = 'Related' | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Subjects with Any SAEs >= Grade 3 AESER = 'Y', TOXGGR1 = 'Grade 3 or Higher' | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Subjects with Any SAEs Related& to T Cell Therapy and Grade >= 3 AESER = 'Y', PELCEL No. 1 TOYCORI - Young 2 or Wicher! | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| RELGR1='Related', TOXGGR1='Grade 3 or Higher' Subjects with Any SAEs with Fatal Outcome AESER = 'Y', AEOUT = 'FATAL' | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |

```
Period 1 = from date of informed consent through end of study.

& Treatment-related: definitely related, probably related, possibly related, or unlikely related to T cell infusion.
File Name: S:\.....\&prog_name
Repeat Table 8.1001 template for:

Table 8.1003

Overall Summary of Adverse Events for Period 2.

mITT Population

(replace Period 1 footnote with: Period 2 = from start date of lymphodepletion through end of study.)

ADAE.PER02FL = 'Y'

MITTFL = 'Y'

Do not use treatment-emergent flag.

Use ARM.
```

SAE = serious adverse event.

Protocol: GSK208466/ADP-04511 

Population: Intent-To-Treat (Data as of: 24APR2018)

Table 8.1101

Incidence of Adverse Events by System Organ Class and Preferred Term for Period 1

ITT Population

ADAE.PER01FL = 'Y'

ITTFL = 'Y'

Do not use treatment-emergent flag for any tables.

Use ARM for all tables

| System Organ Class/<br>ADAE.AEBODSYS | | | | | Cohort 2-4 | |
|---|---|---|---|---|---|---|
| Preferred Term<br>ADAE.AEDECOD | Cohort 1<br>(N=xx) | Cohort 2<br>(N=xx) | Cohort 3 (N=xx) | Cohort 4 (N=xx) | Total (N=xx) | Overall<br>(N=xx) |
| Any Adverse Event | xx(xx.x %) | xx(xx.x %) | xx(xx.x %) | xx(xx.x %) | xx(xx.x %) | xx(xx.x %) |
| SOC1 | xx(xx.x %) | xx(xx.x %) | xx(xx.x %) | xx(xx.x %) | xx(xx.x %) | xx(xx.x %) |
| Term 1 | xx(xx.x %) | xx(xx.x %) | xx(xx.x %) | xx(xx.x %) | xx(xx.x %) | xx(xx.x %) |
| Term 2 | xx(xx.x %) | xx(xx.x %) | xx(xx.x %) | xx(xx.x %) | xx(xx.x %) | xx(xx.x %) |
| SOC2 | xx(xx.x %) | xx(xx.x %) | xx(xx.x %) | xx(xx.x %) | xx(xx.x %) | xx(xx.x %) |
| Term 1 | xx(xx.x %) | xx(xx.x %) | xx(xx.x %) | xx(xx.x %) | xx(xx.x %) | xx(xx.x %) |
| Term 2 | xx(xx.x %) | xx(xx.x %) | xx(xx.x %) | xx(xx.x %) | xx(xx.x %) | xx(xx.x %) |

Etc.

Programming Note: Sort SOCs by descending frequency of subjects in Overall column, then alphabetically. Within each SOC, sort PTs by descending frequency of subjects Overall column, then alphabetically.

Period 1 = from date of informed consent through end of study.

Note 1: Subjects are counted once for each system organ class and once for each preferred term.

Note 2: System organ classes (and preferred terms within each) are sorted by descending frequency according to the Overall group.

File Name: S:\.... \&prog name

# Repeat Table 8.1101 template for:

```
Table 8.1103
Incidence of Adverse Events by System Organ Class and Preferred Term for Period 2
(replace Period 1 footnote with: Period 2 = from start date of lymphodepletion through end of study.)
ADAE.PER02FL = 'Y'
MITTFL = 'Y'
Use ARM
Table 8.1104
Summary of Adverse Events Grouped by Similarity of Preferred Terms for Period 1
ADAE.PER01FL = 'Y'
TTTFI = 'Y'
Use ARM
Table 8.1106
Summary of Adverse Events Grouped by Similarity of Preferred Terms for Period 2
(replace Period 1 footnote with: Period 2 = from start date of lymphodepletion through end of study.)
ADAE.PER02FL = 'Y'
MITTFL = 'Y'
Use ARM
Footnotes for 8.1104, 8.1101:
Period 1 = from date of informed consent through end of study.
Note 1: Subjects are counted once for each synonym and once for each preferred term
Note 2: Synonyms (and preferred terms within each) are sorted by descending frequency according to the Overall group.
File Name: S:\.....\&prog name
```


Population: Intent-To-Treat (Data as of: 24APR2018)

Table 8.1201

Incidence of Adverse Events by Toxicity Grade and Preferred Term for Period 1

ITT Population

Cohort 1 (N=xxx)

| | Maxim | num Grade | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Preferred Term | 1 | 2 | 3 | 4 | 5 | 3+4+5 | Unknown | Total |
| Any Adverse Event | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Term 1 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Term 2 | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Term 3 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Term 4 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Term 5 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |

Period 1 = from date of informed consent through end of study.

Note 1: Subjects are counted once for each system organ class and once for each preferred term under the most severe toxicity grade.

Note 2: System organ classes (and preferred terms within each) are sorted by descending frequency in the Overall group.

Note 3: Synonymous preferred terms are combined.

Note to programmer: Include only Grades with frequency > 0 for Overall columns. Please only present synonym terms as described in appendix 2.

File Name: S:\.....\&prog name

208466/ADP-04511


Population: Intent-To-Treat (Data as of: 24APR2018)

Table 8.1201

Incidence of Adverse Events by Toxicity Grade Preferred Term for Period 1

ITT Population
Cohort 2 (N=xxx)

| | Maxin | num Grade | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Preferred Term | 1 | 2 | 3 | 4 | 5 | 3+4+5 | Unknown | Total |
| Any Adverse Event | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Term 1 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Term 2 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Term 3 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Term 4 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Term 5 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |

Period 1 = from date of informed consent through end of study.

File Name: S:\.... \&prog name

Note 1: Subjects are counted once for each system organ class and once for each preferred term under the most severe toxicity grade.

Note 2: System organ classes (and preferred terms within each) are sorted by descending frequency in the Overall group.

Note 3: Synonymous preferred terms are combined.

Note to programmer: Include only Grades with frequency > 0 for Overall columns. Please only present synonym terms as described in appendix 2.


Population: Intent-To-Treat (Data as of: 24APR2018)

Table 8.1201

Incidence of Adverse Events by Toxicity Grade Preferred Term for Period 1

ITT Population
Cohort 3 (N=xxx)

| | Maxim | Maximum Grade | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Preferred Term | 1 | 2 | 3 | 4 | 5 | 3+4+5 | Unknown | Total |
| Any Adverse Event | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Term 1 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Term 2 | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Term 3 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Term 4 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Term 5 | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| *** | | | | | | | | |

Period 1 = from date of informed consent through end of study.

File Name: S:\.... \&prog name

Note 1: Subjects are counted once for each system organ class and once for each preferred term under the most severe toxicity grade.

Note 2: System organ classes (and preferred terms within each) are sorted by descending frequency in the Overall group.

Note 3: Synonymous preferred terms are combined.

Note to programmer: Include only Grades with frequency > 0 for Overall columns. Please only present synonym terms as described in appendix 2.


Population: Intent-To-Treat (Data as of: 24APR2018)

Table 8.1201

Incidence of Adverse Events by Toxicity Grade and Preferred Term for Period 1

ITT Population
Cohort 4 (N=xxx)

| | Maxim | Maximum Grade | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Preferred Term | 1 | 2 | 3 | 4 | 5 | 3+4+5 | Unknown | Total |
| Any Adverse Event | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Term 1 | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Term 2 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Term 3 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Term 4 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Term 5 | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |

Period 1 = from date of informed consent through end of study.

Note 1: Subjects are counted once for each system organ class and once for each preferred term under the most severe toxicity grade.

Note 2: System organ classes (and preferred terms within each) are sorted by descending frequency in the Overall group.

Note 3: Synonymous preferred terms are combined.

Note to programmer: Include only Grades with frequency > 0 for Overall columns. Please only present synonym terms as described in appendix 2.

# 208466/ADP-04511

Page 1 of n (Data as of: 24APR2018)

Protocol: GSK208466/ADP-04511
Population: Intent-To-Treat

Table 8.1201

Incidence of Adverse Events by Toxicity Grade and Preferred Term for Period 1

ITT Population
Cohort 2-4 (N=xxx)

| | Maxim | num Grade | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Preferred Term | 1 | 2 | 3 | 4 | 5 | 3+4+5 | Unknown | Total |
| Any Adverse Event | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Term 1 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Term 2 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Term 3 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Term 4 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Term 5 | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |

Period 1 = from date of informed consent through end of study.

Note 1: Subjects are counted once for each system organ class and once for each preferred term under the most severe toxicity grade.

Note 2: System organ classes (and preferred terms within each) are sorted by descending frequency in the Overall group.

Note 3: Synonymous preferred terms are combined.

Note to programmer: Include only Grades with frequency > 0 for Overall columns. Please only present synonym terms as described in appendix 2.

File Name: S:\.... \&prog name

## 208466/ADP-04511

Page 1 of n (Data as of: 24APR2018)

Protocol: GSK208466/ADP-04511 Population: Intent-To-Treat

Table 8.1201

Incidence of Adverse Events by Toxicity Grade and Preferred Term for Period 1

ITT Population
Cohort 1-4 (N=xxx)

| | Maxim | Maximum Grade | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Preferred Term | 1 | 2 | 3 | 4 | 5 | 3+4+5 | Unknown | Total |
| Any Adverse Event | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Term 1 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Term 2 | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Term 3 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Term 4 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Term 5 | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |

Period 1 = from date of informed consent through end of study.

Note 1: Subjects are counted once for each system organ class and once for each preferred term under the most severe toxicity grade.

Note 2: System organ classes (and preferred terms within each) are sorted by descending frequency in the Overall group.

Note 3: Synonymous preferred terms are combined.

Note to programmer: Include only Grades with frequency > 0 for Overall columns. Please only present synonym terms as described in appendix 2.

File Name: S:\.....\&prog\_name
Repeat Table 8.1201 template for:

### Table 8.1203

Incidence of Adverse Events by Toxicity Grade Class and Preferred Term for Period 2 mITT Population

(replace Period 1 footnote with: Period 2 = from start date of lymphodepletion through end of study.)

ADAE.PER02FL = 'Y'

MITTFL = 'Y'

Use ARM

Include only Grades with frequency > 0 for Overall columns.

### Table 8.1204

Incidence of Treatment Adverse Events by Toxicity Grade Class and Preferred Term for Period 2 mITT Population

(replace Period 1 footnote with: Period 2 = from start date of lymphodepletion through end of study.)

208466/ADP-04511

Protocol: GSK208466/ADP-04511
Population: Modified Intent-To-Treat (Data as of: 24APR2018)

Table 8.1205

Incidence of Treatment Related Adverse Events by System Organ Class and Preferred Term for Period 1

mITT Population

ADAE.PER01FL = 'Y'

MITTFL = 'Y'

Use ARM

Include only related AEs (RELGR1 = 'Related').

| System Organ<br>Class/ADAE.AEBODSYS<br>Preferred Term ADAE.AEDECOD | Cohort 1<br>(N=xx) | Cohort 2<br>(N=xx) | Cohort 3<br>(N=xx) | Cohort 4<br>(N=xx) | Cohort 2-4<br>Total<br>(N=xx) | Overall<br>(N=xx) |
|---|---|---|---|---|---|---|
| Any Adverse Event | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| SOC1 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Term 1 Term 2 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |

Etc.

File Name: S:\.....\&prog name

Period 1 = from date of informed consent through end of study.

Note 1: Subjects are counted once for each system organ class and once for each preferred term under the strongest relationship.

Note 2: Related adverse events have a relationship of definitely related, probably related, possibly related, or unlikely related to T cell infusion or lymphodepletion chemotherapy (cyclophosphamide and/or Mesna).

Note 3: System organ classes (and preferred terms within each) are sorted by descending frequency in the Overall group.

208466/ADP-04511

# Use 8.1205 as a template for the following Tables:

```
Table 8.1206
Incidence of Treatment Related Adverse Events by System Organ Class and Preferred Term for Period 2 mITT Population
(replace Period 1 footnote with: Period 2 = from start date of lymphodepletion through end of study.)
ADAE.PER02FL = 'Y'
MITTFL = 'Y'
Use ARM
Include only related AEs (RELGR1 = 'Related').
```

# Use 8.1101 as a template for the following Tables:

## Table 8.1301

```
Incidence of Adverse Events with Toxicity Grade >=3 by System Organ Class and Preferred Term for Period 1
ITT Population
ADAE.PER01FL = 'Y'
ITTFL = 'Y'
TOXGGR1 = 'Grade 3 or Higher'
Use ARM
```

### Table 8.1303

Incidence of Adverse Events with Toxicity Grade  $\geq$ 3 by System Organ Class and Preferred Term for Period 2 mITT Population

(replace Period 1 footnote with: Period 2 = from start date of lymphodepletion through end of study.)
ADAE.PER02FL = 'Y'
MITTFL = 'Y'
TOXGGR1 = 'Grade 3 or Higher'
Use ARM

208466/ADP-04511

# Use 8.1205 as a template for the following Tables:

```
Table 8.1305
Incidence of Treatment Related Adverse Events with Toxicity Grade >=3 by System Organ Class and Preferred Term for Period 1
mITT Population
ADAE.PER01FL = 'Y'
MITTFL = 'Y'
Use Include only related AEs (RELGR1 = 'Related').
TOXGGR1 = 'Grade 3 or Higher'
Use ARM
Table 8.1306
Incidence of Treatment Related Adverse Events with Toxicity Grade >=3 by System Organ Class and Preferred Term for Period 2
(replace Period 1 footnote with: Period 2 = from start date of lymphodepletion through end of study.)
ADAE.PER02FL = 'Y'
MITTFL = 'Y'
Use Include only related AEs (RELGR1 = 'Related').
TOXGGR1 = 'Grade 3 or Higher'
Use ARM
```

Use Table 8.1101 as a template for the following Tables:

#### Table 8.1401

Incidence of Serious Adverse Events by System Organ Class and Preferred Term for the Pre-leukapheresis Period ITT Population

ADAE.PRELEUFL = 'Y'
(no pop specified)
AESER = 'Y'

Use ARM [it looks like there are no AEs meeting criteria at this point]

Programming note: Change the "Population: Modified Intent-To-Treat" in the upper left to "Population: Intent-to-Treat".

### Footnotes for Table 8.1401:

Note 1: Subjects are counted once for each system organ class and once for each preferred term.

Note 2: Serious adverse events that occur after the date of informed consent and prior to date of leukapheresis are included.

Note 3: System organ classes (and preferred terms within each) are sorted by descending frequency in the Overall group.

### Table 8.1402

Incidence of Serious Adverse Events by System Organ Class and Preferred Term for Period 1 ITT Population

ADAE.PER01FL = 'Y'
ITTFL = 'Y'
AESER = 'Y'
Use ARM

## Table 8.1404

Incidence of Serious Adverse Events by System Organ Class and Preferred Term for the Period 2 mITT Population

(replace Period 1 footnote with: Period 2 = from start date of lymphodepletion through end of study.)

ADAE.PER02FL = 'Y'
MITTFL = 'Y'
AESER = 'Y'
Use ARM

208466/ADP-04511

Use 8.1205 as a template for the following Tables:

```
Table 8.1502
```

Incidence of Treatment Related Serious Adverse Events by System Organ Class and Preferred Term for Period 1 mITT Population

ADAE.PER01FL = 'Y'
MITTFL = 'Y'
AESER = 'Y'
RELGR1 = 'Related'
Use ARM

## Table 8.1503

Incidence of Treatment Related Serious Adverse Events by System Organ Class and Preferred Term for Period 2 mITT Population

(replace Period 1 footnote with: Period 2 = from start date of lymphodepletion through end of study.)

ADAE.PER02FL = 'Y'
MITTFL = 'Y'
AESER = 'Y'
RELGR1 = 'Related'
Use ARM

## Repeat Table 8.1201 template for:

#### Table 8.1504

Incidence of Serious Adverse Events by Toxicity Grade and Preferred Term for Period 1 ITT population

### Table 8.1505

Incidence of Serious Adverse Events by Toxicity Grade and Preferred Term for Period 2 mITT population

(replace Period 1 footnote with: Period 2 = from start date of lymphodepletion through end of study.)

#### Table 8.1506

Incidence of Treatment Related Serious Adverse Events by Toxicity Grade and Preferred Term for Period 2 mITT population

(replace Period 1 footnote with: Period 2 = from start date of lymphodepletion through end of study.)

## Use 8.1101 as a template for the following Tables:

#### Table 8.1601

Incidence of Serious Adverse Events with Toxicity Grade >= 3 by System Organ Class and Preferred Term for the Pre-leukapheresis Period ITT Population

#### Footnotes:

Note 1: Subjects are counted once for each system organ class and once for each preferred term.

Note 2: Serious adverse events that occur after the date of informed consent and prior to date of leukapheresis are included.

Note 3: System organ classes (and preferred terms within each) are sorted by descending frequency in the Overall group.

ADAE.PRELEUFL = 'Y'

(no pop specified)

AESER = 'Y'

TOXGGR1 = 'Grade 3 or Higher'

Use ARM [it looks like there are no AEs meeting criteria at this point]

Programming note: Change the "Population: Modified Intent-To-Treat" in the upper left to "Population: Intent-to-Treat".

### Table 8.1602

```
Incidence of Serious Adverse Events with Toxicity Grade >=3 by System Organ Class and Preferred Term for Period 1
ITT Population
ADAE.PER01FL = 'Y'
ITTFL = 'Y'
AESER = 'Y'
TOXGGR1 = 'Grade 3 or Higher'
Use ARM
```

### Table 8.1604

208466/ADP-04511

Incidence of Serious Adverse Events with Toxicity Grade >=3 by System Organ Class and Preferred Term for Period 2 mITT Population

(replace Period 1 footnote with: Period 2 = from start date of lymphodepletion through end of study.)
ADAE.PER02FL = 'Y'
MITTFL = 'Y'
AESER = 'Y'
TOXGGR1 = 'Grade 3 or Higher'
Use ARM

208466/ADP-04511

# Use 8.1205 as a template for the following Tables:

### Table 8.1606

Incidence of Treatment Related Serious Adverse Events with Toxicity Grade >=3 by System Organ Class and Preferred Term for Period 1
mITT Population

ADAE.PER01FL = 'Y'
MITTFL = 'Y'
AESER = 'Y'
RELGR1 = 'Related'
TOXGGR1 = 'Grade 3 or Higher'
Use ARM

## Table 8.1607

Incidence of Treatment Related Serious Adverse Events with Toxicity Grade >=3 by System Organ Class and Preferred Term for Period 2
mITT Population

(replace Period 1 footnote with: Period 2 = from start date of lymphodepletion through end of study.)

ADAE.PER02FL = 'Y'
MITTFL = 'Y'
AESER = 'Y'
RELGR1 = 'Related'
TOXGGR1 = 'Grade 3 or Higher'
Use ARM

## Use 8.1101 as a template for the following Tables:

#### Table 8.1608

Incidence of Serious Adverse Events Resulting in Death by System Organ Class and Preferred Term for the Pre-leukapheresis Period
ITT Population
ADAE.PRELEUFL = 'Y'
(no pop specified)
AESER = 'Y'
AEOUT = 'FATAL'
Use ARM [it looks like there are no AEs meeting criteria at this point]

#### Footnotes:

Note 1: Subjects are counted once for each system organ class and once for each preferred term.

Note 2: Serious adverse events that occur after the date of informed consent and prior to date of leukapheresis are included.

Note 3: System organ classes (and preferred terms within each) are sorted by descending frequency in the Overall group.

Programming note: Change the "Population: Modified Intent-To-Treat" in the upper left to "Population: Intent-to-Treat".

AESER = 'Y'
AEOUT = 'FATAL'

#### Table 8.2101

Incidence of Serious Adverse Events Resulting in Death by System Organ Class and Preferred Term for Period 1
ITT Population
ADAE.PER01FL = 'Y'
MITTFL = 'Y'
AESER = 'Y'
AEOUT = 'FATAL'

## Table 8.2103

Incidence of Serious Adverse Events Resulting in Death by System Organ Class and Preferred Term for Period 2 mITT Population (replace Period 1 footnote with: Period 2 = from start date of lymphodepletion through end of study.)

ADAE.PER02FL = 'Y'
MITTFL = 'Y'
AESER = 'Y'
AEOUT = 'FATAL'

208466/ADP-04511

Protocol: GSK208466/ADP-04511
Population: Modified Intent-To-Treat

(Data as of: 24APR2018)


Table 8.3001

Overall Summary of Adverse Events for the Post-lymphodepletion Period for the Second T Cell Infusion Subjects with a Second T Cell Infusion

ADAE.INF2FL = 'Y'

TRT02A = 'T-CELL' (denominator)

| Category | Overall (N=xx) |
|---|---|
| Subjects with Any AEs | x (xx.x%) |
| Subjects with Any AEs Related& to T Cell Therapy RELGR1 = 'Related' | x (xx.x%) |
| Subjects with Any AEs >= Grade 3 TOXGGR1 = 'Grade 3 or Higher' | x (xx.x%) |
| Subjects with Any Serious AEs (SAE) AESER = 'Y' | x (xx.x%) |
| Subjects with Any SAEs with Fatal Outcome AESER = 'Y', AEOUT = 'FATAL' | x (xx.x%) |

SAE = serious adverse event.

& Treatment-related: definitely related, probably related, or possibly related to T cell infusion.

File Name: S:\.....\&prog\_name

208466/ADP-04511

Protocol: GSK208466/ADP-04511
Population: Modified Intent-To-Treat

(Data as of: 24APR2018)

Table 8.3002

Incidence of Adverse Events by System Organ Class and Preferred Term for the Post-lymphodepletion Period for the Second T Cell Infusion Subjects with a Second T Cell Infusion

ADAE.INF2FL = 'Y'
TRT02A = 'T-CELL' (denominator)

| Preferred Term ADAE.AEDECOD | Overall (N=xx) |
|-----------------------------|----------------|
| Any Adverse Event | xx(xx.x %) |
| SOC1 | xx(xx.x %) |
| Term 1 | xx(xx.x %) |
| Term 2 | xx(xx.x %) |
| SOC2 | xx(xx.x %) |
| Term 1 | xx(xx.x %) |
| Term 2 | xx (xx . x %) |

Note 1: Subjects are counted once for each system organ class and once for each preferred term.

Note 2: System organ classes (and preferred terms within each) are sorted by descending frequency according to the Overall group.

File Name: S:\.....\&prog name

(Data as of: 24APR2018)


Protocol: GSK208466/ADP-04511
Population: Modified Intent-To-Treat

Table 8.3003

Incidence of Adverse Events by Toxicity Grade and Preferred Term for the Post-lymphodepletion Period for the Second T-Cell Infusion Period Subjects with a Second T-Cell Infusion

Total (N=xxx)

| | Ma | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Preferred Term | 1 | 2 | 3 | 4 | 5 | 3+4+5 | Unknown | Total |
| Any Adverse Event | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) |
| Term 1 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Term 2 | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Term 3 | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Term 4 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Term 5 | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |

Note 1: Subjects are counted once for each system organ class and once for each preferred term under the most severe toxicity grade.

Note 2: System organ classes (and preferred terms within each) are sorted by descending frequency in the Overall group.

Note 3: Synonymous preferred terms are combined.

Note to programmer: Include only Grades with frequency > 0 for Overall columns. Please only present synonym terms as described in appendix 2.

File Name: S:\.... \&prog name

208466/ADP-04511

## Use 8.3002 as a template for the following Tables:

### Table 8.3004

Incidence of Treatment Related Adverse Events by System Organ Class and Preferred Term for the Post-lymphodepletion Period for the Second T-Cell Infusion Subjects with a Second T Cell Infusion

Add footnote: Note 2: Related adverse events have a relationship of definitely related, probably related, or possibly related to T cell infusion or lymphodepletion chemotherapy (cyclophosphamide and/or Mesna).

ADAE.INF2FL = 'Y'

TRT02A = 'T-CELL' (denominator)

RELGR1 = 'Related'

#### Table 8.3005

Incidence of Serious Adverse Events by System Organ Class and Preferred Term for the Post-lymphodepletion Period for the Second T Cell Infusion Subjects with a Second T Cell Infusion

ADAE.INF2FL = 'Y'

TRT02A = 'T-CELL' (denominator)

AESER = 'Y'

208466/ADP-04511

## Use 8.3003 as a template for the following Tables:

### Table 8.3006

Incidence of Treatment Related Adverse Events by Toxicity Grade and Preferred Term for the Post-lymphodepletion Period for the Second T-Cell Infusion

Population: Subjects with a Second T-Cell Infusion

## Table 8.3007

Incidence of Serious Adverse Events by Toxicity Grade and Preferred Term for the Post-lymphodepletion Period for the Second T-Cell Infusion

Population: Subjects with a Second T-Cell Infusion

## Table 8.3008

Incidence of Treatment Related Serious Adverse Events by Toxicity Grade and Preferred Term for the Post-lymphodepletion Period for the Second T-Cell Infusion

Population: Subjects with a Second T-Cell Infusion

# 208466/ADP-04511


(Data as of: 24APR2018)

Protocol: GSK208466/ADP-04511

Population: Modified Intent-To-Treat

Table 8.3101

Summary of Adverse Events of Special Interest by Cohort (All Infusions)

Cohort 1 (N=xx)

| | | Maximum Grade | | | | | | |
|---|---|---|---|---|---|---|---|---|
| AESI Category | 1 | 2 | 2 | 4 | F | 2.4.5 | II.a lan assa | maka 1 |
| Preferred Term | Ι | ۷ | 3 | 4 | 5 | 3+4+5 | Unknown | Total |
| ANY EVENT | 1 (1%) | 4 (5%) | 6 (7%) | 71 (86%) | 0 | 77 (93%) | 0 | 82 (99%) |
| Potential symptoms of GVHD | | | | | | | | |
| Any Event | 24 (29%) | 31 (37%) | 26 (31%) | 0 | 0 | 26 (31%) | 0 | 81 (98%) |
| Nausea | 40 (48%) | 26 (31%) | 5 (6%) | 0 | 0 | 5 (6%) | 0 | 71 (86%) |
| Diarrhoea | 23 (28%) | 14 (17%) | 11 (13%) | 0 | 0 | 11 (13%) | 0 | 48 (58%) |
| Rash maculo-papular | 17 (20%) | 8 (10%) | 6 (7%) | 0 | 0 | 6 (7%) | 0 | 31 (37%) |
| Abdominal pain | 15 (18%) | 6 (7%) | 4 (5%) | 0 | 0 | 4 (5%) | 0 | 25 (30%) |

Programming note: AESI list will be provided by GSK. Please use the AESI list and report the synonym terms as described in appendix 2.

•

Note 1: Subjects are counted once for each preferred term under the most severe grade.

Note 2: Preferred terms are sorted by descending frequency of 'Total' AEs.

Note 3: Adverse events with missing grade are only included in 'Unknown' and 'Total' columns.

Note 4: Synonymous preferred terms are combined.

# 208466/ADP-04511


(Data as of: 24APR2018)

Protocol: GSK208466/ADP-04511

Population: Modified Intent-To-Treat

Table 8.3101

Summary of Adverse Events of Special Interest by Cohort (All Infusions)

Cohort 2 (N=xx)

| | | Maximum Grade | | | | | | |
|---|---|---|---|---|---|---|---|---|
| AESI Category Preferred Term | 1 | 2 | 2 | 4 | E | 3+4+5 | Unknown | Total |
| Preferred Term | 1 | | 3 | 4 | 5 | 37473 | Ulikilowii | IOLAI |
| ANY EVENT | 1 (1%) | 4 (5%) | 6 (7%) | 71 (86%) | 0 | 77 (93%) | 0 | 82 (99%) |
| Potential symptoms of GVHD | | | | | | | | |
| Any Event | 24 (29%) | 31 (37%) | 26 (31%) | 0 | 0 | 26 (31%) | 0 | 81 (98%) |
| Nausea | 40 (48%) | 26 (31%) | 5 (6%) | 0 | 0 | 5 (6%) | 0 | 71 (86%) |
| Diarrhoea | 23 (28%) | 14 (17%) | 11 (13%) | 0 | 0 | 11 (13%) | 0 | 48 (58%) |
| Rash maculo-papular | 17 (20%) | 8 (10%) | 6 (7%) | 0 | 0 | 6 (7%) | 0 | 31 (37%) |
| Abdominal pain | 15 (18%) | 6 (7%) | 4 (5%) | 0 | 0 | 4 (5%) | 0 | 25 (30%) |

Programming note: AESI list will be provided by GSK. Please use the AESI list and report the synonym terms as described in appendix 2.

Note 1: Subjects are counted once for each preferred term under the most severe grade.

Note 2: Preferred terms are sorted by descending frequency of 'Total' AEs.

Note 3: Adverse events with missing grade are only included in 'Unknown' and 'Total' columns.

Note 4: Synonymous preferred terms are combined.

(Data as of: 24APR2018)


Protocol: GSK208466/ADP-04511

Population: Modified Intent-To-Treat

Table 8.3101

Summary of Adverse Events of Special Interest by Cohort (All Infusions)

Cohort 3 (N=xx)

| | | Maximum G | rade | | | | | |
|---|---|---|---|---|---|---|---|---|
| AESI Category<br>Preferred Term | 1 | 2 | 3 | 4 | 5 | 3+4+5 | Unknown | Total |
| ANY EVENT | 1 (1%) | 4 (5%) | 6 (7%) | 71 (86%) | 0 | 77 (93%) | 0 | 82 (99%) |
| Potential symptoms of GVHD | | | | | | | | |
| Any Event | 24 (29%) | 31 (37%) | 26 (31%) | 0 | 0 | 26 (31%) | 0 | 81 (98%) |
| Nausea | 40 (48%) | 26 (31%) | 5 (6%) | 0 | 0 | 5 (6%) | 0 | 71 (86%) |
| Diarrhoea | 23 (28%) | 14 (17%) | 11 (13%) | 0 | 0 | 11 (13%) | 0 | 48 (58%) |
| Rash maculo-papular | 17 (20%) | 8 (10%) | 6 (7%) | 0 | 0 | 6 (7%) | 0 | 31 (37%) |
| Abdominal pain | 15 (18%) | 6 (7%) | 4 (5%) | 0 | 0 | 4 (5%) | 0 | 25 (30%) |

Note 1: Subjects are counted once for each preferred term under the most severe grade.

Note 2: Preferred terms are sorted by descending frequency of 'Total' AEs.

Note 3: Adverse events with missing grade are only included in 'Unknown' and 'Total' columns.

Note 4: Synonymous preferred terms are combined.

Programming note: AESI list will be provided by GSK. Please use the AESI list and report the synonym terms as described in appendix 2.


(Data as of: 24APR2018)

Protocol: GSK208466/ADP-04511

Population: Modified Intent-To-Treat

Table 8.3101

Summary of Adverse Events of Special Interest by Cohort (All Infusions)

Cohort 4 (Nevv)

| | | Maximum Gr | rade | | | | | |
|---|---|---|---|---|---|---|---|---|
| AESI Category<br>Preferred Term | 1 | 2 | 3 | 4 | 5 | 3+4+5 | Unknown | Total |
| ANY EVENT | 1 (1%) | 4 (5%) | 6 (7%) | 71 (86%) | 0 | 77 (93%) | 0 | 82 (99%) |
| Potential symptoms of GVHD | | | | | | | | |
| Any Event | 24 (29%) | 31 (37%) | 26 (31%) | 0 | 0 | 26 (31%) | 0 | 81 (98%) |
| Nausea | 40 (48%) | 26 (31%) | 5 (6%) | 0 | 0 | 5 (6%) | 0 | 71 (86%) |
| Diarrhoea | 23 (28%) | 14 (17%) | 11 (13%) | 0 | 0 | 11 (13%) | 0 | 48 (58%) |
| Rash maculo-papular | 17 (20%) | 8 (10%) | 6 (7%) | 0 | 0 | 6 (7%) | 0 | 31 (37%) |
| Abdominal pain | 15 (18%) | 6 (7%) | 4 (5%) | 0 | 0 | 4 (5%) | 0 | 25 (30%) |

Programming note: AESI list will be provided by GSK. Please use the AESI list and report the synonym terms as described in appendix 2.

Note 1: Subjects are counted once for each preferred term under the most severe grade.

Note 2: Preferred terms are sorted by descending frequency of 'Total' AEs.

Note 3: Adverse events with missing grade are only included in 'Unknown' and 'Total' columns.

Note 4: Synonymous preferred terms are combined.
208466/ADP-04511

Page 1 of n

(Data as of: 24APR2018)

Protocol: GSK208466/ADP-04511 Population: Modified Intent-To-Treat

Table 8.3101

Summary of Adverse Events of Special Interest by Cohort (All Infusions)

Overall (Nevy)

| | | Maximum Gr | ade | | | | | |
|---|---|---|---|---|---|---|---|---|
| AESI Category<br>Preferred Term | 1 | 2 | 3 | 4 | 5 | 3+4+5 | Unknown | Total |
| ANY EVENT | 1 (1%) | 4 (5%) | 6 (7%) | 71 (86%) | 0 | 77 (93%) | 0 | 82 (99%) |
| Potential symptoms of GVHD | | | | | | | | |
| Any Event | 24 (29%) | 31 (37%) | 26 (31%) | 0 | 0 | 26 (31%) | 0 | 81 (98%) |
| Nausea | 40 (48%) | 26 (31%) | 5 (6%) | 0 | 0 | 5 (6%) | 0 | 71 (86%) |
| Diarrhoea | 23 (28%) | 14 (17%) | 11 (13%) | 0 | 0 | 11 (13%) | 0 | 48 (58%) |
| Rash maculo-papular | 17 (20%) | 8 (10%) | 6 (7%) | 0 | 0 | 6 (7%) | 0 | 31 (37%) |
| Abdominal pain | 15 (18%) | 6 (7%) | 4 (5%) | 0 | 0 | 4 (5%) | 0 | 25 (30%) |

Note 1: Subjects are counted once for each preferred term under the most severe grade.

Note 2: Preferred terms are sorted by descending frequency of 'Total' AEs.

Note 3: Adverse events with missing grade are only included in 'Unknown' and 'Total' columns.

Note 4: Synonymous preferred terms are combined.

Programming note: AESI list will be provided by GSK. Please use the AESI list and report the synonym terms as described in appendix 2.

#### Use 8.3101 as a template for the following Table:

#### Table 8.3102

Summary of Adverse Events of Special Interest for the First Infusion Programming note: Please use the AESI list and report the synonym terms as described in appendix 2.

#### Use 8.3101 as a template for the following Table:

#### Table 8.3103

Overall Summary of Adverse Events of Special Interest by Cohort for the Second Infusion Programming note: Please use the AESI list and report the synonym terms as described in appendix 2. Protocol: GSK208466/ADP-04511

 Population: Modified Intent-To-Treat (Data as of: 24APR2018)

Table 8.3104


Summary of Characterisics of Guillain-Barre Syndrome (All Infusions)

| | Cohort 1<br>(N=xx) | Cohort 2<br>(N=xx) | Cohort 3<br>(N=xx) | Cohort 4<br>(N=xx) | Cohort 2 -4 Total (N=xx) | Overall (N=xx) |
|---|---|---|---|---|---|---|
| Number of Subjects with Events | 50 (50%) | 40 (40%) | 50 (50%) | 40 (40%) | 50 (50%) | 40 (40%) |
| Number of Events | 60 | 40 | 60 | 40 | 60 | 40 |
| Event Characteristics [1] | | | | | | |
| n | 50 | 40 | 50 | 40 | 50 | 40 |
| Serious | 10/50 (20%) | 4/40 (10%) | 10/50 (20%) | 4/40 (10%) | 10/50 (20%) | 4/40 (10%) |
| Drug-related | 5/50 (10%) | 3/40 (8%) | 5/50 (10%) | 3/40 (8%) | 5/50 (10%) | 3/40 (8%) |
| Fatal | 0 | 0 | 0 | 0 | 0 | 0 |
| Number of occurrences | | | | | | |
| n | 50 | 40 | 50 | 40 | 50 | 40 |
| One | 40/50 (80%) | 40/40 (100%) | 40/50 (80%) | 40/40 (100%) | 40/50 (80%) | 40/40 (100%) |
| Two | 10/50 (20%) | 0 | 10/50 (20%) | 0 | 10/50 (20%) | 0 |
| Three or more | 0 | 0 | 0 | 0 | 0 | 0 |
| Outcome [2] | | | | | | |
| n | 50 | 40 | 50 | 40 | 50 | 40 |
| Recovered/Resolved | 50/50 (100%) | 30/40 (75%) | 50/50<br>(100%) | 30/40 (75%) | 50/50 (100%) | 30/40 (75%) |
| Recovering/Resolving | 0 | 6/40 (15%) | 0 | 6/40 (15%) | 0 | 6/40 (15%) |
| Not Recovered/Not Resolved | 0 | 0 | 0 | 0 | 0 | 0 |
| Recovered/Resolved w/sequelae | 10/50 (20%) | 4/40 (10%) | 10/50 (20%) | 4/40 (10%) | 10/50 (20%) | 4/40 (10%) |
| Fatal | 0 | 0 | 0 | 0 | 0 | 0 |

<sup>[1]</sup> Subjects may be included in more than one category for 'Event Characteristics'.

Programming note: Please use the AESI list of Guillain-Barre Syndrome; for No. of Events, n, No. of occurrences, outcome and grade counts please follow the AE collapsing rule in the RAP AESI section.

### PPD

Protocol: GSK208466/ADP-04511

Population: Modified Intent-To-Treat (Data as of: 24APR2018)

Table 8.3104

<sup>[2]</sup> Outcome worst case hierarchy: Fatal > Not Recovered/Not Resolved > Recovered/Resolved with sequelae > Recovering/Resolving > Recovered/Resolved

Summary of Characterisics of Guillain-Barre Syndrome (All Infusions)

| | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 2 - 4 | Overall |
|---|---|---|---|---|---|---|
| | (N=200) | (N=100) | (N=200) | (N=100) | Total<br>(N=200) | (N=100) |
| | | · | | | | · |
| Maximum Grade | | | | | | |
| n | 50 | 40 | 50 | 40 | 50 | 40 |
| Grade 1 | 5/50 (10%) | 4/40 (10%) | 5/50 (10%) | 4/40 (10%) | 5/50 (10%) | 4/40 (10%) |
| Grade 2 | 2/50 (4%) | 0 | 2/50 (4%) | 0 | 2/50 (4%) | 0 |
| Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 |
| Grade 4 | 40/50 (80%) | 35/40 (88%) | 40/50 (80%) | 35/40 (88%) | 40/50 (80%) | 35/40 (88%) |

<sup>[1]</sup> Subjects may be included in more than one category for 'Event Characteristics'.

Programming note: Please use the AESI list of Guillain-Barre Syndrome; for No. of Events, n, No. of occurrences, outcome and grade counts please follow the AE collapsing rule in the RAP AESI section.

PPD

Use 8.3104 as a template for the following Table:

Table 8.3105

Summary of Characteristics of Cytokine Release Syndrome (All Infusions)

Table 8.3106

Summary of Characteristics of Cytokine Release Syndrome (All Infusions)

Table 8.3107

<sup>[2]</sup> Outcome worst case hierarchy: Fatal > Not Recovered/Not Resolved > Recovered/Resolved with sequelae > Recovering/Resolving > Recovered/Resolved

208466/ADP-04511

Summary of Characteristics of Recurrent Pancytopenia/Aplastic Anaemia (All Infusions)

Table 8.3108

Summary of Characteristics of Encephalopathy (All Infusions)

Table 8.3109

Summary of Characterisics of Guillain-Barre Syndrome (Second Infusions) Programming note: population: subjects with a second T-cell infusion

Table 8.3110

Summary of Characteristics of Graft versus Host Disease (Second Infusions)

Programming note: population: subjects with a second T-cell infusion

Table 8.3111

Summary of Characteristics of Cytokine Release Syndrome (Second Infusions)

Programming note: population: subjects with a second T-cell infusion

Table 8.3112

Summary of Characteristics of Recurrent Pancytopenia/Aplastic Anaemia (Second Infusions)

Programming note: population: subjects with a second T-cell infusion

Table 8.3113

Summary of Characteristics of Encephalopathy (Second Infusions)

Programming note: population: subjects with a second T-cell infusion

## 208466/ADP-04511


Protocol: GSK208466/ADP-04511 Population: Modified Intent-To-Treat (Data as of: 24APR2018)

Table 8.3114

Summary of Onset and Duration of the First Occurrence of Guillain-Barre Syndrome

| | Cohort 1<br>(N=100) | Cohort 2<br>(N=100) | Cohort 3<br>(N=100) | Cohort 4<br>(N=100) | Cohort 2 - 4<br>Total<br>(N=100) | Overall (N=100) |
|---|---|---|---|---|---|---|
| Number of Subjects with Events | 50 (50%) | 40 (40%) | 50 (50%) | 40 (40%) | 50 (50%) | 40 (40%) |
| Time of onset, days | | | | | | |
| Subjects with event | | | | | | |
| 1-14 | 40 | 40 | 40 | 40 | 40 | 40 |
| 15-28 | 10 | 0 | 10 | 0 | 10 | 0 |
| >28 | 0 | 0 | 0 | 0 | 0 | 0 |
| Mean | 2.5 | 2.1 | 2.5 | 2.1 | 2.5 | 2.1 |
| SD | 1.44 | 1.24 | 1.44 | 1.24 | 1.44 | 1.24 |
| Median | 4 | 3 | 4 | 3 | 4 | 3 |
| Min. | 1 | 1 | 1 | 1 | 1 | 1 |
| Max. | 8 | 5 | 8 | 5 | 8 | 5 |
| Duration, days | | | | | | |
| n | 50 | 40 | 50 | 40 | 50 | 40 |
| 1-5 | 40 (80%) | 40 (100%) | 40 (80%) | 40 (100%) | 40 (80%) | 40 (100% |
| 6-10 | 10 (20%) | 0 | 10 (20%) | 0 | 10 (20%) | 0 |
| >10 | 0 | 0 | 0 | 0 | 0 | 0 |
| Mean | 2.5 | 2.1 | 2.5 | 2.1 | 2.5 | 2.1 |
| SD | 1.44 | 1.24 | 1.44 | 1.24 | 1.44 | 1.24 |
| Median | 4 | 3 | 4 | 3 | 4 | 3 |
| Min. | 1 | 1 | 1 | 1 | 1 | 1 |
| Max. | 8 | 5 | 8 | 5 | 8 | 5 |

Note: Subjects at risk is calculated as the number at risk at the start of the interval.

PPD

Programming note: Please use the AESI list of Guillain-Barre Syndrome; for duration please follow the AE collapsing rule in the RAP AESI section.

Use 8.3114 as a template for the following Table:

Table 8.3115, Table 8.3116, Table 8.3117, Table 8.3118, Table 8.3119, Table 8.3120, Table 8.3121, Table 8.3122 and Table 8.3123

Use 8.3101 as a template for the table 8.3124 (programming note: please use the Comprehensive AESI flag) Use 8.3102 as a template for the table 8.3125 (programming note: please use the Comprehensive AESI flag) Use 8.3103 as a template for the table 8.3126 (programming note: please use the Comprehensive AESI flag) Use 8.3104 as template for the table:

Table 8.3127 Summary of Characteristics of Haematopoietic Cytopenias (Comprehensive List-All Infusions)

Population: mITT

Programming note: please use AESI comprehensive AESI list and use the AESI term "Haematopoietic cytopenias" to report this table.

Use 8.3104 as template for the table:

Table 8.3128 Summary of Characteristics of Haematopoietic Cytopenias (Comprehensive List-Second Infusions)

Population: Subjects with a Second T-Cell Infusion

Programming note: please use AESI comprehensive AESI list and use the AESI term "Haematopoietic cytopenias" to report this table.

Use 8.3114 as a template for the table:

Table 8.3129 Summary of Onset and Duration of the First Occurrence of Haematopoietic Cytopenias (Comprehensive List)

Population: mITT

Programming note: please use AESI comprehensive AESI list and use the AESI term "Haematopoietic cytopenias" to report this table.

### 208466/ADP-04511

Protocol: GSK208466/ADP-04511

Population: Modified Intent-To-Treat


(Data as of: 24APR2018)

Table 8.3201

Time to Resolution of Grade >= 3 Haematopoietic Cytopenias (Comprehensive List)

| | Cohort 1<br>(N=100) | Cohort 2 (N=100) | Cohort 3<br>(N=100) | Cohort 4<br>(N=100) | Cohort 2 - 4<br>Total<br>(N=100) | Overall<br>(N=100) |
|---|---|---|---|---|---|---|
| Number of Subjects with Events | 50 (50%) | 40 (40%) | 50 (50%) | 40 (40%) | 50 (50%) | 40 (40%) |
| Time to Resolution<br>Subjects with event | | | | | | |
| ≤ 28 days | 40 | 40 | 40 | 40 | 40 | 40 |
| 29 days - 3 months | 10 | 0 | 10 | 0 | 10 | 0 |
| > 3 months | 0 | 0 | 0 | 0 | 0 | 0 |

Note: Time to resolution is defined as time from T-cell infusion to the last date of end dates of AESI preferred terms.

Programming note: Please use the comprehensive list AESI term Haematopoietic cytopenias.

#### Use table 8.3201 as a template for the following tables:

Table 8.3202 Time to Resolution of Grade >=3 Recurrent Pancytopenia/Aplastic Anaemia

Population: mITT

Programming note: Please use the focused list AESI term 'Recurrent Pancytopenia/Aplastic Anaemia'

Table 8.3203 Time to Resolution of Grade >=3 Graft versus Host Disease

Population: mITT

Programming note: Please use the focused list AESI term GVHD.

Table 8.3204 Time to Resolution of Grade >= 3 Cytokine Release Syndrome

Population: mITT

Programming note: Please use the focused list AESI term CRS.

208466/ADP-04511


Protocol: GSK208466/ADP-04511

Population: Modified Intent-To-Treat (Data as of: 24APR2018)

Table 8.4101

Change from Baseline to Each Scheduled Visit for Hematology Parameters for the Post-lymphodepletion Period mITT Population

MITTFL = 'Y' and ADLB.PARCAT1 = 'HEMATOLOGY' and ADLB.ANLXXFL = 'Y' (if analysis flag for mean change tables)

| Parameter | | | | | | Cohort 2-4 | |
|---|---|---|---|---|---|---|---|
| Study Visit | | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total | Overall |
| Timepoint | Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Parameter 1 (units) | | | | | | | |
| Day 1 | | | | | | | |
| Baseline | N | X | X | X | X | X | X |
| | Mean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | SD | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| | Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Min,Max | xx.x,xx.x | xx.x,xx.x | xx.x,xx.x | xx.x,xx.x | xx.x,xx.x | xx.x,xx.x |
| Visit | N | Х | х | X | X | Х | Х |
| | Mean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | SD | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| | Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Min,Max | xx.x,xx.x | xx.x,xx.x | xx.x,xx.x | xx.x,xx.x | xx.x, xx.x | xx.x,xx.x |
| Change from Baseline | N | х | х | Х | Х | Χ | X |
| | Mean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | xx.xx |
| | SD | XX.XXX | XX.XXX | XX.XXX | xx.xxx | XX.XXX | XX.XXX |
| | Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Min,Max | XX.X,XX.X | XX.X,XX.X | xx.x,xx.x | xx.x,xx.x | XX.X,XX.X | xx.x,xx.x |

Etc

Continue for remaining scheduled visits

SD = Standard Deviation.

Note: Baseline is within 7 days prior to intitiating lymphodepletion.

File Name: S:\.....\&prog name

## Use 8.4101 as a template for the following Table:

Table 8.4102

Protocol: GSK208466/ADP-04511

Population: Modified Intent-To-Treat


(Data as of: 24APR2018)

Table 8.4201

Shifts from Baseline to Worst Post-Baseline NCI-CTCAE Grade for Hematology Parameters for the Post-lymphodepletion Period mITT Population

SAFFL = 'Y' and ADLB.PARCAT1 = 'HEMATOLOGY' and ADLB.ANLXXFL = 'Y' (if analysis flag for shift tables)

Use ADLB.SHIFT1 for record with LVOTFL = 'Y'. If SHIFT1 is not in dataset, use ADLB.ANRIND and ADLB.BNRIND.

BNRIND contains baseline value, and ANRIND contains End of Treatment Value.

| | | Worst On-Study | Grade | | | |
|---|---|---|---|---|---|---|
| Parameter/ | Baseline | 0 | 1 | 2 | 3 | 4 |
| Cohort | Grade | n/N (%) | n/N (%) | n/N (%) | n/N (%) | n/N (%) |
| arameter 1 | | | | | | |
| Cohort 1 (N=xx) | 0 | x/x ( $xx.x$ ) | x/x ( $xx.x$ ) | x/x ( $xx.x$ ) | x/x (xx.x) | x/x ( $xx.x$ ) |
| | 1 | x/x ( $xx.x$ ) | x/x (xx.x) | x/x (xx.x) | x/x (xx.x) | x/x (xx.x) |
| | 2 | x/x (xx.x) | x/x (xx.x) | x/x (xx.x) | x/x (xx.x) | x/x (xx.x) |
| | 3 | x/x (xx.x) | x/x (xx.x) | x/x (xx.x) | x/x (xx.x) | x/x (xx.x) |
| | 4 | x/x ( $xx.x$ ) | x/x (xx.x) | x/x (xx.x) | x/x (xx.x) | x/x (xx.x) |
| Cohort 2 (N=xx) | 0 | x/x (xx.x) | x/x (xx.x) | x/x (xx.x) | x/x (xx.x) | x/x (xx.x) |
| | 1 | x/x (xx.x) | x/x ( $xx.x$ ) | x/x (xx.x) | x/x (xx.x) | x/x ( $xx.x$ ) |
| | 2 | x/x (xx.x) | x/x ( $xx.x$ ) | x/x ( $xx.x$ ) | x/x (xx.x) | x/x (xx.x) |
| | 3 | x/x ( $xx.x$ ) | x/x ( $xx.x$ ) | x/x ( $xx.x$ ) | x/x ( $xx.x$ ) | x/x ( $xx.x$ ) |
| | 4 | x/x ( $xx.x$ ) | x/x ( $xx.x$ ) | x/x ( $xx.x$ ) | x/x (xx.x) | x/x ( $xx.x$ ) |
| Cohort 3 (N=xx) | 0 | x/x (xx.x) | x/x (xx.x) | x/x (xx.x) | x/x (xx.x) | x/x (xx.x) |
| | 1 | x/x ( $xx.x$ ) | x/x ( $xx.x$ ) | x/x ( $xx.x$ ) | x/x ( $xx.x$ ) | x/x ( $xx.x$ ) |
| | 2 | x/x (xx.x) | x/x ( $xx.x$ ) | x/x (xx.x) | x/x (xx.x) | x/x (xx.x) |
| | 3 | x/x (xx.x) | x/x (xx.x) | x/x (xx.x) | x/x (xx.x) | x/x (xx.x) |
| | 4 | x/x ( $xx.x$ ) | x/x ( $xx.x$ ) | x/x ( $xx.x$ ) | x/x (xx.x) | x/x ( $xx.x$ ) |
| Cohort 4 (N=xx) | 0 | x/x (xx.x) | x/x (xx.x) | x/x (xx.x) | x/x (xx.x) | x/x (xx.x) |
| | 1 | x/x (xx.x) | x/x ( $xx.x$ ) | x/x ( $xx.x$ ) | x/x (xx.x) | x/x (xx.x) |
| | 2 | x/x (xx.x) | x/x ( $xx.x$ ) | x/x ( $xx.x$ ) | x/x (xx.x) | x/x (xx.x) |
| | 3 | x/x (xx.x) | x/x ( $xx.x$ ) | x/x ( $xx.x$ ) | x/x (xx.x) | x/x (xx.x) |
| | 4 | x/x ( $xx.x$ ) | x/x ( $xx.x$ ) | x/x ( $xx.x$ ) | x/x ( $xx.x$ ) | x/x (xx.x) |
| Cohort 2-4 combined (N=xx) | 0 | x/x (xx.x) | x/x (xx.x) | x/x (xx.x) | x/x (xx.x) | x/x (xx.x) |
| | 1 | x/x (xx.x) | x/x ( $xx.x$ ) | x/x ( $xx.x$ ) | x/x (xx.x) | x/x ( $xx.x$ ) |
| | 2 | x/x (xx.x) | x/x ( $xx.x$ ) | x/x ( $xx.x$ ) | x/x (xx.x) | x/x ( $xx.x$ ) |
| | 3 | x/x (xx.x) | x/x ( $xx.x$ ) | x/x ( $xx.x$ ) | x/x (xx.x) | x/x ( $xx.x$ ) |
| | 4 | x/x ( $xx.x$ ) | x/x (xx.x) | x/x (xx.x) | x/x (xx.x) | x/x (xx.x) |

Cohort 1-4 conbined (N=xx)

······· • •

NCI-CTCAE = National Cancer Institute - Common Terminology Criteria for Adverse Events.

Note 1: For n/N, n=number of subjects who meet the criterion, N=number of subjects with both baseline and post-baseline results.

Note 2: Baseline is within 7 days prior to intitiating lymphodepletion.

208466/ADP-04511
File Name: S:\.....\&prog\_name

## Use 8.4201 as a template for the following Table:

Table 8.4202
Shifts from Baseline to Worst Post-Baseline NCI-CTCAE Grade for Chemistry Parameters for the Post-lymphodepletion Period mITT Population

Protocol: GSK208466/ADP-04511

Population: Modified Intent-To-Treat


(Data as of: 24APR2018)

Table 8.4301

Number and Proportion of Subjects with Potentially Clinically Significant Hepatic Post-Baseline Results for the Post-lymphodepletion Period mITT Population

Select records with ADLB.CRITXXFL = 'Y'

| | | | | | | | Cohort 2- | - 4 |
|---|---|---|---|---|---|---|---|---|
| Parameter ADLB.PARAM | Criterion | Statistic | Cohort 1<br>(N=xx) | Cohort 2<br>(N=xx) | Cohort 3<br>(N=xx) | Cohort 4<br>(N=xx) | Total<br>(N=xx) | Overall (N=xx) |
| ALT, AST and BIL<br>Elevations | ( $\geq$ 3xULN AST and/or ALT) and $\geq$ 2xULN BIL | n/N (%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) |
| | ( $\geq$ 3xULN AST and/or ALT) and $\geq$ 1.5xULN BIL | n/N (%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) |
| ALT Elevations | ≥20xULN | n/N (%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) |
| | ≥10xULN | n/N (%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) |
| | ≥5xULN | n/N (%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) |
| | ≥3xULN | n/N (%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) |
| BIL Elevations | >2 xULN | n/N (%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) |
| | >1.5 xULN | n/N (%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) |

ALT = Alanine aminotransferase, AST = Aspartate aminotransferase, BIL = Total bilirubin.

Note 1: Baseline is within 7 days prior to initiating lymphodepletion.

Note 2: For n/N, n=number of subjects who meet the criterion at least once, N=number of subjects with post-baseline results.

# 208466/ADP-04511


(Data as of: 24APR2018)

Protocol: GSK208466/ADP-04511

Population: Modified Intent-To-Treat

Table 8.5001

Maximum Persistence and Time to Maximum Persistence for Responders, Non-Responders, and Overall for the First Infusion

mITT Population

| | | | | | | Cohort 2- | 4 |
|---|---|---|---|---|---|---|---|
| | | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total | Overall |
| Parameter | Statistic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Responders | | | | | | | |
| Maximum Persistence | N | Х | Х | Х | Х | X | Х |
| | Mean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | SD | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| | Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Min,Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Mine to Mariana Brazilatora | N. | | | | | | |
| Time to Maximum Persistence | N | X | X | X | X | X | Х |
| | Mean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | SD | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| | Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Min,Max | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | XX.X,XX.X | xx.x,xx.x |

Maximum Cell Persistence (/µL)

Time to Maximum Cell Persistence (Days)

Maximum Gene marked cells per total lymphocyte

Time to Maximum Gene marked cells per total

lymphocyte (%) (Days)

Repeast for Non-Responders and Overall.

Note 1: Time to maximum persistence is defined as date of maximum persistence for Infusion 1 visits - date of T Cell infusion + 1.

Note 2: Cell Persistence = Absolute peripheral gene-marked cell number/ $\mu$ L = (Psi result number/151515) X (lymphocyte count + monocyte count) X 1000, where Psi is value collected on eCRF.

Note 3: Percent of gene marked cells per total lymphocyte compartment = ((Absolute peripheral gene marked cell number/µL)/Lymphocyte count x 1000)) X 100.

# 208466/ADP-04511

Protocol: GSK208466/ADP-04511

Population: Modified Intent-To-Treat

 (Data as of: 24APR2018)

Table 8.5002

Number and Proportion of RCL Positive Subjects  $\ensuremath{\mathsf{mITT}}$  Population

| | | | | | | Cohort | 2- |
|---|---|---|---|---|---|---|---|
| | Statistic | Cohort 1 (N=xx) | Cohort 2<br>(N=xx) | Cohort 3 (N=xx) | Cohort 4 (N=xx) | 4<br>Total | Overall (N=xx) |
| Parameter | | | | | | (N=xx) | |
| RCL Positive | n/N | xx/XX (xx.x% | ) xx/XX<br>(xx.x%) | xx/XX<br>(xx.x%) | xx/XX (xx.) | ⟨%) xx/XX (xx. | x%) xx/XX (xx.x%) |

Note: n = number of subjects who are RCL positive at any time after initial T Cell infusion, <math>N = number of subjects tested for RCL at least once after initial T Cell infusion.

# 208466/ADP-04511

Protocol: GSK208466/ADP-04511

Population: Modified Intent-To-Treat

 (Data as of: 24APR2018)

Table 8.5003

Number and Percentage of Subjects with Potentially Clinically Significant Post-Baseline Vital Signs Results MITT Population

| | | | | | | | Cohort 2- | 1 |
|---|---|---|---|---|---|---|---|---|
| Parameter | Criterion | Statistic | Cohort 1 (N=xx) | Cohort 2<br>(N=xx) | Cohort 3 (N=xx) | Cohort 4<br>(N=xx) | Total<br>(N=xx) | Overall (N=xx) |
| raramotor | Olicelion . | Deacibeic | (14 222) | (14 122) | (IV ZZZ) | (IV III) | (21 2112) | (14 222) |
| Heart Rate | < 60 bpm | n/N (%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) |
| | > 100 bpm | n/N (%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) |
| Systolic Blood Pressure | >=140 mmHg | n/N (%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) |
| Systolic Blood Pressure | >=140 mmHg | n/N (%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | X | x/xx(%) |
| iastolic Blood Pressure | >=90mmHg | n/N (%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/x |

Note 1: Baseline is within 7 days of initiating lymphodepletion.

Note 2: For n/N, n=number of subjects who meet the criterion at least once, N=number of subjects with post-baseline results.

File Name: S:\.....\&prog name

Protocol: GSK208466/ADP-04511

Population: Modified Intent-To-Treat

Table 8.6101

Summary of ECOG Performance Status at Each Visit

MITT Population

 (Data as of: 24APR2018)

| | | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 2-4 | Overall |
|---|---|---|---|---|---|---|---|
| Jisit/ | | (N=xx) | (N=xx) | (N=xx) | (N=xx) | Total | (N=xx) |
| Score | Statistic | | | | | (N=xx) | |
| Screening | | | | | | | |
| 0 | n/N(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) |
| 1 | n/N(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) |
| 2 | n/N(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) |
| 3 | n/N(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) |
| 4 | n/N(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) |
| 5 | n/N(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) |
| Baseline | | | | | | | |
| 0 | n/N(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) |
| 1 | n/N(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) |
| 2 | n/N(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) |
| 3 | n/N(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) |
| 4 | n/N(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) |
| 5 | n/N(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) |
| T-CELL INFUSIO | N | | | | | | |
| 0 | n/N(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) |
| 1 | n/N(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) |
| 2 | n/N(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) |
| 3 | n/N(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) |
| 4 | n/N(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) |
| 5 | n/N(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) | xx/xx(%) |

ECOG = Eastern Cooperative Oncology Group.

File Name: S:\....\&prog\_name
Protocol: GSK208466/ADP-04511


Population: Modified Intent-To-Treat

(Data as of: 24APR2018)

Figure 17.0001

Note 1: Baseline is within 7 days of initiating lymphodepletion.

Note 2: ECOG Score: 0 - Fully active and able to carry on all pre-disease activities without restriction, 1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light sedimentary nature, 2 - Ambulatory and capable of all self-care but unable to carry out any work activities, 3 - Capable of only limited self-care, 4 - Completely disabled, 5 - Dead.

Maximal Reduction in Sum of Diameters of Target Lesions from Baseline through Progression or Prior to Subsequent Anti-Cancer Therapy for the First Infusion




Protocol: GSK208466/ADP-04511
Population: Modified Intent-To-Treat

Figure 17.0001

Maximal Reduction in Sum of Diameters of Target Lesions from Baseline through Progression or Prior to Subsequent Anti-Cancer Therapy for the First Infusion



Protocol: GSK208466/ADP-04511

Population: Modified Intent-To-Treat

(Data as of: 24APR2018)

Figure 17.0001

Maximal Reduction in Sum of Diameters of Target Lesions from Baseline through Progression or Prior to Subsequent Anti-Cancer Therapy for the First Infusion



Protocol: GSK208466/ADP-04511

Population: Modified Intent-To-Treat

Figure 17.0001


(Data as of: 24APR2018)

Maximal Reduction in Sum of Diameters of Target Lesions from Baseline through Progression or Prior to Subsequent Anti-Cancer Therapy for the First Infusion



Protocol: GSK208466/ADP-04511
Population: Modified Intent-To-Treat (Data as of: 24APR2018)

Figure 17.0002

Maximal Reduction in Sum of Diameters of Target Lesions from the Second Infusion through Progression or Prior to Subsequent Anti-Cancer Therapy



Programming note: for subjects who received 2<sup>nd</sup> infusion report them all together in in graph and if possible mark the corresponding cohort under the subject ID.

Programming note: please also exclude recordes after anti-cancer treatment.


(Data as of: 24APR2018)

Protocol: GSK208466/ADP-04511

Population: Modified Intent-To-Treat

Figure 17.1001

Kaplan-Meier Plot of Progression-Free Survival



Programming note: please plot all KM curves in on graph and provide legend.

Protocol: GSK208466/ADP-04511

Population: Modified Intent-To-Treat

Figure 17.1002

Kaplan-Meier Plot of Overall Survival



Programming note: please plot all KM curves in on graph and provide legend.


Protocol: GSK208466/ADP-04511 Population: Modified Intent-To-Treat

Figure 17.2001

Response Characteristics via RECIST 1.1 and Follow-up

Cohort 1



Programming note: please repeat for cohort 2-4 and add 2<sup>nd</sup> infusion info. (add a symbol for the start timepoint of the 2<sup>nd</sup> infusion.) And also change the X-axis label to Time from the First Tcell Infusion (Weeks); please change "x Surgical Resection" to "x Surgical Resection/Anti-Cancer Therapy" in the lengend and so please also mark the anti-cancer therapy in the plot.

208466/ADP-04511


(Data as of: 24APR2018)

Protocol: GSK208466/ADP-04511

Population: Modified Intent-To-Treat

Figure 17.3001

Boxplots for Peak Expansion by Responders vs. Non-Responders for the First Infusion

Cohort 1



Note: Within each boxplot, the horizontal line is the median and the diamond is the mean.

Protocol: GSK208466/ADP-04511

Population: Modified Intent-To-Treat

Figure 14.4001

Spider Plots for Persistence Results over Time (Truncated at 60 Days) by Responders vs. Non-Responders for the First Infusion Cohort 1



Note: Y-axis is log-transformed. Values below the lower limit of quantitation are set to 1. The R and NR before the subject number indicate responders and non-responders, respectively.

Protocol: GSK208466/ADP-04511

Population: Modified Intent-To-Treat

Figure 17.4002

Spider Plots for Persistence Results over Time (Truncated at 100 Days) by Responders vs. Non-Responders for the First Infusion Cohort 1



Note: Y-axis is log-transformed. Values below the lower limit of quantitation are set to 1. The R and NR before the subject number indicate responders and non-responders, respectively.


Protocol: GSK208466/ADP-04511

Population: Modified Intent-To-Treat

Figure 17.4003

Spider Plots for Persistence Results over Time by Responders vs. Non-Responders for the First Infusion

Cohort 1



Note: Y-axis is log-transformed. Values below the lower limit of quantitation are set to 1. The R and NR before the subject number indicate responders and non-responders, respectively.

Protocol: GSK208466/ADP-04511


Population: Modified Intent-To-Treat

(Data as of: 24APR2018)

Figure 17.4004

Spider Plots of Change from Baseline in Target Lesion through Progression and Prior to Subsequent Anti-Cancer Therapy Over Time by Response Status for the First Infusion

Cohort 1



Note: The R and NR before the subject number indicate responders and non-responders, respectively.

Programming note: please repeat for cohort 2-4. Please also exclude data after anti-cancer therapy (including anti-cancer surgery)

Figure 17.4005: Spider Plots for Persistence Results over Time (Truncated at 60 Days) by Responders vs. Non-Responders for the Second Infusion Programming note: Repeat Figure 17.4001 for subjects who had  $2^{nd}$  infusion. Please report all subjects who received the  $2^{nd}$  infusion from different cohorts in one plot. Responders/non-responders are only for the  $2^{nd}$  infusion period. please also mark the patient cohort in the legend.

### 208466/ADP-04511

Figure 17.4006: Spider Plots for Persistence Results over Time (Truncated at 100 Days) by Responders vs. Non-Responders for the Second Infusion Programming note: Repeat Figure 17.4002 for subjects who had  $2^{nd}$  infusion. Please report all subjects who received the  $2^{nd}$  infusion from different cohorts in one plot. Responders/non-responders are only for the  $2^{nd}$  infusion period. please also mark the patient cohort in the legend.

Figure 17.4007: Spider Plots for Persistence Results over Time by Responders vs. Non-Responders for the Second Infusion

Programming note: Repeat Figure 17.4003 for subjects who had  $2^{nd}$  infusion. Please report all subjects who received the  $2^{nd}$  infusion from different cohorts in one plot. Responders/non-responders are only for the  $2^{nd}$  infusion period. please also mark the patient cohort in the legend.

Figure 17.4008: Spider Plots of Change from Baseline in Target Lesion through Progression and Prior to Subsequent Anti-Cancer Therapy Over Time by Response Status for the Second Infusion

Programming note: Repeat Figure 17.4004 for subjects who had  $2^{nd}$  infusion. Please report all subjects who received the  $2^{nd}$  infusion from different cohorts in one plot. Responders/non-responders are only for the  $2^{nd}$  infusion period. please also mark the patient cohort in the legend.

Protocol: GSK208466/ADP-04511 Population: Modified Intent-To-Treat

Figure 18.5003

Characteristics of CRS Plot for the First Infusion

Cohort 1



Programming note: please repeat for cohort 2-4. Please use the focused scope AESI list. Change the x-axis label to "Time from the First Tcell Infusion (Days)"

208466/ADP-04511

#### Use Figure 18.5003 as a template for the following figures:

Figure 18.5004

Characteristics of CRS Plot for the Second Infusion Population: Subjects with a Second T-Cell Infusion

Programming note: please repeat for cohort 2-4. Please use the focused AESI list. Change the x-axis label to "Time from the Second Tcell Infusion (Days)"

Figure 18.5005

Characteristics of Recurrent Pancytopenia with Bone Marrow Failure/Aplastic Anemia plot for the First Infusion

Population: MITT

Programming note: please repeat for cohort 2-4. Please use the focused AESI list of Recurrent Pancytopenia with Bone Marrow Failure/Aplastic Anemia.

Figure 18.5006

Characteristics of Recurrent Pancytopenia with Bone Marrow Failure/Aplastic Anemia plot for the Second Infusion

Population: MITT

Programming note: please repeat for cohort 2-4. Please use the focused AESI list of Recurrent Pancytopenia with Bone Marrow Failure/Aplastic Anemia. Change the x-axis label to "Time from the Second Tcell Infusion (Days)"

Protocol: GSK208466/ADP-04511


Population: Modified Intent-To-Treat

(Data as of: 24APR2018)

Figure 18.5101

Profile of INF-Gamma by CRS Status and Subject (First Infusion)

Cohort 1



Programming note: please repeat for cohort 2-4. Please use the focused scope AESI list. By CSR (None or Non-Serious CRS vs. Serious CRS) and add legend for start and stop of CRS event. Change color of label for end of event.

# Use Figure 18.5101 as a template for the following figures:

Figure 18.5102

Profile of IL-6 by CRS Status and Subject (First Infusion)

Population: Modified Intent-To-Treat

Figure 18.5103

Profile of IL-8 by CRS Status and Subject (First Infusion)

Population: Modified Intent-To-Treat

Profile of IL-12 by CRS Status and Subject (First Infusion) Population: Modified Intent-To-Treat Figure 18.5105 Profile of IL-13 by CRS Status and Subject (First Infusion) Figure 18.5106 Profile of TNF-Alpha by CRS Status and Subject (First Infusion) Population: Modified Intent-To-Treat Figure 18.5107 Profile of TNF-Gamma by Response and Subject (First Infusion) Population: Modified Intent-To-Treat Programming note: Change the graph tile to "Responder" and "Non-Responder" Figure 18.5108 Profile of IL-6 by Response and Subject (First Infusion) Population: Modified Intent-To-Treat Programming note: Change the graph tile to "Responder" and "Non-Responder" Figure 18.5109 Profile of IL-8 by Response and Subject (First Infusion) Population: Modified Intent-To-Treat Programming note: Change the graph tile to "Responder" and "Non-Responder" Figure 18.5110 Profile of IL-12 by Response and Subject (First Infusion) Population: Modified Intent-To-Treat Programming note: Change the graph tile to "Responder" and "Non-Responder" Figure 18.5111 Profile of IL-13 by Response and Subject (First Infusion) Population: Modified Intent-To-Treat Programming note: Change the graph tile to "Responder" and "Non-Responder" Figure 18.5112 Profile of TNF-Alpha by Response and Subject (First Infusion) Population: Modified Intent-To-Treat Programming note: Change the graph tile to "Responder" and "Non-Responder"

Figure 18.5104


(Data as of: 24APR2018)

Protocol: GSK208466/ADP-04511

Population: Modified Intent-To-Treat

Figure 18.5113

Peak Cytokine Expression of INF-Gamma by CRS Status (First Infusion)

Cohort 1



Programming note: please repeat for cohort 2-4. By CSR (None or Non-Serious CRS vs. Serious CRS).

# Use Figure 18.5113 as a template for the following figures:

Figure 18.5114

Peak Cytokine Expression of IL-6 by CRS Status (First Infusion)

Population: Modified Intent-To-Treat

Figure 18.5115


(Data as of: 24APR2018)

```
Peak Cytokine Expression of IL-8 by CRS Status (First Infusion)
Population: Modified Intent-To-Treat
Figure 18.5116
Peak Cytokine Expression of IL-12 by CRS Status (First Infusion)
Population: Modified Intent-To-Treat
Figure 18.5117
Peak Cytokine Expression of IL-13 by CRS Status (First Infusion)
Population: Modified Intent-To-Treat
Figure 18.5118
Peak Cytokine Expression of TNF-Alpha by CRS Status (First Infusion)
Population: Modified Intent-To-Treat
Figure 18.5119
Peak Cytokine Expression of INF-Gamma by Response (First Infusion)
Population: Modified Intent-To-Treat
Programmingn note: by responder and non-responder. Please change the x-axis labels to "Responder" and "Non-Responder"
Figure 18.5120
Peak Cytokine Expression of IL-6 by Response (First Infusion)
Population: Modified Intent-To-Treat
Programmingn note: by responder and non-responder. Please change the x-axis labels to "Responder" and "Non-Responder"
Figure 18.5121
Peak Cytokine Expression of IL-8 by Response (First Infusion)
Population: Modified Intent-To-Treat
Programmingn note: by responder and non-responder. Please change the x-axis labels to "Responder" and "Non-Responder"
Figure 18.5122
Peak Cytokine Expression of IL-12 by Response (First Infusion)
Population: Modified Intent-To-Treat
Programmingn note: by responder and non-responder. Please change the x-axis labels to "Responder" and "Non-Responder"
Figure 18.5123
Peak Cytokine Expression of IL-13 by Response (First Infusion)
Population: Modified Intent-To-Treat
Programmingn note: by responder and non-responder. Please change the x-axis labels to "Responder" and "Non-Responder"
Figure 18.5124
Peak Cytokine Expression of TNF-Alpha by Response (First Infusion)
Population: Modified Intent-To-Treat
```

Programmingn note: by responder and non-responder. Please change the x-axis labels to "Responder" and "Non-Responder"

Protocol: GSK208466/ADP-04511
Population: Intent-To-Treat

Listing 26.0001 Subject Disposition

208466/ADP-04511

Screening Treatment Informed Informed

Second Second Date Subject Consent Consent Protocol Subject Discontinu-Reason for T-Cell Infusion of ADSL.SUBJID Date Date Version Status \$ ation Date Discontinuation Infusion? Consent Date Death

Cohort: ADSL.ACTARM

Programmer: If reason for discontinuation is 'Protocol Violation' or 'Failed manufacture of cell product', report this as Reason (e.g. Protocol): <specify> where the specify is from SUPPDS.

There are up to 3 Informed Consent Dates: 1) at Screening visit for study, 2) for treatment, and for second infusion. Patient Status will be 'End of Infusion 1' or= 'Infusion 2', depending on when the subject exited the study.

Note: Study Day is relative to the date of the first T cell infusion, which is Study Day 1. \$ Subject Status = 'Infusion 1' or 'Infusion 2', depending on when subject exited the study.

Y = Yes, N = No.
# 208466/ADP-04511

Protocol: GSK208466/ADP-04511
Population: Intent-To-Treat

 (Data as of: 24APR2018)

Listing 26.0002 Study Visits

Cohort Subject Visit Date Reason for ADSL.ACTARM ADSL.SUBJID Visit (Study Day) Unscheduled Visit

Note: Study Day is relative to the date of the first T cell infusion, which is Study Day 1.

208466/ADP-04511

Protocol: GSK208466/ADP-04511

 (Data as of: 24APR2018) Population: Intent-To-Treat

Listing 26.1401

Inclusion and Exclusion Criteria Not Met Prior to Leukapheresis

Criterion Type Cohort Subject Criterion Number ADSL.SUBJID Violated ADSL.ACTARM Violated

Note to programmer: Criterion Type Violated = 'Inclusion' or 'Exclusion'. If all criteria were met, insert statement into listing: 'All subjects met inclusion and exclusion criteria'

Note: Only subjects who did not meet all inclusion/exclusion criteria prior to leukapheresis are listed.

208466/ADP-04511

Protocol: GSK208466/ADP-04511 Population: Intent-To-Treat  (Data as of: 24APR2018)

Listing 26.1403
Protocol Deviations

| | | | Date Of | |
|----|-------------|--------------|-------------|-------------|
| | | | Deviation | |
| Co | phort | Subject | (Study Day) | Description |
| ΑT | OSI. ACTARM | ADSI, SUBJID | DV.DVSTDTC | DV. DVTERM |

Note to programmer: exact layout of the listing will not be known until later. Deviations not collected on eCRF.

Note 1: Study Day is relative to the date of the first T cell infusion, which is Study Day 1.

Note 2: Only subjects with protocol deviations are listed.

208466/ADP-04511

Protocol: GSK208466/ADP-04511 Population: Intent-To-Treat

 (Data as of: 24APR2018)

Listing 26.1101

Demographics and Baseline Characteristics

| | | | | | | Child- | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Cohort | Cohort | Subject | Date of | Age | | Bearing | | Weight | Height | BMI | BSA |
| ADSL.ACTARM | Number | ADSL.SUBJID | Birth | (Years) | Sex | Potetnial? Race | Ethnicity | (kg) | (cm) | (kg/m2) | (m2) |

Strip number from ADSL.ARCMD, this should match number in ACTARM except for subjects with treatment of 'Not Assigned'

Note to programmer: If race is Other, report this as Other: <specify>.

BMI = Body Mass Index (calculated from weight and height), BSA = Body Surface Area (from eCRF).

File Name: S:\.....\&prog name

148

# 208466/ADP-04511

Protocol: GSK208466/ADP-04511 Population: Intent-To-Treat  (Data as of: 24APR2018)

Listing 26.3101 Medical History

MHCAT = 'GENERAL MEDICAL HISTORY'

| | | S:System Organ Class | | | |
|---|---|---|---|---|---|
| | | P:Preferred Term | | End Date | |
| Cohort | Subject | V:Verbatim Term | Start Date | Or Ongoing | Treated? |
| ADSL.ACTARM | ADSL.SUBJID | S: MH.MHBODSYS | MH.MHSTDTC | MH.MHENDTC | |
| | | P: MH.MHDECOD | | Or ONGOING | |
| | | V: MH.MHTERM` | | | |

Note to Programmer: medical history will be coded with MedDRA.

Y = Yes, N = No.

Note 1: Only subjects with medical history reported are listed.

208466/ADP-04511

Population: Intent-To-Treat (Data as of: 24APR2018)

Listing 26.3102

HLA and NY-ESO-1 Antigen

Sample Date for Other Cohort Subject Cancer Testis HLA

ADSL.ACTARM ADSL.SUBJID Antigen Expression HLA-A\*0201 HLA-A\*0205 HLA-A\*0206 Status NY-ESO-1 Status

Note to programmer: The HLA and NY-ESO-1 status in this listing is from the Screening Enrollment CRF and the data is in S.SC.

A subject may have more than one HLA status. If HLA Status is Other, report the <specify> in the Other column. A subject will have only one NY-ESO-1 status.

Y = Yes, N = No.

# 208466/ADP-04511

Protocol: GSK208466/ADP-04511 Population: Intent-To-Treat

Listing 26.2101

Disease Characteristics

 (Data as of: 24APR2018)

Cohort Subject Primary/Original Primary Disease Disease Stage Grade of
ADSL.ACTARM ADSL.SUBJID Diagnosis Date Site at Screening at Screening Histology

MHSTDTC when MHCAT =
'PRIMARY DIAGNOSIS'

Note to programmer: if Disease Stage or Type of Histology is Other, report this as Other:

208466/ADP-04511

Protocol: GSK208466/ADP-04511 Population: Intent-To-Treat  (Data as of: 24APR2018)

Listing 26.4001 Prior Cancer Surgery

Organ - Site Surgery
Cohort Subject of Surgery Description of Surgery Date

ADSL.ACTARM ADSL.SUBJID

N = No, Y = Yes.

Note: Only subjects with prior cancer surgery are listed.

# 208466/ADP-04511

Protocol: GSK208466/ADP-04511 Population: Intent-To-Treat  (Data as of: 24APR2018)

Listing 26.4002

Prior Oncology Treatment

| Subject | Therapy | | Dose | Start | End | |
|---|---|---|---|---|---|---|
| ADSL.SUBJID | Class | Therapy Description | Ordered | Date | Date | Best Response |

Cohort: ADSL.ACTARM

Note to programmer: All prior treatments from CM except for Radiation which is in S.PR

Note: Only subjects reporting prior oncology treatment are listed.

208466/ADP-04511

Protocol: GSK208466/ADP-04511

 (Data as of: 24APR2018) Population: Intent-To-Treat

Listing 28.0001

Dates of Leukapheresis, Lymphodepleting Chemotherapy, and T-Cell Infusion

Cohort Subject Date of Treatment ADSL.ACTARM ADSL.SUBJID Visit Treatment (Study Day)

Note to programmer: Treatment will be Leukapheresis, Lymhodepleting Chemotherapy (list which med was given), or T-Cell

Note: Study Day is relative to the date of the first T cell infusion, which is Study Day 1.

# 208466/ADP-04511

Protocol: GSK208466/ADP-04511 Population: Intent-To-Treat  (Data as of: 24APR2018)

Listing 28.0002

Lymphodepleting Chemotherapy

| Subject | | Date of Med | Start | End | Time | Hospital- | Dose | Infusion |
|---|---|---|---|---|---|---|---|---|
| ADGI GIIR.TID | Medication | (Study Day) | Time | Time | Point | 170d2 # | (ma/m^2) | Duration @ |

Cohort:

Note to Programmers: Include Fludarabine, Cyclophosphamide, and Mesna. Time Point is Pre-CTX or Post-CTX for Mesna.

Note: Study Day is relative to the date of the first T cell infusion, which is Study Day 1.

# For Cyclophosphamide treatment.

@ Duration follows ISO 8601 format. P indicates that the value is a duration, T = Time, H = Hours, M = Minutes, D = Days.

208466/ADP-04511

Protocol: GSK208466/ADP-04511

 Population: Intent-To-Treat (Data as of: 24APR2018)

Listing 28.0003 T Cell Infusion

| | | | | Total | Percent of | | | Vector | = | |
|---|---|---|---|---|---|---|---|---|---|---|
| | T-Cell | | | Cells | Cells | Reason | | Сору | | Reaction |
| Subject | Infusion Date | Start Time/ | Total Cell | Transduced | Infused | Whole Bag | Duration | Number | Lot Number | To |
| ADSL.SUBJID | (Study Day) | End Time | Dose (x10^9) | $(x10^9)$ | (응) # | Not Infused # | of Infusion | (copies) | (PCT Unit #) | Infusion? |
| EXADJ | ECDUR or | | | | | | | | | |

Cohort: EXDUR

 $<sup>\</sup>overline{Y} = Yes, N = No.$ 

Note 1: Only subjects who received T Cell Infusion are listed.

Note 2: Study Day is relative to the date of the first T cell infusion, which is Study Day 1.

<sup>#</sup> If whole bag was not infused.

208466/ADP-04511

Protocol: GSK208466/ADP-04511  (Data as of: 24APR2018) Population: Intent-To-Treat

Listing 27.0001

Lesion Measurements and Assessments by RECIST v1.1

ADTRREC.

PCHG for SDIAM for BASETYPE =

PARAMCD= SDIAM

TRTESTCD =

NADIR 1

Sum of

Short Longest

TR.TRDTC TR. Assessment

Visit (Study Day)

TRVISIT Date

Lesion Method ID \$

Tumor Organ Site Type

Criterion TRTESTCD=

Diameter (mm)

Longest

Axis Diameter (mm) (mm)

% Change From Baseline from Nadir

% Change

Assessment @

Cohort:

Subject

TRMETHOD TRLNKID

SUPPTU.SITE TRCAT TRGRPID

T.D.T.A.M

PCHG for TRTESTCD=

SDIAM for

TR.TUMSTATE

TULOC

SAXTS

BASETYPE =

PRETREATMENT BASELINE 1

Organ, Site, Sum of Longest Diameter and Sum of Short Axis only occur for first row per subject per visit. Tumor Type is Index, Non-Index, Target, Target Nodal, Non-Target, and New. Criterion is IRRC or RECIST v1.1. Assessment is Tumor State.

ND = Not Done.

Note 1: Study Day is relative to the date of the first T cell infusion, which is Study Day 1.

Note 2: Sum of Longest Diameter is sum of the longest diameter for non-nodal lesions and short axis for nodal lesions. Sum of Short Axis is sum of the short axis for all nodal lesions.

Note 3: Listing includes subjects who received at least one T cell infusion.

@ Assessment was performed by investigator and applies to Non-target lesions and New lesions.

\$ T = Target lesion, NT = Non-target lesion, NEW = New lesion.

208466/ADP-04511

Protocol: GSK208466/ADP-04511  Population: Intent-To-Treat (Data as of: 24APR2018)

Listing 27.0003

Response Assessments and Overall Response by RECIST v1.1 for the First Infusion

| | | Date of<br>T Cell | Assessment<br>Date | Target<br>Lesion | Non-Target<br>Lesion | New | Visit E |
|---|---|---|---|---|---|---|---|
| Subject | Visit | Infusion | (Study Day) | Evaluation | Evaluation | Lesions? | Response Res |
| ADSL.SUBJID | TRTSDT ADT | AVALC | AVALC AVALC AVALC | | | | * |
| Cohort: | | for | for for for | | | | |

for for for TRGRESP NTRGRESP NEWLES VISRESP

Y = Yes, N = No, PD = Progressive Disease, SD = Stable Disease, NE = Not Evaluable, CR = Complete Response, PR = Partial Response. RECIST = Response Evaluation Criteria in Solid Tumors.

Note 1: Study Day is relative to the date of the first T cell infusion, which is Study Day 1.

Note to programmer: Put 'ND' under Assessment Date if tumor was NOT assessed on a visit.

Note 2: Evaluation of target and non-target lesions does not take into account the presence of new lesions.

The overall response does take new lesions into account.

Note 3: Subject PPD had a Day 3 assessment of PD that was not used in derivation of Best Overall Response.

208466/ADP-04511

#### Use Template for Listing 27.0003 for

#### Listing 27.0004

#### Response Assessments and Overall Response by RECIST v1.1 Following a Second T Cell Infusion

(Programming note: Please use the following footnotes:

Y = Yes, N = No, PD = Progressive Disease, SD = Stable Disease, NE = Not Evaluable, CR = Complete Response, PR = Partial Response.

RECIST = Response Evaluation Criteria in Solid Tumors.

Note 1: Listing includes only subjects who had a second T cell infusion.

Note 2: 1st Study Day is relative to the date of the first T cell infusion, 2nd study day is relative to date of the second T cell infusion.)

208466/ADP-04511

Protocol: GSK208466/ADP-04511  Population: Intent-To-Treat

(Data as of: 24APR2018)

Listing 27.0005

Investigator RECIST v1.1 Response Assessments and Overall Response for the First Infusion

| Date of Assessment | Target | Non-Target | | Visit | Best |
|---|---|---|---|---|---|
| T Cell Date | Lesions | Lesions | New | Overall | Overall |
| Subject Visit Infusion (Study Day) | Evaluation | Evaluation | Lesions? | Response | Response |

ADSL.SUBJID TRTSDT ADT AVALC AVALC AVALC AVALC Cohort: for for for for TRGRESP NTRGRESP NEWLES VISRESP

Note to programmer: Put 'ND' under Assessment Date if tumor was NOT assessed on a visit.

Y = Yes, N = No, PD = Progressive Disease, SD = Stable Disease, NE = Not Evaluable, CR = Complete Response, PR = Partial Response.

RECIST = Response Evaluation Criteria in Solid Tumors.

Note 1: Listing includes subjects who received at least one T cell infusion. Note 2: Study Day is relative to the date of the first T cell infusion, which is Study Day 1.

Note 3: Subjects PPD received anti-cancer therapy on PPD

File Name: S:\.....\&prog name

Use Template for Listing 27.0005 for

#### Listing 27.00051

#### Investigator RECIST v1.1 Response Assessments and Overall Response Following a Second T Cell Infusion

Programming note: Please using the following footnotes:

Y = Yes, N = No, PD = Progressive Disease, SD = Stable Disease, NE = Not Evaluable, CR = Complete Response, PR = Partial Response.

RECIST = Response Evaluation Criteria in Solid Tumors.

Note 1: Listing includes only subjects who had a second T cell infusion.

Note 2: 1st Study Day is relative to the date of the first T cell infusion, 2nd study day is relative to date of the second T cell infusion.

208466/ADP-04511

Protocol: GSK208466/ADP-04511

Population: Intent-To-Treat

(Data as of: 24APR2018)

Listing 27.0007

Progression-Free Survival and Overall Survival

ADTTEREC.PARAMCD = 'PFS' for Reason for PD, Death, Date of PD/Death, Progression-Free Survival.

ADTTEREC.PARAMCD = 'OS' for Date of Death or Censoring and Overall Survival

| | | Date of | | Reason | Date of PD/Death | Progression- | Date of Death | Overall |
|---|---|---|---|---|---|---|---|---|
| | | T cell | | For | or Censoring | Free Survival | or Censoring | Survival |
| Cohort | Subject | Infusion | PD? | PD | (Study Day) | (Weeks) | (Study Day) | (Weeks) |
| | | TRTSDT | Y/N | | ADT, ADY | AVAL | ADT, ADY | AVAL |

Y if CNSR = 0 N if CNSR = 1

From ADTTEREC

Note to programmer: there may be multiple reasons for PD. Each can go on a different row. These will be Increased Tumor Burden, Surgical Resection, Prohibited Medications

N = No, Y = Yes, OS = Overall Survival PFS = Progression-Free Survival, PD = Progressive Disease.

Note 1: PFS is defined as the interval between the date of first T cell infusion and the earliest documented evidence of disease progression or death due to any cause or surgical resection or start of prohibited medications. Subjects who do not have a documented date of progression, death, surgical resection, or prohibited medication are censored at the date of last assessment.

Note 2: OS is defined as the interval between the date of first T cell infusion and date of death from any cause. Subjects who are still alive or who are lost to follow-up are censored at the date of last contact.

Note 3: Study Day is relative to the date of the first T cell infusion, which is Study Day 1.

Note 4: Listing includes subjects who received at least one T cell infusion.

Protocol: GSK208466/ADP-04511
Population: Intent-To-Treat
(Data as of: 24APR2018)

Listing 27.0008

Time to Confirmed Response, Duration of Response, and Duration of Stable Disease, and Best Overall Response Note: one row per subject.

| | | | ADT for ADRSREC. PARAMCD = 'RSPSTUS' | | | |
|---|---|---|---|---|---|---|
| | | AVALC for | When AVALC = | | | |
| | | ADRSREC. | 'RESPONDER' | | | |
| | | PARAMCD = | And DTYPE = | | | |
| | | 'BESTRESP' | 'INFUSION 1 | AVAL for | AVAL for | |
| | | And DTYPE = | RESPONSE' | ADTTEREC.PARAMCD | ADTTEREC.PARAMCD | |
| | | 'INFUSION 1 | Date of | = 'TTR' and | = 'DOR' and | AVAL for ADTTEREC.PARAMCD |
| | | RESPONSE' | Confirmed | CNSR = 0. | CNSR = 0. | = 'DOSD' and |
| | | Best | Response | Time to | Duration of Response | CNSR = 0. |
| | Date of T Cell | Overall Response | (CR or PR) | Response | (DOR) | Duration of Stable Disease |
| Cohort Subject | Infusion | (BOR) | (Study Day) | (Weeks) | (Weeks) | (Weeks) |
| · | TRTSDT | CR, PR, SD, PD, | | | | |
| | | NE | | | | |

Programming Note: Subjects who do not have confirmed response of CR or PR will not have values for Date of Confirmed Response, Time to Response. Duration of Response.

#### From ADRSREC and ADTTEREC

BOR = Best Overall Response, CR = Complete Response, DOR = Duration of Response, PD = Progressive Disease, PR = Partial Response, NE = Not Evaluable, SD = Stable Disease, TTR = Time to Response.

Note 1: TTR is defined as the interval between the date of first T-cell infusion and the earliest date of first documented confirmed CR or confirmed PR among participants with a confirmed PR or CR.

Note 2: Duration of response is defined as the time from first documented evidence of confirmed CR or PR until first documented date of disease progression or death due to any cause or surgical resection or start of prohibited medications. Responders who are still alive and who do not have documented disease progression, surgical resection, or prohibited medication are censored at the date of the last assessment.

Note 3: Listing includes subjects who received at least one T-cell infusion.

Note 4: Study Day is relative to the date of the first T cell infusion, which is Study Day 1.

Note 5: Duration of response or duration of stable disease with a "+" sign means the subject did not have documented disease progression.

 (Data as of: 24APR2018)

Listing 28.1001

Adverse Events for First T Cell Infusion

| Subject | S:System Organ Class<br>P:Preferred Term | Start Date | End Date<br>(Study Day) | Serious?/ | Reason<br>Serious @ Toxicity @ | Relationship<br>Grade to T Cell | Action Taker with T Cell | Other<br>Action | |
|---|---|---|---|---|---|---|---|---|---|
| ADSL.SUBJID | V:Verbatim Term | (Study Day) | or Ongoing | Pre? # | \$ | Infusion | Infusion | Taken | Outcome |
| | | | ADAE.AEENDTC | | | | | | |
| Cohort: | ADAE.AEBODSYS | | (ADAE.AEENDY) | ADAE.TRTEMFL | | ADAE.AEREL | | | ADAE.AEOUT |
| ADSL.ACTARM | ADAE.AEDECOD | ADAE.AESTDTC | | ADAE.AESER | | | ADAE.AEACN | | |
| | ADAE AETERM | (ADAE.AESTDY) | | | | | | | |

Note 1: Only subjects with adverse events are listed. Includes all adverse events from date of informed consent through end of study or start of lymphodepletion for second T cell infusion, whichever is earlier.

Note 2: Study Day is relative to the date of the first T cell infusion, which is Study Day 1.

Note 3: Adverse events are graded using NCI CTCAE Version 4.03.

<sup>#</sup> If Serious = 'Y' and the AE started prior to leukapheresis, response to Pre? = 'Y'. Otherwise, response to Pre is missing.

<sup>@</sup> DE = Death, DI = Disability, CA = Congenital Anomaly, LF = Life Threatening, HO = Hospitalization, MS = Medically Significant Event.

<sup>\$ &#</sup>x27;C' after the toxicity grade indicates a change in severity.

## 208466/ADP-04511

Protocol: GSK208466/ADP-04511 Population: Intent-To-Treat  (Data as of: 24APR2018)

Listing 28.1002

Adverse Events for Second T-Cell Infusion

| | S:System Organ Cla | ss Start Date | End Date | | Reason | | Relationship | Action Taken | Other | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject | P:Preferred Term | (Study Day 1/ | (Study Day) | | Serious | Toxicity | to T Cell | with T Cell | Action | |
| ADSL.SUBJID | V:Verbatim Term | Study Day 2) | or Ongoing | Serious? | @ | Grade \$ | Infusion | Infusion | Taken | Outcome |
| | | | ADAE.AEENDTC | | | | | | | |
| Cohort: | ADAE.AEBODSYS | | (ADAE.AEENDY) | ADAE.TRTEMFL | | | ADAE.AEREL | | | ADAE.AEOUT |
| ADSL.ACTARM | ADAE.AEDECOD | ADAE.AESTDTC | | ADAE.AESER | | | | ADAE.AEACN | | |
| | ADAE.AETERM | (ADAE.AESTDY) | | | | | | | | |

#### Note to Programmer:

Note 1: Only subjects with adverse events are listed. Includes all adverse events beginning with start of lymphodepletion for second T cell infusion.

Note 2: 1st Study Day is relative to the date of the first T cell infusion, 2nd study day is relative to date of the second T cell infusion.

Note 3: Adverse events are graded using NCI CTCAE Version 4.03.

@ DE = Death, DI = Disability, CA = Congenital Anomaly, LF = Life Threatening, HO = Hospitalization, MS = Medically Significant Event.

\$ 'C' after the toxicity grade indicates a change in severity.

File Name: S:\.... \&prog name

Protocol: GSK208466/ADP-04511 Population: Intent-To-Treat

Listing 28.1003

Adverse Events with CTCAE Grade 3 or Higher

 (Data as of: 24APR2018)

| Subject | S:System Organ Class<br>P:Preferred Term | Start Date<br>(Study Day)/ | End Date<br>(Study Day) | Serious?/ | Reason<br>Serious @ Toxicity | Relationship<br>Gradeto T Cell | Action Taker<br>with T Cell | | |
|---|---|---|---|---|---|---|---|---|---|
| ADSL.SUBJID | V:Verbatim Term | Infusion | or Ongoing | Pre? # | \$ | Infusion | Infusion | Taken | Outcome |
| | | | ADAE.AEENDTC | | | | | | |
| Cohort: | ADAE.AEBODSYS | | (ADAE.AEENDY) | ADAE.TRTEMFL | | ADAE.AEREL | | | ADAE.AEOUT |
| ADSL.ACTARM | ADAE.AEDECOD | ADAE.AESTDTC | | ADAE.AESER | | | ADAE.AEACN | | |
| | ADAE.AETERM | (ADAE.AESTDY) | | | | | | | |

Note to programmers: Infusion is First or Second. If there are no values for a column, omit the column.

Note 1: Only subjects with adverse events with toxicity grade of 3 or more are listed.

Note 2: Study Day is relative to the date of the first T cell infusion, which is Study Day 1.

Note 3: Adverse events are graded using NCI CTCAE Version 4.03.

<sup>#</sup> If Serious = 'Y' and the AE started prior to leukapheresis, response to Pre? = 'Y'. Otherwise, response to Pre is missing.

<sup>@</sup> DE = Death, DI = Disability, CA = Congenital Anomaly, LF = Life Threatening, HO = Hospitalization, MS = Medically Significant Event.

<sup>\$ &#</sup>x27;C' after the toxicity grade indicates a change in severity.

 (Data as of: 24APR2018)

Listing 28.2001

Serious Adverse Events

| Subject | S:System Organ Class<br>P:Preferred Term | Start Date<br>(Study Day) | End Date<br>(Study Day) | Serious?/ | Reason<br>Serious @ Toxicity | Relationship<br>Gradeto T Cell | Action Taken with T Cell | Other<br>Action | |
|---|---|---|---|---|---|---|---|---|---|
| ADSL.SUBJID | V:Verbatim Term | Infusion | or Ongoing | Pre? # | \$ | Infusion | Infusion | Taken | Outcome |
| | | | ADAE.AEENDTC | | | | | | |
| Cohort: | ADAE.AEBODSYS | | (ADAE.AEENDY) | ADAE.TRTEMFL | | ADAE.AEREL | | | ADAE.AEOUT |
| ADSL.ACTARM | ADAE.AEDECOD | ADAE.AESTDTC | | ADAE.AESER | | | ADAE.AEACN | | |
| | ADAE.AETERM | (ADAE.AESTDY) | | | | | | | |

Note to programmers: Infusion is First or Second.

Note 1: Only subjects with serious adverse events are listed.

Note 2: Study Day is relative to the date of the first T cell infusion, which is Study Day 1.

Note 3: Adverse events are graded using NCI CTCAE Version 4.03.

<sup>#</sup> If the SAE started prior to leukapheresis, response to Pre? = 'Y'. Otherwise, response to Pre is missing.

<sup>@</sup> DE = Death, DI = Disability, CA = Congenital Anomaly, LF = Life Threatening, HO = Hospitalization, MS = Medically Significant Event.

<sup>\$ &#</sup>x27;C' after the toxicity grade indicates a change in severity.

 (Data as of: 24APR2018)

Listing 28.3001

Cytokine Release Syndrome (CRS)

| Subject | S:System Organ Class<br>P:Preferred Term | Start Date<br>(Study Day)/ | End Date<br>(Study Day) | Serious?/ | Reason<br>Serious @ Toxicity | Relationship<br>Gradeto T Cell | Action Taker<br>with T Cell | | |
|---|---|---|---|---|---|---|---|---|---|
| ADSL.SUBJID | V:Verbatim Term | Infusion | or Ongoing | Pre? # | \$ | Infusion | Infusion | Taken | Outcome |
| | | | ADAE.AEENDTC | | | | | | |
| Cohort: | ADAE.AEBODSYS | | (ADAE.AEENDY) | ADAE.TRTEMFL | | ADAE.AEREL | | | ADAE.AEOUT |
| ADSL.ACTARM | ADAE.AEDECOD | ADAE.AESTDTC | | ADAE.AESER | | | ADAE.AEACN | | |
| | ADAE.AETERM | (ADAE.AESTDY) | | | | | | | |

Note to programmers: Infusion is First or Second. List of preferred terms to include is in Appendix 2 of SAP.

Note 1: Only subjects with adverse events coded to the MedDRA PT cytokine release syndrome or cytokine storm are listed.

Note 2: Study Day is relative to the date of the first T cell infusion, which is Study Day 1.

Note 3: Adverse events are graded using NCI CTCAE Version 4.03.

<sup>#</sup> If Serious = 'Y' and the AE started prior to leukapheresis, response to Pre? = 'Y'. Otherwise, response to Pre is missing.

<sup>@</sup> DE = Death, DI = Disability, CA = Congenital Anomaly, LF = Life Threatening, HO = Hospitalization, MS = Medically Significant Event.

<sup>\$ &#</sup>x27;C' after the toxicity grade indicates a change in severity.

 (Data as of: 24APR2018)

Listing 28.3002

Graft Versus Host Disease (GVHD)

| Subject | S:System Organ Class<br>P:Preferred Term | Start Date<br>(Study Day)/ | End Date<br>(Study Day) | Serious?/ | Reason<br>Serious @ Toxicity ( | Relationship<br>Gradeto T Cell | Action Taken with T Cell | Other<br>Action | |
|---|---|---|---|---|---|---|---|---|---|
| ADSL.SUBJID | V:Verbatim Term | Infusion | or Ongoing | Pre? # | \$ | Infusion | Infusion | Taken | Outcome |
| | | | ADAE.AEENDTC | | | | | | |
| Cohort: | ADAE.AEBODSYS | | (ADAE.AEENDY) | ADAE.TRTEMFL | | ADAE.AEREL | | | ADAE.AEOUT |
| ADSL.ACTARM | ADAE.AEDECOD | ADAE.AESTDTC | | ADAE.AESER | | | ADAE.AEACN | | |
| | ADAE.AETERM | (ADAE.AESTDY) | | | | | | | |

Note to programmers: Infusion is First or Second. List of preferred terms to include is in Appendix 2 of SAP.

File Name: S:\.....\&prog name

Programming note:

Use Listing 28.3001 template for:

Listing 28.3003 Recurrent pancytopenia with bone marrow failure/Aplastic anemia

Listing 28.3004 Guillain-Barre syndrome

Listing 28.3005 Encephalopathy syndrome

Note 1: Only subjects with adverse events coded to the MedDRA PT terms associated with GVHD are listed.

Note 2: Study Day is relative to the date of the first T cell infusion, which is Study Day 1.

Note 3: Adverse events are graded using NCI CTCAE Version 4.03.

<sup>#</sup> If Serious = 'Y' and the AE started prior to leukapheresis, response to Pre? = 'Y'. Otherwise, response to Pre is missing.

<sup>@</sup> DE = Death, DI = Disability, CA = Congenital Anomaly, LF = Life Threatening, HO = Hospitalization, MS = Medically Significant Event.

<sup>\$ &#</sup>x27;C' after the toxicity grade indicates a change in severity.

208466/ADP-04511

Protocol: GSK208466/ADP-04511
Population: Intent-To-Treat

 (Data as of: 24APR2018)

Listing 28.3101

Hematology Evaluations - Part 1

Collection Date

Subject Visit (Study Day)

ADSL.SUBJID LB.VIIST LB.LBDTC (LB.LBDY)

Parameter1 (unit) (unit) Parameter3 (unit) Parameter4 (unit) Parameter5 (unit) Parameter5 (unit)

Cohort:

LB.LBSTRESC concatenated with LB.LBNRIND for 'L' or 'H' for each LBTESTCD

ADSL.ACTARM

Notes to programmer: If sample not collected, put ND under Collection Date. If test is not done on a parameter on a certain visit put ND as result corresponding to that parameter on that visit. Listing includes Coagulation parameters

List L or H for values outside the reference range. LB.LBNRIND

Include as many parts as needed to accommodate all parameters. If multiple parts, numbering will be 28.3101, 28.3102, etc.

ND = Not Done.

L = Below lower limit of laboratory reference range, H = Above upper limit of laboratory reference range. Note: Study Day is relative to the date of the first T cell infusion, which is Study Day 1.

File Name: S:\.....\&prog name

Programming note:

Use Listing 28.3101 template for: Listings 28.3111, 28.3121.

208466/ADP-04511

Protocol: GSK208466/ADP-04511 Population: Intent-To-Treat

Listing 28.3131

Clinically Significant Hematology Findings

 (Data as of: 24APR2018)

Collection Date Parameter Reference
Subject ADSL.SUBJID Visit (Study Day) (unit) Result Range

LB.VISIT LB.LBDTC (LB.LBDY)

Cohort: ADSL.ACTARM

Note to programmer: Include only clinically significant values.

L = Below lower limit of laboratory reference range, H = Above upper limit of laboratory reference range.

Note: Study Day is relative to the date of the first T cell infusion, which is Study Day 1.

File Name: S:\.....\&prog name

Protocol: GSK208466/ADP-04511


Population: Modified Intent-To-Treat

(Data as of: 24APR2018)

Listing 28.3132

Listing of Subjects with Potentially Clinically Significant Hepatic Post-Baseline Results for the Post-lymphodepletion Period

mITT Population

Collection
Date/Time

Criterion Cohort Subject Visit (Study Day) Parameter Value

(≥3xULN AST and/or ALT) and ≥2xULN BIL

208466/ADP-04511

.

ALT = Alanine aminotransferase, AST = Aspartate aminotransferase, BIL = Total bilirubin.

Note 1: Baseline is within 7 days of initiating lymphodepletion.

Note 2: Study Day is relative to the day of the first T Cell infusion (Day 1).

File Name: S:\.....\&prog\_name

Programming Note: List all of a subject's values for parameters listed in the criterion if a subject meets criterion for at least one visit.

# 208466/ADP-04511

Protocol: GSK208466/ADP-04511 Population: Intent-To-Treat

Listing 28.3201

Clinical Chemistry Evaluations - Part 1

 (Data as of: 24APR2018)

Same template as Listing 28.3101

Note to Programmer: Include as many Parts as needed to accommodate all parameters. If multiple parts, numbering will be 28.3202, 28.3203 etc.

File Name: S:\.....\&prog name

Programming note:

Use Listing 28.3201 template for Listings 28.3211, 28.3221.

208466/ADP-04511

Protocol: GSK208466/ADP-04511
Population: Intent-To-Treat

(Data as of: 24APR2018)

Listing 28.3231

Clinically Significant Clinical Chemistry Findings

Same template as Listing 28.3131

File Name: S:\.....\&prog\_name

173

208466/ADP-04511

Protocol: GSK208466/ADP-04511
Population: Intent-To-Treat

(Data as of: 24APR2018)

Listing 28.3301

Urinalysis Evaluations - Part 1

Same template as Listing 28.3101

Note to Programmer: Include as many Parts as needed to accommodate all parameters. If multiple parts, numbering will be 28.3302, 28.3303 etc.

File Name: S:\....\&prog\_name

Programming note:

Use Listing 28.3301 template for: Listings28.3311, 28.3321.

208466/ADP-04511

Protocol: GSK208466/ADP-04511
Population: Intent-To-Treat

(Data as of: 24APR2018)

Listing 28.3331

Clinically Significant Urinalysis Findings

Same template as Listing 28.3131

208466/ADP-04511

Protocol: GSK208466/ADP-04511
Population: Intent-To-Treat

 (Data as of: 24APR2018)

Listing 28.3341

Additional Laboratory Assessments

Collection Date Rheumatoid TSH T3 T4

Cohort Subject Visit (Study Day) ANA Factor (units) (units)

Notes to programmer: If all of the tests are not done on a visit, put 'ND' under Collection Date for that visit. If a particular test is not done on a visit, put 'ND' under that test for that visit.

ND = Not Done.

Note: Study Day is relative to the date of the first T cell infusion, which is Study Day 1.

208466/ADP-04511

Protocol: GSK208466/ADP-04511
Population: Intent-To-Treat

(Data as of: 24APR2018)

Listing 28.3342

Clinically Significant Additional Laboratory Findings

Same template as Listing 28.3131

208466/ADP-04511


(Data as of: 24APR2018)

Protocol: GSK208466/ADP-04511
Population: Intent-To-Treat

Listing 28.3343

Renal Function Findings

LBSP.TESTCD = CREATEXR LBSP.TESTCD = Creatinine Clearance CREATCLR LBSP.TESTCD = Creatinine Excretion EDTACLR Collection Date Clearance Rate EDTA GFR Cohort Subject Visit (Study Day) (mL/min) (g/day) (mL/min)

LBSP.LBCAT = 'RENAL FUNCTION TEST' Notes to programmer: If all of the tests are not done on a visit, put 'ND' under Collection Date for that visit. If a particular test is not done on a visit, put 'ND' under that test for that visit.

ND = Not Done.

Note: Study Day is relative to the date of the first T cell infusion, which is Study Day 1.

208466/ADP-04511

Protocol: GSK208466/ADP-04511

 (Data as of: 24APR2018) Population: Intent-To-Treat

Listing 28.4001

Replication Competent Lentivirus (RCL)

Collection Date (Study

Cohort Subject Visit Result

Notes to programmer: If test are not done on a visit, put 'ND' under Collection Date for that visit. Data to come from vendor.

ND = Not Done.

Note: Study Day is relative to the date of the first T cell infusion, which is Study Day 1.


(Data as of: 24APR2018)

Protocol: GSK208466/ADP-04511

Population: Modified Intent-To-Treat

Listing 28.4002 Persistence

| Cohort Subject Visi | Collection<br>Date<br>it (Study Day) | Result # (copies/mcg DNA) | Lymphocytes (10^9/L) | Monocytes<br>(10^9/L) | Cell<br>Persistence \$ | % Gene Marked<br>Cells per<br>Lymphocyte & | Coefficient<br>of<br>Variation/<br>Number of<br>Possitive<br>Replicates | | Peak Persistence/ Time to Peak Persistence (Days) | Time to 25% Loss of<br>Peak Persistence<br>(Days) / 50% / 75%<br>/ Duration of<br>Detectable<br>Persistence |
|---|---|---|---|---|---|---|---|---|---|---|
| Cohort 1 200 Baseli | ne 010CT2012(- | -28)50.55 | 0.02 | 0.02 | 0.1234546 | 0.364748 | N/A/<br>1 | NEGATIVE | 586978.1/<br>2 | 3/<br>14/ |
| | | | | | | | | | | 14/<br>28+ |

Notes to programmer: If test are not done on a visit, put 'ND' under Collection Date for that visit. There is a pre-infusion sample on Day 0. Need to map data

ND = Not Done.

Note: Study Day is relative to the date of the first T cell infusion, which is Study Day 1.

<sup>#</sup> As collected on eCRF.

<sup>\$</sup> Cell Persistence = Absolute peripheral gene-marked cell number/ $\mu L$  = (Psi result number/151515) x (lymphocyte count + monocyte count) x 1000, where Psi is value collected on eCRF.

<sup>&</sup>amp; Percent of gene marked cells per total lymphocyte compartment = ((Absolute peripheral gene marked cell number/ $\mu$ L)/Lymphocyte count x 1000)) x 100.
208466/ADP-04511

Protocol: GSK208466/ADP-04511

 Population: Intent-To-Treat (Data as of: 24APR2018)

Listing 28.4101 Cytokines - Part 1

T Cell

Infusion Collection Date Time Cohort Subject Visit Timepoint Dates (Study Day) Point Param 1 Param 2 Etc.

Notes to programmer: If test are not done on a visit, put 'ND' under Collection Date for that visit. There is a pre-infusion sample on Day 0. Subjects with an AE of CRS will have # after their subject number.

Note to Programmer: Include as many Parts as needed to accommodate all parameters. If multiple parts, numbering will be 28.4102, 28.4103 etc. Data will come from vendor

ND = Not Done.

Note: Study Day is relative to the date of the first T cell infusion, which is Study Day 1. # Subject has an adverse event of cytokine release syndrome (CRS).

File Name: S:\.....\&prog name

Porgramming note:

Repeat Listing 28.4101 format for Listing 28.4102.

208466/ADP-04511

Protocol: GSK208466/ADP-04511 Population: Intent-To-Treat  (Data as of: 24APR2018)

Listing 28.4201

Biopsy-Tumor Antigen Results

Cohort Subject Visit Collection Date (Study Type of Media of Any Antigen Date of Antigen Sample Storage Expression? Expression

ND = Not Done.

Note: Study Day is relative to the date of the first T cell infusion, which is Study Day 1.

208466/ADP-04511

Protocol: GSK208466/ADP-04511

 Population: Intent-To-Treat (Data as of: 24APR2018)

Listing 28.4301 Flow Cytometry

T Cell

Infusion Collection Date Subject Visit Dates (Study Day) Cohort

ND = Not Done.

Note: Study Day is relative to the date of the first T cell infusion, which is Study Day 1.

208466/ADP-04511

Protocol: GSK208466/ADP-04511 Population: Intent-To-Treat  (Data as of: 24APR2018)

Listing 28.5001

Pregnancy Test Results

Date Performed

Cohort Subject Visit (Study Day) Specimen Type Result

Notes to programmer: If pregnancy test not performed, put ND under Date Performed.

Result = Positive or Negative.

ND = Not Done.

Note: Study Day is relative to the date of the first T cell infusion, which is Study Day 1.

### 208466/ADP-04511

Protocol: GSK208466/ADP-04511 Population: Intent-To-Treat  (Data as of: 24APR2018)

Listing 28.5101 Vital Signs

| Subject<br>ADSL.SUBJID | Visit | Date/Time<br>Performed<br>(Study Day) | ) Time-poin | Blood Pressure<br>Systolic/Diastolic<br>t (mmHg) | Pulse<br>Rate<br>(bpm) | Temperature (C) | Respiratory Rate<br>(Breaths/min) | e Weight<br>(kg) | BSA<br>(m^2) | Oxygen<br>Saturation<br>(%) |
|---|---|---|---|---|---|---|---|---|---|---|
| | VS.VISIT | VS.VSDTC<br>(VS.VSDY) | VS.VSTPT | VS.VSSTRESC for<br>VS.VSTESTCD in<br>'SYSBP'/'DIABP' | VS.VSSTRESC<br>for<br>VS.VSTESTCD<br>'HR' | = | VS.VSSTRESC for<br>VS.VSTESTCD =<br>'RESP' | | VS.VSSTRESC<br>for<br>VS.VSTESTCD<br>'BMI' | = |
| Cohort:<br>ADSL.ACTARM | | | | | | VS.VSSTRESC<br>for<br>VS.VSTESTCD<br>'TEMP' | = | VS.VSSTRESC<br>for<br>VS.VSTESTCD<br>'WEIGHT' | = | VS.VSSTRESC<br>for<br>VS.VSTESTCD<br>'OXYSAT' |

Notes to programmer: If all of the tests are not done on a visit, put ND under Date Performed for that visit. If all of the tests are not done on a time-point on a certain visit put ND under each test corresponding to that time-point. If a particular test is not done on a visit or on a time point, put 'ND' under that test for that visit or time point.

ND = Not Done.

BSA = Body Surface Area.

Note: Study Day is relative to the date of the first T cell infusion, which is Study Day 1.


(Data as of: 24APR2018)

Protocol: GSK208466/ADP-04511

Population: Modified Intent-To-Treat

Listing 28.5102

Listing of Subjects with Potentially Clinically Significant Post-Baseline Vital Signs

| Subject | | Date/Time<br>Performed | | Blood Pressure<br>Systolic/Diastolic | Pulse<br>Rate | |
|---|---|---|---|---|---|---|
| ADSL.SUBJID | Visit | (Study Day) | Time-point | (mmHg) | (bpm) | |
| Cohort • | VS.VISIT | VS.VSDTC<br>(VS.VSDY) | VS.VSTPT | VS.VSSTRESC for<br>VS.VSTESTCD in<br>'SYSBP'/'DIABP' | VS.VSSTRESC<br>for<br>VS.VSTESTCD<br>'HR' | = |

Cohort:
ADSL.ACTARM

Notes to programmer: If all of the tests are not done on a visit, put ND under Date Performed for that visit. If all of the tests are not done on a time-point on a certain visit put ND under each test corresponding to that time-point. If a particular test is not done on a visit or on a time point, put 'ND' under that test for that visit or time point. The listing will contain all of a subject's values for parameters meeting the criteria.

ND = Not Done.

BSA = Body Surface Area.

Note 1: Potentially clinically significant vital signs criteria: heart rate is either less than 60 bpm or greater than 100 bpm; systolic blood pressure  $\geq$  140 mmHg; Diastolic  $\geq$  90 mmHg.

Note 2: Study Day is relative to the date of the first T cell infusion, which is Study Day 1.

208466/ADP-04511

Protocol: GSK208466/ADP-04511
Population: Intent-To-Treat

(Data as of: 24APR2018)


Listing 28.5201

ECOG Performance Status, Karnofsky Score, and Lansky Score

Cohort Date Performed Karnofsky Lansky
Subject Visit (Study Day) ECOG Score# Score (%) Score (%)

ND = Not Done, ECOG = Eastern Cooperative Oncology Group.

Note 1: The Lansky Score was assessed for children <= 10 years of age. The Karnofsky Score was optional.

Note 2: Study Day is relative to the date of the first T cell infusion, which is Study Day 1

# ECOG Score

0 = Fully active and able to carry on all pre-disease activities without restriction,

1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature,

2 = Ambulatory and capable of all self-care but unable to carry out any work activities,

3 = Capable of only limited self-care,

4 = Completely disabled,

5 = Dead.

208466/ADP-04511

Protocol: GSK208466/ADP-04511
Population: Intent-To-Treat

 (Data as of: 24APR2018)

Listing 28.6101 Electrocardiogram

| | | | Date/Time | | | Reason for |
|---|---|---|---|---|---|---|
| | | | Performed | | | Unscheduled |
| Cohort | Subject | Visit | (Study Day) | Assessment | Abnormalities | Assessment |

Notes to programmer: If all of the tests are not done on a visit(EGTESTCD = 'EGALL'), put 'ND' under Date Performed for that visit. If a particular test is not done on a visit, put 'ND' under that test for that visit.

\_\_\_\_\_

ND = Not Done.

Note: Study Day is relative to the date of the first T cell infusion, which is Study Day 1.

208466/ADP-04511

Protocol: GSK208466/ADP-04511 Population: Intent-To-Treat  (Data as of: 24APR2018)

Listing 28.6201
Physical Examination

Cohort Subject Date Performed

ADSL.ACTARM ADSL.SUBJID Visit (Study Day) Body System Abnormality

Notes to programmer: If Physical Examination is not performed, put ND under Date Performed. If Body System result was not done, put ND under Abnormality.

ND = Not Done.

Note 1: Only abnormalities and body systems not assessed are listed.

Note: Study Day is relative to the date of the first T cell infusion, which is Study Day 1.

Protocol: GSK208466/ADP-04511 Population: Intent-To-Treat  (Data as of: 24APR2018)

Listing 28.6301

Concomitant Medications

| | A:ATC-3 | | End Date | | | | |
|---|---|---|---|---|---|---|---|
| Subject | P:Preferred Name | Start Date | (Study Day) | Dose | | | |
| ADSL.SUBJID | V:Verbatim Name | (Study Day) | or Ongoing | (units) | Frequency | Route | Indication |
| | | | | | | | CM.CMINDC |
| Cohort | A: QVAL when QNAM = | | | | | | |
| ADSL.ACTARM | ATC3 | CM.CMSTDTC | CM.CMENDTC | | | | |
| | P: CM.CMDECOD | (CM.CMSTDY) | (CM.CMENDY) | | | | |
| | V: CM.CMTRT | | Or CM.CMENRF | | | | |

Note to programmer: If Unit, Frequency, or Route is Other, report this as Other: <Specify>.

Note 1: Only subjects reporting medications are listed.

Note 2: Medications are coded by WHO Drug Dictionary 2015-Dec.

Note 3: Study Day is relative to the date of the first T cell infusion, which is Study Day 1.

Note 4: If the 3rd level term is not available, the next available level is used.

# 208466/ADP-04511

Protocol: GSK208466/ADP-04511 Population: Intent-To-Treat  (Data as of: 24APR2018)

Listing 28.6401 Bridging Therapies

| Cohort | Subject | Start Date | Stop Date | Hospitalized | Therapy | Therapy | Dose | Disease |
|---|---|---|---|---|---|---|---|---|
| ADSL.ACTARM | ADSL.SUBJID | (Study Day) | (Study Day) | for Therapy? | Class | Description | Ordered | Status |

Note 1: Only subjects with cancer therapies given after apheresis and before lymphodepletion are listed.

Note 2: Study Day is relative to the date of the first T cell infusion, which is Study Day 1.

208466/ADP-04511

Protocol: GSK208466/ADP-04511 Population: Intent-To-Treat  (Data as of: 24APR2018)

Listing 28.6402 On-Study Surgery

T-Cell

Infusion Dates Organ - Site of Surgery

Description of Surgery

Surgery Date

ADSL.ACTARM

Cohort

Subject
ADSL.SUBJID

N = No, Y = Yes.

Note: Only subjects with surgery following T-cell administration are listed.

208466/ADP-04511

Protocol: GSK208466/ADP-04511 Population: Intent-To-Treat  (Data as of: 24APR2018)

Listing 28.6403

On-Study Oncology Treatment

CM.CMCAT = 'ON STUDY ONCOLOGY TREATMENT'
PR.PRCAT = 'ON STUDY ONCOLOGY TREATMENT'

| Cohort | Subject | T-Cell<br>Infusion | Therapy | Therapy | Dose | Start Date | End Date |
|---|---|---|---|---|---|---|---|
| ADSL.ACTARM | ADSL.SUBJID | Dates | Class | Description | Ordered | (Study Day) | (Study Day) |
| | | | 'RADIATION' | PRTRT | PRDOSTXT | | |
| | | | If from PR | CMTRT | CMDOSTXT | | |
| | | | CM.CMSCAT | | | | |

Note to programmer: All prior treatments from CM except for Radiation which is in S.PR

\_\_\_\_\_\_Note: Only subjects

reporting prior oncology treatment are listed.

208466/ADP-04511

Protocol: GSK208466/ADP-04511 Population: Intent-To-Treat  (Data as of: 24APR2018)

Listing 28.6404

Echocardiogram or Multigated Acquisition Scan (MUGA)

| | Subject | | Date Performed | Test | | Details of | LVEF |
|---|---|---|---|---|---|---|---|
| Cohort ADSL.ACTARM | ADSL.SUBJID | Visit | (Study Day) | Performed | Result | CS Abnormality | (%) |
| | | | | ECHO | | | |
| | | | | MUGA | | | |

CS = Clinically Significant, NCS = Not Clinically Significant, LVEF = Left Ventricular Ejection Fraction.

Note: Study Day is relative to the date of the first T cell infusion, which is Study Day 1.

208466/ADP-04511

Protocol: GSK208466/ADP-04511 Population: Intent-To-Treat  (Data as of: 24APR2018)

Listing 28.6502

EBV and Anti-CMV Status

Collection

Cohort Subject Visit (Study Day) EBV Status Anti-CMV Status

ADLBSP

ND = Not Done.

Note: Study Day is relative to the date of the first T cell infusion, which is Study Day 1.

208466/ADP-04511

Protocol: GSK208466/ADP-04511 Population: Intent-To-Treat

 (Data as of: 24APR2018)

Listing 28.6503

Infection Disease Testing

Date of Testing

(Study Day) Cohort Subject Visit

ND = Not Done.

Note: Study Day is relative to the date of the first T cell infusion, which is Study Day 1.